NCT #: NCT04590781



# CLINICAL STUDY PROTOCOL

A Phase 1b/2 Multiple-Dose Study to Evaluate the Safety and Efficacy of XmAb®18087 ± Pembrolizumab in Subjects with Advanced Merkel Cell Carcinoma or Extensive-stage Small Cell Lung Cancer (DUET-1-02)

Protocol No.: XmAb18087-02
IND No.: IND 136250
Test Product: XmAb®18087

Indications: Advanced Merkel Cell Carcinoma, Extensive-Stage Small Cell

Lung Cancer

Sponsor: Xencor, Inc.

111 West Lemon Avenue

Monrovia, CA 91016

Development Phase: Phase 1b/2

Sponsor Medical Expert:

Telephone:

Email:

Version and Date: Version 1.0 (18 August 2020)

## **Confidentiality Statement**

The confidential information in this document is provided to you as an Investigator, potential Investigator or consultant for review by you, your staff and applicable Independent Ethics Committee and/or Institutional Review Board. It is understood that the information will not be disclosed to others without written authorization from Xencor, Inc. except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

Version 1.0 

## SIGNATURE PAGES

## **Declaration of Sponsor or Responsible Medical Expert**

PROTOCOL TITLE: A Phase 1b/2 Multiple-Dose Study to Evaluate the Safety and Efficacy of XmAb®18087 ± Pembrolizumab in Subjects with Advanced Merkel Cell Carcinoma or Extensive-stage Small Cell Lung Cancer (DUET-1-02)

PROTOCOL NUMBER: XmAb18087-02

Xencor, Inc.

This clinical study protocol was subjected to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the investigational medicinal product (IMP), as well as with the moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (Version 2013), and the current guidelines on good clinical practices (GCP) applicable to this clinical study.

{See appended electronic signature page at the end of the document}

Xencor, Inc.


**Principal Investigator** 

## SIGNATURE PAGE

## **Declaration of the Principal Investigator**

PROTOCOL TITLE: A Phase 1b/2 Multiple-Dose Study to Evaluate the Safety and Efficacy of XmAb®18087 ± Pembrolizumab in Subjects with Advanced Merkel Cell Carcinoma or Extensive-stage Small Cell Lung Cancer (DUET-1-02)

This clinical study protocol was subjected to critical review and has been released by the Sponsor. I have read this protocol and agree that the information it contains is consistent with current risk and benefit evaluation of the IMP, as well as with the moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki (Version 2013), and the current guidelines on GCP applicable to this clinical study.

I will provide copies of the protocol and of the clinical and preclinical information on the investigational product, which was furnished to me by the Sponsor, to all members of the study team responsible to me who participate in the study. I will discuss this material with them to assure that they are fully informed regarding the study drug and the conduct of the study.

I will perform the study according to specifications outlined in the protocol and agree to implement protocol requirements only after this protocol version and the subject information/informed consent forms (ICF) have been approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). I will not modify this protocol without obtaining the prior approval of the Sponsor and of the IRB/IEC. I will submit any protocol modifications (amendments) and/or any ICF modifications to the Sponsor and the IRB/IEC, and approval will be obtained before any modifications are implemented.

I understand that the information presented in this study protocol is confidential, and I hereby assure that no information based on the conduct of the study will be released without prior consent from the Sponsor, Xencor, Inc., unless this requirement is superseded by a regulatory authority, eg, United States (US) Food and Drug Administration (FDA).

I agree to conduct the study as outlined in this clinical study protocol dated 18 August 2020. Any modification of the clinical study protocol must be agreed upon by the Sponsor and the Investigator(s) and must be documented in writing.

| <del>-</del> | |
|--------------|--------------------------|
| Name, Title | Date<br>(Day/Month/2020) |


# **GENERAL INFORMATION**

| Protocol Title: | A Phase 1b/2 Multiple-Dose Study to Evaluate the Safety and Efficacy of XmAb®18087 ± Pembrolizumab in Subjects with Advanced Merkel Cell Carcinoma or Extensive-stage Small Cell Lung Cancer (DUET-1-02) |
|---|---|
| Protocol No.: | XmAb18087-02 |
| Protocol Date: | Version 1.0, Original (18 August 2020) |
| Sponsor: | Xencor, Inc 111 West Lemon Avenue Monrovia, CA 91016 |
| Sponsor Medical Monitor: | Telephone: Email: |
| Adverse Event Reporting: | ICON Clinical Research Emergency phone number: (Toll free for US) (Toll number for US and outside of US) E-mail: (Americas) (Europe) |
| Clinical Research<br>Organization: | ICON Clinical Research Ltd South County Business Park Leopardstown Ireland |
| Clinical Laboratories: | ICON Laboratory Services 123 Smith Street Farmingdale, NY 11735 |
| Bioanalytical Laboratory (PK): | See Laboratory Manual for contact information. |
| Cytokine Laboratory: | See Laboratory Manual for contact information. |
| Immunogenicity (ADA) Assessment Laboratory: | See Laboratory Manual for contact information. |
| Flow Cytometry, B Cell,<br>NK Cell T Cell Assessment,<br>and Immunohistochemistry<br>Laboratory | See Laboratory Manual for contact information. |
| Merkel cell polyoma virus<br>antibody assay and<br>Immunohistochemistry<br>Laboratory | See Laboratory Manual for contact information. |


## 2. SYNOPSIS

Name of Sponsor/Company:

Xencor, Inc.

Name of Investigational Product:

XmAb®18087

Name of Active Ingredient:

XmAb18087

Protocol Number: XmAb18087-02 | Phase: 1b/2 | Country: United States

Title of Study:

A Phase 1b/2 Multiple-Dose Study to Evaluate the Safety and Efficacy of XmAb®18087 ± Pembrolizumab in Subjects with Advanced Merkel Cell Carcinoma or Extensive-stage Small Cell Lung Cancer (DUET-1-02)

**Study Center(s):** 

It is planned that up to 25 study centers will be initiated for this study in the United States.

**Publications:** 

None

**Planned Study Period:** 

Estimated date first subject enrolled: 31 March 2021

Estimated date last subject completed: 30 June 2024

**Development Phase:** 

Phase 1b/2

**Objectives:** 

## **Primary Objectives:**

The primary objectives of the study are as follows:

- 1. To determine the safety and efficacy (by overall response rate [ORR], complete response [CR], and partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria) of XmAb18087 monotherapy in subjects with advanced Merkel cell carcinoma (MCC) that has progressed after treatment with standard therapies
- 2. To determine the safety and efficacy (by ORR, CR, and PR per RECIST 1.1 criteria) of XmAb18087 in combination with pembrolizumab in subjects with advanced MCC who have not received prior anti-programmed cell death 1 (PD1) or anti-programmed cell death ligand 1 (PDL1) therapies, and for whom pembrolizumab as a single agent is indicated
- 3. To determine the safety and efficacy (by ORR, CR, and PR per RECIST 1.1 criteria) of XmAb18087 monotherapy in subjects with extensive-stage small cell lung cancer (SCLC) that has progressed after treatment with standard therapies

#### **Secondary Objectives:**

The secondary objectives of the study are as follows:

- 1. To assess antitumor activity of XmAb18087 by progression-free survival (PFS) per RECIST 1.1 criteria, as well as overall survival (OS) and duration of response, when administered with and without pembrolizumab in subjects with advanced MCC, and as monotherapy in subjects with extensive-stage SCLC
- 2. To characterize the pharmacokinetics (PK) and immunogenicity of XmAb18087 administered with and without pembrolizumab in subjects with advanced MCC, and as monotherapy in subjects with extensive-stage SCLC
- 3. To assess the PK profile (maximum observed serum concentration [C<sub>max</sub>] and C<sub>min[trough]</sub>) of pembrolizumab when co-administered with XmAb18087

## **Exploratory Objectives:**

The exploratory objectives of the study are as follows:


- 1. To assess the incidence, timing, and severity of cytokine release syndrome (CRS) by the following:
  - a. CRS-related adverse events (AEs), incidence and grade of AEs and incidence of serious adverse events [SAEs])
  - b. Biomarkers of CRS
- 2. To characterize the response to administration of XmAb18087 with and without pembrolizumab by assessment of cell surface markers on selected immune system cells in peripheral blood, including changes in lymphocyte subsets and in T-cell activation/exhaustion by flow cytometry and similar bioanalytical methods
- 3. To characterize pharmacodynamics (PD) by correlation of response with NETSPOT® (gallium 68 dotatate) positron emission tomography/computed tomography (PET/CT) scan results after XmAb18087 administration with and without pembrolizumab
- 4. To evaluate by immunohistochemistry tumor-cell expression of somatostatin receptor 2 (SSTR2) and PDL1 on tumor cells and tumor-infiltrating T cells for expression of proliferation markers and PD1/PDL1 after XmAb18087 administration with and without pembrolizumab, as well as changes in other immune cell subsets
- 5. To characterize the pharmacodynamic changes in the intratumoral inflammatory response using immunostaining of immune cells and analysis of RNA signatures
- 6. To correlate response in MCC subjects to Merkel cell polyomavirus (MCPyV) status as determined by serology and immunohistochemistry

#### Methodology:

This is a Phase 1b/2, multiple-dose study designed to describe safety and efficacy, and to assess PK and immunogenicity of XmAb18087 monotherapy and in combination with pembrolizumab in subjects with metastatic MCC or locoregional MCC that has recurred after locoregional therapy with surgery and/or radiation therapy, and XmAb18087 monotherapy in subjects with extensive-stage SCLC that has progressed after standard therapies.

Part A of the study will enroll safety run-in cohorts of subjects with advanced MCC that has progressed after treatment with standard therapies to confirm the safety and tolerability of the XmAb18087 monotherapy administered intravenously (IV) with weekly step-up dosing for 42-day cycles. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 monotherapy using the recommended dose (RD) identified following the safety run-in.

Part B of the study will enroll safety run-in cohorts of subjects with advanced MCC not previously treated with anti-PD1 or anti-PDL1 agents, and for whom pembrolizumab as a single agent is indicated, to confirm the safety and tolerability of XmAb18087 in combination with pembrolizumab. Subjects will receive step-up IV dosing of XmAb18087 on Days 1, 8, 22, 29, and 36, and IV dosing of pembrolizumab on Day 15 of each 42-day cycle. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 plus pembrolizumab combination therapy using the RD identified following the safety run-in.

Enrollment into the first safety run-in cohort of Part B (Cohort 1B) may begin after the first safety run-in cohort in Part A (Cohort 1A, one dose level higher than Cohort 1B) has completed the first cycle and the regimen has been demonstrated to be tolerable.

Part C of the study will enroll safety run-in cohorts of subjects with extensive-stage SCLC that has progressed after treatment with standard therapies to confirm the safety and tolerability the same XmAb18087 monotherapy. The safety run-in will follow the same cohort schema as described for Part A to identify a RD for expansion in SCLC. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 monotherapy using the RD identified following the safety run-in.

Enrollment into Part C may begin concurrently with Part A.

## **Termination of Study**

If the Investigator or the Sponsor becomes aware of conditions or events that suggest a possible hazard to subjects should the clinical study continue, the clinical study may be terminated after appropriate consultation among the involved parties. The clinical study also may be terminated at the Sponsor's discretion, also in the absence of such a finding.

Conditions that may warrant termination of the clinical study include, but are not limited to:

The discovery of an unexpected, relevant, or unacceptable risk to the subjects enrolled in the clinical study.


- Failure to enroll subjects at the required rate.
- A decision of the Sponsor to suspend or discontinue development of the investigational medicinal product (IMP).

Should the study be terminated and/or the site closed for whatever reason, all documentation pertaining to the study and IMP must be returned to the Sponsor. Any actions required for assessing or maintaining subject safety will continue as required, despite termination of the study by the Sponsor.

#### **Treatment Plan:**

Part A, which will enroll subjects with previously treated advanced MCC, consists of safety-run in cohorts followed by an expansion cohort. For the first safety run-in cohort (Cohort 1A), 3 to 6 subjects will be enrolled and will receive step-up dosing as follows: 0.3 μg/kg on Day 1, followed by 1.0 μg/kg on Days 8, 15, 22, 29, and 36 of the first cycle, and Days 1, 8, 15, 22, 29, and 36 of all subsequent cycles. If the Cohort 1A regimen is not tolerated, lower dose levels may be explored. If the Cohort 1A regimen is tolerated, 3 to 6 subjects will be enrolled in Cohort 2A and will receive step-up dosing as follows: 0.3 μg/kg on Day 1, 1.0 μg/kg on Day 8, and 2.0 μg/kg on Days 15, 22, 29, and 36 of the first cycle and Days 1, 8, 15, 22, 29, and 36 of all subsequent cycles. If this regimen is tolerated, 3 to 6 subjects will be enrolled in Cohort 3A and will receive step-up dosing as follows: 0.3 μg/kg on Day 1, 1.0 μg/kg on Day 8, 2.0 μg/kg on Day 15, and 4.0 μg/kg on Days 22, 29, and 36 of the first cycle and Days 1, 8, 15, 22, 29, and 36 of the first cycle and Days 1, 8, 15, 22, 29, and 36 of all subsequent cycles. See Cohort Table A.

Based on assessments of tolerability, safety, and PK data from all the safety run-in cohorts in Part A, an RD regimen for expansion will be selected. Up to 9 subjects will be enrolled at the RD. If at least 1 subject shows a response by RECIST 1.1 criteria, then enrollment will continue up to a total of 22 subjects to evaluate efficacy.

Part B, which will enroll subjects with advanced MCC not previously treated with anti-PD1 or anti-PDL1 agents, consists of safety run-in cohorts followed by an expansion cohort. Safety run-in Cohort 1B (one dose level below Cohort 1A) will begin enrolling after Cohort 1A is completed and the dosing regimen is deemed tolerable. For all Part B cohorts, 400 mg pembrolizumab will be administered IV on Day 15 of each 42-day cycle. Three to 6 subjects will be enrolled in Cohort 1B and will receive XmAb18087 administered IV as follows: 0.3  $\mu$ g/kg on Days 1, 8, 22, 29, and 36 of all cycles. If this regimen is tolerated, 3 to 6 additional safety run-in subjects will be enrolled in Cohort 2B and will receive step-up IV dosing of XmAb18087 as follows: 0.3  $\mu$ g/kg on Day 1, then 1.0  $\mu$ g/kg on Days 8, 22, 29, and 36 of the first cycle and Days 1, 8, 22, 29, and 36 of all subsequent cycles. If this regimen is tolerated, 3 to 6 subjects will be enrolled in Cohort 3B and will receive step-up IV dosing of XmAb18087 as follows: 0.3  $\mu$ g/kg on Day 1, 1.0  $\mu$ g/kg on Days 8 and 22, then 2.0  $\mu$ g/kg on Days 29 and 36 of the first cycle and Days 1, 8, 22, 29, and 36 of all subsequent cycles. If this regimen is tolerated, 3 to 6 subjects will be enrolled in Cohort 4B and will receive step-up IV dosing of XmAb18087 as follows: 0.3  $\mu$ g/kg on Day 1, 1.0  $\mu$ g/kg on Days 8 and 22, 2.0  $\mu$ g/kg on Days 29 and 36 of the first cycle and Day 1 of all subsequent cycles, and 4.0  $\mu$ g/kg and Days 1, 8, 22, 29, and 36 of all cycles after the first cycle. See Cohort Table B.

Based on assessments of tolerability, safety, and PK data from all the safety run-in cohorts in Part B, an RD for expansion will be selected. Up to 12 subjects will be enrolled at the RD. If at least 4 subjects show a response by RECIST 1.1 criteria, enrollment will continue up to a total of 30 subjects to evaluate efficacy.

Part C will enroll subjects with previously treated extensive-stage SCLC and consists of safety-run in cohorts followed by an expansion cohort. Part C will follow the same safety run-in schema as described for Part A. See Cohort Table C.

Based on assessments of tolerability, safety, and PK data from all the safety run-in cohorts in Part C, an RD for expansion will be selected. Up to 9 subjects will be enrolled at the RD. If at least 1 subject shows a response by RECIST 1.1 criteria, then enrollment will continue up to a total of 30 subjects to evaluate efficacy. Throughout the study, SSTR2 expression levels and prevalence will be assessed histologically using tumor biopsies from enrolled subjects; a higher number of subjects may be enrolled in the Part C expansion cohort based on these assessments.

Parts A, B, and C: The decision to advance to higher dose levels after each safety run-in cohort will be made by a Safety Review Committee (SRC) based on review of the aggregate safety data for all subjects in that cohort as well as cumulative safety data for the study overall. The SRC will be allowed to make adaptations to the dosing schema, if needed, in accordance with evolving trial safety and tolerability findings, as long as adaptations do not significantly increase subject risk. Any such adaptations would require a protocol amendment and Institutional Review Board (IRB) approval.




MCC = Merkel cell carcinoma; PD1 = programmed cell death protein 1; PDL1 = programmed cell death ligand 1; SCLC = small cell lung cancer.

#### **Number of Subjects:**

Up to 142 subjects will be enrolled.

## Diagnosis and Main Criteria for Inclusion/Exclusion:

#### **Inclusion Criteria for All Cohorts**

Each subject must meet all of the following inclusion criteria to be enrolled in the study:

- Able to provide written informed consent
- Adult subjects  $\geq$  18 years
- Disease measurable by RECIST 1.1 criteria using either CT or magnetic resonance imaging (MRI) scan
- Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
- All subjects must have adequate archival tumor sample (slides or archival formalin-fixed paraffin-embedded [FFPE] block[s] containing tumor that has not been previously irradiated; FFPE blocks are preferred to slides, and newly obtained biopsies are preferred to archived tissue. Refer to the laboratory manual for further instructions). Excepted are subjects who consent to having a fresh tumor biopsy to provide a fresh tumor sample instead of the archival tumor sample.
- Female subjects of childbearing potential must agree to use a highly effective method of birth control during and for 4 weeks after completion of study. Women are considered to be of childbearing potential unless it is documented that they are over the age of 60 OR postmenopausal by history with no menses for 1 year and confirmed by follicle-stimulating hormone (FSH; using local reference ranges) OR have a history of hysterectomy and/or bilateral oophorectomy OR have a history of bilateral tubal ligation. Highly effective methods of birth control include combined hormonal birth control (oral, intravaginal, or transdermal), or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or intrauterine), intrauterine devices (IUDs), intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner (provided partner is the sole sexual partner and there has been a medical assessment of surgical success), or sexual abstinence as defined in Section 8.9.1.
- Fertile male subjects must be willing to practice a highly effective method of birth control for the duration of the study and continuing for 4 weeks after the last dose of XmAb18087 or pembrolizumab (when applicable).


Highly effective methods of birth control include vasectomy or a condom in combination with double-barrier methods, spermicide, hormonal birth control, or IUD (nonhormonal) used by the woman.

· Able and willing to complete the entire study according to the study schedule

#### Additional Inclusion Criteria for Part A and Part B Cohorts:

In addition to the inclusion criteria above, the following criteria are required for Parts A and B safety run-in and expansion cohorts:

• Histologically or cytologically confirmed metastatic MCC or locoregional MCC that has recurred following standard locoregional therapy with surgery and/or radiation therapy

#### **Additional Inclusion Criteria for Part A Cohorts:**

In addition to the inclusion criteria above, the following criteria are required for Part A safety run-in and expansion cohorts:

Subjects must have progressed on or been ineligible for treatment with anti-PD1 or anti PDL1 therapy.

#### **Additional Inclusion Criteria for Part B Cohorts:**

In addition to the inclusion criteria above, the following criteria are required for Part B safety run in and expansion cohorts:

• Subjects must be eligible to receive pembrolizumab as standard of care.

#### **Additional Inclusion Criteria for Part C Cohorts:**

In addition to the inclusion criteria above, the following criteria are required for Part C safety run-in and expansion cohorts:

 Histologically or cytologically confirmed extensive-stage SCLC that has progressed following standard therapies

#### **Exclusion Criteria for All Cohorts**

Subjects who meet any of the following criteria will be excluded from the study:

- · History of prior organ or bone marrow transplant
- History of chronic lymphocytic leukemia
- Subjects currently receiving anticancer therapies
- Subjects who have received anticancer therapies within 2 weeks of the start of study drug (including chemotherapy, radiation therapy, immunotherapy, etc.)
- Prior therapy with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA4, OX40, CD137) AND were permanently discontinued from that treatment due to an immune-related adverse event (IRAE)
- Failure to recover from any IRAE from prior cancer therapy to  $\leq$  Grade 1 (participants with  $\leq$  Grade 2 neuropathy or endocrinopathies controlled by hormone replacement are eligible)
- Failure to recover from any other toxicity (other than immune-related toxicity) from previous anticancer treatment to ≤ Grade 2
- Known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days prior to trial treatment.
- Have a history of (noninfectious) pneumonitis that required steroids or have current pneumonitis (history of radiographically visible but asymptomatic radiation pneumonitis is allowed)
- Platelet count  $< 50 \times 10^9/L$
- Absolute neutrophil count  $< 1.0 \times 10^9/L$
- Aspartate aminotransferase (AST) ≥ 3 × upper limit of normal (ULN), or if subject has known liver metastases, AST ≥ 7 × ULN
- Alanine aminotransferase (ALT)  $\geq 3 \times ULN$ , or if subject has known liver metastases, ALT  $\geq 7 \times ULN$


- Estimated creatinine clearance < 50 mL/min calculated by the Cockcroft Gault or Modification of Diet in Renal Disease formulas at screening
- Treatment with immunosuppressive therapy within 28 days of first dose of study drug
- History or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary, renal, metabolic, hematologic, or psychiatric) other than their primary malignancy that in the opinion of the Investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
- Treatment for any serious bacterial, viral, parasitic, or systemic fungal infections within the 30 days prior to study entry
- Active known or suspected COVID-19 disease
- Active known or suspected autoimmune disease (except that subjects are permitted to enroll if they have
  vitiligo; type 1 diabetes mellitus; residual hypothyroidism due to an autoimmune condition that is treatable
  with hormone replacement therapy only; psoriasis, atopic dermatitis, or another autoimmune skin condition
  that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral
  acetaminophen and nonsteroidal anti-inflammatory drugs [NSAIDS])
- Positive test for human immunodeficiency virus (HIV) or hepatitis C antibodies
- Positive test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb; a subject whose HBsAg is negative and HBcAb is positive may be enrolled if a hepatitis B virus [HBV] DNA test is negative and either the subject is treated with potent antiviral therapy or is retested for HBsAg and HBV DNA every month)
- Subject is pregnant or breastfeeding, planning to become pregnant, or expecting to conceive or father children while enrolled in the study, up to the end of study (EOS) visit.
- Positive serum pregnancy test (ie, urine human chorionic gonadotropin) at screening

#### Additional Exclusion Criteria for Part B Cohorts:

In addition to the exclusion criteria above, subjects will be excluded from Part B cohorts administered XmAb18087 in combination with pembrolizumab if they meet the following criteria:

- Prior treatment with therapeutics directed at anti-programmed cell death 1 (anti-PD1) or anti-programmed cell death ligand 1 (anti-PDL1)
- Have severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients

#### Test Product, Dose, and Mode of Administration:

XmAb18087 is a humanized bispecific antibody (bsAb) that binds both the tumor antigen SSTR2 and CD3 antigen to recruit cytotoxic T cells for killing of SSTR2<sup>+</sup> tumor cells.

The cohorts and dose levels to be administered in this clinical trial are shown below.


## Cohorts

Cohort Table A: Part A (MCC) Monotherapy Safety Run-in and Expansion Cohorts

| | C 1 | | | Cycle 1 | | | | | | Cycle 2+ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cycle<br>and Day | <b>D</b> 1 | D8 | D15 | D22 | D29 | D36 | <b>D40</b> | <b>D</b> 1 | D8 | D15 | D22 | D29 | D36 | <b>D40</b> | |
| | | | | | | | | ± 2 | | | | | | | ± 2 | |
| | Drug | | | XmA | b1808 | 7 | | EA | | 2 | XmAb | 18087 | | | EA | |
| | | | | (μ <u>ε</u> | g/kg) | | | | | | (μg/ | kg) | | | | |
| | Study | 1 | 8 | 15 | 22 | 29 | 36 | 40 | 43 | 50 | 57 | 64 | 71 | 78 | 82 | |
| | Day | | | | | | | | | | | | | | | |
| Part A | 1A | 0.3 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 3 – 6 |
| (Safety | 2A | 0.3 | 1.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 3 - 6 |
| Run-in) | 3A | 0.3 | 1.0 | 2.0 | 4.0 | 4.0 | 4.0 | 1 | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | | 3 - 6 |
| Part A | Expansion | | | | | | | Δ+1 | RD coho | rt | | | | | | Up to 22 |
| (Expansion) | A | | | | | | | Atı | XD COIIO | 1 t | | | | | | Op 10 22 |

D = day; EA = efficacy assessment (no drug administered). Maximum escalated dose for each cohort in bold.


Cohort Table B: Part B (MCC) Combination Therapy Safety Run-in and Expansion Cohorts

| | Cycle | | Cycle 1 | | | | | | | | Subjects | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | and Day | D1 | D8 | D15 | D22 | D29 | D36 | D40 | D1 | D8 | D15 | D22 | D29 | D36 | D40 | |
| | Drug | VmAh | 10007 | Pem | V. | n 4 h 1 9 | 0007 | ± 2 | VmAh | 19097 | Pem | Vn | a A b 1 Q | 007 | ± 2<br>EA | |
| | Drug | XmAb18087<br>(μg/kg) | | (mg) | XmAb18087 ΕΑ<br>(μg/kg) | | | LA | XmAb18087<br>(µg/kg) | | (mg) | | KmAb18087<br>(μg/kg) | | LA | |
| | Study<br>Day | 1 | 8 | 15 | 22 | 29 | 36 | 40 | 43 | 50 | 57 | 64 | 71 | 78 | 82 | |
| | 1B | 0.3 | 0.3 | 400 | 0.3 | 0.3 | 0.3 | | 0.3 | 0.3 | 400 | 0.3 | 0.3 | 0.3 | | 3 – 6 |
| Part B<br>(Safety | 2B | 0.3 | 1.0 | 400 | 1.0 | 1.0 | 1.0 | | 1.0 | 1.0 | 400 | 1.0 | 1.0 | 1.0 | | 3 – 6 |
| Run-in) | 3B | 0.3 | 1.0 | 400 | 1.0 | 2.0 | 2.0 | | 2.0 | 2.0 | 400 | 2.0 | 2.0 | 2.0 | | 3 – 6 |
| | 4B | 0.3 | 1.0 | 400 | 1.0 | 2.0 | 2.0 | | 2.0 | 4.0 | 400 | 4.0 | 4.0 | 4.0 | | 3 – 6 |
| Part B (Expansion) | Expansion B | | | | | | | At RD | cohort | | | | | | | Up to 30 |

D = day; EA = efficacy assessment (no drug administered); Pem = pembrolizumab. Maximum escalated dose for each cohort in bold.


| | , |
|---------|----------------|
| Protoco | l XmAb18087-02 |

| Cohort Table C: | Part C (SCLC) | ) Mon | otheraj | y Safe | ty Run- | in and I | Expansi | on Cohor | ts | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | G 1 | | Cycle 1 Cycle 2+ | | | | | | | | | | | | Subjects | |
| | Cycle and Day | D1 | D8 | D15 | D22 | D29 | D36 | D40 | D1 | D8 | D15 | D22 | D29 | D36 | D40 | |
| | | | | | | | | ± 2 | | | | | | | ± 2 | |
| | Drug | | | XmA | b1808 | 7 | | EA | | | XmAb | 18087 | | | EA | |
| | | | (μg/kg) | | | | | | (μg/kg) | | | | | | | |
| | Study<br>Day | 1 | 8 | 15 | 22 | 29 | 36 | 40 | 43 | 50 | 57 | 64 | 71 | 78 | 82 | |
| Part C | 1C | 0.3 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 3 - 6 |
| (Safety | 2C | 0.3 | 1.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 3 – 6 |
| Run-in) | 3C | 0.3 | 1.0 | 2.0 | 4.0 | 4.0 | 4.0 | | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | | 3 - 6 |
| Part C<br>(Expansion) | Expansion C | | | | | | | At ] | RD coho | rt | | | | | | Up to 30 |

D = day; EA = efficacy assessment (no drug administered). Maximum escalated dose for each cohort in bold.


## Reference Therapy, Dosage, and Mode of Administration:

None

#### **Duration of Treatment:**

Each treatment cycle (Parts A, B, and C) is 42 days long. In Parts A and C, each cycle will consist of 6 weekly doses of XmAb18087 (on Days 1, 8, 15, 22, 29, and 36). In Part B, each cycle will consist of 6 weekly doses of either XmAb18087 or pembrolizumab: 5 doses of XmAb18087 (on Days 1, 8, 22, 29, and 36) and 1 dose of pembrolizumab (on Day 15).

#### **Criteria for Evaluation:**

#### Safety:

As assessed by AEs, vital signs, physical examination (PE) findings, clinical laboratory safety assessments, and electrocardiogram (ECG) parameters:

• Incidence of treatment-emergent AEs (TEAEs), treatment-emergent serious adverse events (TESAEs), treatment-related TEAEs and TESAEs, TEAEs by severity as defined in the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, and TEAEs resulting in the permanent discontinuation of XmAb18087 or pembrolizumab.

#### **Efficacy:**

Antitumor activity of XmAb18087 as assessed by response rates (ORR, CR rate, PR rate), duration of response, PFS, and OS.

#### **Pharmacokinetics:**

Pharmacokinetic parameters including  $C_{max}$ , time to reach maximum concentration ( $t_{max}$ ), half-life ( $t_{1/2}$ ), area under the serum concentration-time curve from time zero to infinity ( $AUC_{0-\infty}$ ), clearance (CL), volume of distribution (Vd), and volume of distribution at steady state ( $Vd_{ss}$ ) will be estimated using either noncompartmental or compartmental methods, whichever best describes the observed data. Pharmacokinetic parameters for XmAb18087 will be compared with and without pembrolizumab administration.

#### Pharmacodynamics:

Baseline and serial assessment of B-cell, NK-cell, and T-cell numbers and T-cell activation will be assessed in peripheral venous blood.

## **Endpoints:**

## **Primary Endpoints:**

The primary endpoints are as follows:

- Safety of (1) XmAb18087 monotherapy in MCC and SCLC, and (2) XmAb18087 and pembrolizumab combination therapy in MCC, as assessed by the following:
  - Incidence of TEAEs
  - Incidence of clinically significant changes in safety laboratory tests, PE findings, vital signs, and ECGs
  - Incidence and severity of CRS
- Efficacy of (1) XmAb18087 monotherapy in MCC and SCLC, and (2) XmAb18087 and pembrolizumab combination therapy in MCC using RECIST 1.1 assessment of CT/MRI imaging, as well as aggregate data, for the following:
  - ORR
  - CR rate
  - PR rate

## **Secondary Endpoints:**

The secondary endpoints are as follows:

- Efficacy of (1) XmAb18087 monotherapy in MCC and SCLC, and (2) XmAb18087 and pembrolizumab combination therapy in MCC using RECIST 1.1 assessment of CT/MRI imaging, as well as aggregate data, for the following:
  - Duration of response


- PFS
- OS
- PK characterization of XmAb18087, when administered as monotherapy and in combination with pembrolizumab, based on the parameters of C<sub>max</sub>, t<sub>max</sub>, t<sub>1/2</sub>, AUC<sub>0-∞</sub>, CL, Vd, and Vd<sub>ss</sub>. Further details will be defined in a PK analysis plan.
- Assessment of immunogenicity by incidence of anti-XmAb18087 antibodies and qualitative assessment of safety outcomes
- PK characterization of pembrolizumab, when administered in combination with XmAb18087, based on parameters similar to those for XmAb18087, with further details to be provided in a PK analysis plan.

#### **Exploratory Endpoints:**

The exploratory endpoints are as follows:

- Assessment of peripheral blood for cell surface markers by flow cytometry and similar bioanalytical methods
  that evaluate the response of selected immune system cells following administration of XmAb18087 as a
  monotherapy and in combination with pembrolizumab, including changes in lymphocyte subsets and in T-cell
  activation and exhaustion markers
- PD characterized by NETSPOT (gallium 68 dotatate) PET/CT results and by tumor cell expression of SSTR2 and PDL1 and tumor-infiltrating immune-cell expression of PD1/PDL1 and other markers by immunohistochemistry, in response to administration of XmAb18087 monotherapy and in combination with pembrolizumab
- PD: immunohistochemistry (IHC) SSTR2 panel
- PD: MCC and SCLC IHC panels
- Correlation of clinical/radiographic response with MCPyV serology (MCC subjects only)
- Additional exploratory genetic, cellular, and/or serum markers of potential future interest. If evidence of therapeutic activity is seen with XmAb18087, biobanked samples may be assessed for genetic and immunologic factors that might predict response or nonresponse (optional part of study and may be reported separately from the clinical study report). Samples will not be retained for more than 15 years.

#### **Statistical Methods:**

#### **Analysis Populations:**

The populations defined below will be used for analysis:

- Safety population: All subjects who are enrolled and receive at least 1 infusion of XmAb18087.
- Evaluable population: All subjects who are enrolled, receive at least 1 cycle (Parts A and C: 6 doses XmAb18087, Part B: 5 doses XmAb18087 and 1 dose pembrolizumab) of XmAb18087 and have at least 1 postbaseline RECIST 1.1 assessment of tumor imaging available.
- **PD population:** All subjects who are enrolled, receive at least 1 dose of XmAb18087 (and 1 infusion of pembrolizumab, when relevant for a particular PD assessment), and have at least 1 preinfusion and 1 postinfusion set of biomarker data available for analysis.
- **PK populations:** All subjects who are enrolled and receive at least 1 dose of XmAb18087 (ie, the XmAb18087 PK population) or 1 infusion of pembrolizumab, (ie, the pembrolizumab PK population), and have at least 1 set of postinfusion PK data available for analysis.

Continuous data will be presented using descriptive statistics: number of subjects (N), mean, standard deviation, median, minimum, and maximum. Categorical data will be summarized by the number and percentage, where the percentage is presented in brackets to 1 decimal place. Safety and efficacy summaries will be provided for the monotherapy and combination therapy arms separately, as well as for the combined arms.

Date of the Protocol: 18 August 2020


# 3. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

# TABLE OF CONTENTS

| 1. | TITLE PAGE | 1 |
|---|---|---|
| SIGNAT | URE PAGES | 2 |
| GENER! | L INFORMATION | 4 |
| 2. | SYNOPSIS | 5 |
| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 16 |
| LIST OF | TABLES | 21 |
| LIST OF | FIGURES | 22 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 23 |
| 5. | INTRODUCTION | 27 |
| 5.1. | Background | 27 |
| 5.1.1. | Somatostatin and Somatostatin Receptors. | 27 |
| 5.1.2. | Merkel Cell Carcinoma | 27 |
| 5.1.3. | Small Cell Lung Cancer. | 29 |
| 5.1.4. | Therapeutic Bispecific Antibodies | 29 |
| 5.1.5. | XmAb18087 Product Description | 29 |
| 5.1.6. | Preclinical Studies | 30 |
| 5.1.6.1. | Pharmacology | 30 |
| 5.1.6.2. | Pharmacokinetics and Toxicokinetics | 33 |
| 5.1.6.3. | Toxicology | 34 |
| 5.1.7. | Human Experience with XmAb18087 and Related Molecules | 36 |
| 5.2. | Pembrolizumab | 37 |
| 5.2.1. | Pharmaceutical and Therapeutic Background | 37 |
| 5.2.2. | Nonclinical Studies | 38 |
| 5.2.3. | Justification for Pembrolizumab Dose | 38 |
| 5.3. | Rationale for Dose Selection of XmAb18087-01 FIH, XmAb18087-02, and Study Design | 38 |
| 6. | STUDY OBJECTIVES | 40 |
| 6.1. | Primary Objectives | 40 |
| 6.2. | Secondary Objectives | 40 |

| 6.3. | Exploratory Objectives | 40 |
|---|---|---|
| 7. | INVESTIGATIONAL PLAN | 42 |
| 7.1. | Overall Study Design and Plan. | 42 |
| 7.2. | Study Flowcharts | 44 |
| 7.3. | Dosing Schedule | 44 |
| 7.4. | Continuation/Discontinuation of Therapy | 49 |
| 7.4.1. | Continuation Prior to Progression | 49 |
| 7.4.2. | Continuation/Discontinuation at Progression | 49 |
| 7.4.3. | Intrasubject Dose Escalation. | 50 |
| 7.5. | Number of Subjects | 50 |
| 7.6. | Treatment Assignment | 50 |
| 7.7. | Safety Run-in Cohorts | 51 |
| 7.8. | Criteria for Adverse Events of Specific Concern and Dose Adjustment | 51 |
| 7.8.1. | Replacement of Subjects. | 52 |
| 7.8.2. | Criteria for Study Termination | 52 |
| 7.9. | Study Assessments | 53 |
| 7.9.1. | Pretreatment Evaluations | 60 |
| 7.9.1.1. | Screening Period (Day -28 to -2) | 60 |
| 7.9.1.2. | Baseline Assessments (Day -1 or 1) | 61 |
| 7.9.2. | Subject Enrollment | 62 |
| 7.9.3. | Treatment Cycle Assessments | 62 |
| 7.9.3.1. | Clinical Assessments | 62 |
| 7.9.3.2. | Laboratory Assessments | 63 |
| 7.9.3.3. | End-of-Treatment Visit. | 64 |
| 7.9.4. | Post-treatment Follow-up Period (2 Weeks and 4 Weeks After EOT) | 64 |
| 7.9.5. | Long-Term Follow-up Period (6 and 12 Months After EOT) | 64 |
| 7.10. | Discussion of Study Design | 64 |
| 7.10.1. | Risk/Benefit and Ethical Assessment | 65 |
| 7.10.2. | Termination of Study | 65 |
| 8. | SELECTION AND WITHDRAWAL OF SUBJECTS | 66 |
| 8.1. | Inclusion Criteria for All Cohorts | 66 |
| 8.2. | Additional Inclusion Criteria for Part A and Part B Cohorts: | 66 |
| 8.3 | Additional Inclusion Criteria for Part A Cohorts: | 67 |

| 8.4. | Additional Inclusion Criteria for Part B Cohorts: | 67 |
|---|---|---|
| 8.5. | Additional Inclusion Criteria for Part C Cohorts: | 67 |
| 8.6. | Exclusion Criteria for All Cohorts. | 67 |
| 8.7. | Additional Exclusion Criteria for Part B Cohorts: XmAb18087 in Combination with Pembrolizumab | 69 |
| 8.8. | Withdrawal of Subjects | 69 |
| 8.9. | Other Subject Restrictions | 70 |
| 8.9.1. | Avoidance of Pregnancy | 70 |
| 8.9.2. | Use in Nursing Women | 70 |
| 9. | TREATMENT OF SUBJECTS | 71 |
| 9.1. | Identity of Study Treatments | 71 |
| 9.2. | Concomitant Therapy | 71 |
| 9.2.1. | Permitted Medications | 71 |
| 9.2.2. | Excluded Medications | 72 |
| 9.3. | Subject Compliance | 72 |
| 9.4. | Blinding and Randomization of Study Treatment | 72 |
| 9.5. | Procedure for Breaking the Randomization Code | 72 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 73 |
| 10.1. | XmAb18087 | 73 |
| 10.1.1. | Pretreatment of XmAb18087 | 73 |
| 10.1.2. | Prophylaxis of Nausea and Vomiting | 73 |
| 10.1.3. | Prophylaxis of Infusion Reactions/Cytokine Release Syndrome: | 73 |
| 10.1.4. | Administration of XmAb18087 | 74 |
| 10.2. | Pembrolizumab (Keytruda®) | 74 |
| 10.2.1. | Administration of Pembrolizumab | 74 |
| 10.2.2. | Treatment of Overdose | 75 |
| 10.3. | Safety Criteria for Dose Adjustment or Stopping Dose | 75 |
| 10.3.1. | Criteria for Adjustment or Stopping Dose of XmAb18087 | 75 |
| 10.3.2. | Criteria for Adjustment or Stopping Dose of Pembrolizumab | 76 |
| 10.4. | Study Treatment Packaging and Labelling | 76 |
| 10.4.1. | Packaging and Labelling of XmAb18087 | 76 |
| 10.4.2. | Storage of XmAb18087 | 76 |
| 10.4.3. | Preparation of XmAb18087 | 76 |

| 10.4.4. | Packaging and Labeling of Pembrolizumab | 76 |
|---|---|---|
| 10.4.5. | Storage of Pembrolizumab | 77 |
| 10.5. | Study Treatment Accountability, Handling, and Disposal | 77 |
| 11. | ASSESSMENT OF SAFETY | 78 |
| 11.1. | Adverse Events | 78 |
| 11.1.1. | Definitions | 78 |
| 11.1.2. | Recording of Adverse Events | 80 |
| 11.1.2.1. | Intensity | 80 |
| 11.1.2.2. | Causality | 81 |
| 11.1.2.3. | Action Taken with Study Treatment. | 82 |
| 11.1.2.4. | Outcome | 82 |
| 11.1.3. | Preidentified Immune-Mediated Adverse Events. | 83 |
| 11.1.4. | Adverse Events of Special Interest | 83 |
| 11.1.4.1. | Deaths | 83 |
| 11.1.4.2. | Pregnancy | 83 |
| 11.1.5. | Reporting Serious Adverse Events | 84 |
| 11.1.6. | Follow-up of Adverse Events | 85 |
| 11.1.7. | Treatment/Reporting of Overdose | 85 |
| 11.2. | Investigational New Drug Safety Reports | 86 |
| 11.3. | Guidelines for Prophylaxis and Management of Hypersensitivity Reactions, Cytokine Release Syndrome, and Neurological Toxicity Attributed to XmAb18087 | 86 |
| 11.3.1. | Introduction and Grading. | |
| 11.3.2. | Cytokine Release Syndrome Versus Allergic or Hypersensitivity Reactions | |
| 11.3.3. | Treatment Guidelines for Cytokine Release Syndrome | |
| 11.3.3.1. | Use of Tocilizumab for Cytokine Release Syndrome | |
| 11.3.3.2. | Fluid Management | |
| 11.3.3.3. | Cytokine Release Syndrome Treatment Guidelines by Grade | |
| 11.3.3.4. | Neurotoxicity | 91 |
| 11.4. | Guidelines for Prophylaxis and Management of Infusion Reactions Attributed to Pembrolizumab | 94 |
| 11.5. | Laboratory Assessments | 94 |
| 11.6. | Electrocardiogram Assessments | 95 |

| 11.7. | Physical Examination | 95 |
|---|---|---|
| 11.8. | Vital Signs | 95 |
| 12. | ASSESSMENT OF EFFICACY | 97 |
| 13. | PHARMACOKINETIC/PHARMACODYNAMIC ASSESSMENTS | 97 |
| 13.1. | Serum Sampling for Pharmacokinetic Analyses, Anti-drug Antibodies, Cytokines, and Inflammatory Factors | 97 |
| 13.2. | Pharmacokinetics | 97 |
| 13.3. | Pharmacodynamics | 97 |
| 13.4. | Biobanking Samples | 98 |
| 14. | STATISTICAL EVALUATION | 99 |
| 14.1. | Sample Size and Power | 99 |
| 14.2. | Statistical Methods | 99 |
| 14.3. | Study Endpoints | 99 |
| 14.3.1. | Primary Endpoints | 99 |
| 14.3.2. | Secondary Endpoints | 100 |
| 14.3.3. | Exploratory Endpoints | 100 |
| 14.4. | Analysis Populations | 101 |
| 14.5. | Subject Characteristics and Disposition | 101 |
| 14.6. | Safety Assessment | 102 |
| 14.7. | Efficacy Assessment | 103 |
| 14.8. | Pharmacokinetic Analysis | 104 |
| 14.9. | Immunogenicity Assays. | 104 |
| 15. | DIRECT ACCESS TO SOURCE DATA/NOTES | 105 |
| 16. | QUALITY CONTROL AND QUALITY ASSURANCE | 106 |
| 16.1. | Conduct of the Study | 106 |
| 16.2. | Study Monitoring | 106 |
| 17. | ETHICS | 108 |
| 17.1. | Institutional Review Board/Independent Ethics Committee | 108 |
| 17.2. | Good Clinical Practice | 108 |
| 17.3. | Written Informed Consent | 108 |
| 17.4. | Protocol Approval and Amendment(s) | 109 |
| 17.5. | Subject Confidentiality | 109 |
| 18 | DATA HANDI ING AND RECORD KEEPING | 100 |

| 18.1. | Case Report Forms/Source Data Handling | 109 |
|---|---|---|
| 18.2. | Retention of Essential Documents | 110 |
| 18.3. | Principal Investigator's Record Requirements | 110 |
| 19. | PUBLICATION POLICY | 111 |
| 20. | LIST OF REFERENCES | 112 |
| APPENDI | X A. RECIST GUIDELINES | 117 |
| APPENDI | X B. ECOG PERFORMANCE SCALE | 120 |
| APPENDI | X C. PROPHYLAXIS AND MANAGEMENT OF NAUSEA AND VOMITING AND HYPERSENSITIVITY REACTIONS, CYTOKINE RELEASE SYNDROME, AND NEUROLOGICAL TOXICITY | 121 |
| APPENDI | X D. DOSE MODIFICATION AND TOXICITY MANAGEMENT FOR IMMUNE-RELATED ADVERSE EVENTS | 130 |
| APPENDI | X E. NATIONAL COMPREHENSIVE CANCER NETWORK AND AMERICAN SOCIETY OF CLINICAL ONCOLOGY: MANAGEMENT OF IMMUNOTHERAPY-RELATED TOXICITIES (IMMUNE CHECKPOINT INHIBITOR-RELATED TOXICITIES) | 133 |
| Table 1: | LIST OF TABLES Mean Results of Noncompartmental Analysis of XmAm18087 after Multiple IV Dose Administration in Cynomolgus Monkey (Good Laboratory Practice) | 34 |
| Table 2: | Part A (MCC) Monotherapy Safety Run-in and Expansion Cohorts | 46 |
| Table 3: | Part B (MCC) Combination Therapy Safety Run-in and Expansion Cohorts | 47 |
| Table 4: | Part C (SCLC) Monotherapy Safety Run-in and Expansion Cohorts | 48 |
| Table 5: | Boundaries for AESC Incidence: Cohort A | 53 |
| Table 6: | Boundaries for AESC Incidence: Cohorts B and C | 53 |
| Table 7: | Schedule of Assessments | 54 |
| Table 8: | Severity Grading Scale | 81 |
| Table 9: | Causality Grading Scale | 82 |
| Table 10: | American Society for Transplantation and Cellular Therapy Cytokine<br>Release Syndrome Consensus Grading | 87 |
| Table 11: | Immune Effector Cell-associated Encephalopathy Scoring | 92 |
| Table 12: | American Society for Transplantation and Cellular Therapy Immune<br>Effector Cell-associated Neurotoxicity Syndrome Consensus Toxicity | 03 |

| Table 13: | Assessment of Overall Response in Subjects with Target (± Nontarget Disease) | 119 |
|---|---|---|
| Table 14: | ECOG Performance Scale | 120 |
| Table 15. | American Society for Transplantation and Cellular Therapy Cytokine<br>Release Syndrome Consensus Grading | 122 |
| Table 16: | Immune Effector Cell-associated Encephalopathy Scoring | 127 |
| Table 17: | American Society for Transplantation and Cellular Therapy Immune<br>Effector Cell-associated Neurotoxicity Syndrome Consensus Toxicity<br>Grading for Adults | 128 |
| Table 18: | Dose Modification and Toxicity Management Guidelines for Immune-Related Adverse Events in Patients Receiving Pembrolizumab | 131 |
| | LIST OF FIGURES | |
| Figure 1. | Molecular Domain Format of XmAb18087 | 30 |
| Figure 2. | Antitumor Activity in a Mouse Xenograft Model | 32 |
| Figure 3. | XmAb18087 Mean Serum Concentration Versus Time in Cynomolgus<br>Monkeys (Good Laboratory Practice) | 33 |
| Figure 4: | Study Design | 42 |
| Figure 5: | Part A and Part C: XmAb18087 Monotherapy Treatment | 44 |
| Figure 6: | Part B: XmAb18087/Pembrolizumab Combination Therapy Treatment | 44 |


# 4. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| ADA | anti-drug antibody |
|---|---|
| AE(s) | adverse event(s) |
| AESC | adverse event of specific concern |
| AI | accumulation index |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| ASTCT | American Society for Transplantation and Cellular Therapy |
| $AUC_{0-\infty}$ | area under the serum concentration-time curve from time zero to infinity |
| AUC <sub>0-7</sub> | area under the serum concentration-time curve from time zero to seven days postdose |
| AUCt | area under the serum concentration-time curve during a dosing interval (t) |
| β-hCG | beta human chorionic gonadotropin |
| bpm | beats per minute |
| bsAb | bispecific antibody |
| CAR-T | chimeric antigen receptor T cell |
| CBC | complete blood count |
| CFR | Code of Federal Regulations |
| CL | Clearance |
| C <sub>max</sub> | maximum observed serum concentration |
| $C_{min,ss}$ | minimum steady-state concentration |
| $C_{min[trough]}$ | predose or trough concentration |
| $C_{ss}$ | steady-state concentration |
| $C_{trough}$ | trough concentration at predose |
| CR | complete response |
| CRF | case report form |
| CRS | cytokine release syndrome |
| СТ | computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DERC | Dose Escalation Review Committee |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EOI | end of infusion |
| EOS | end of study |


| Fab antigen-binding fragment of an antibody FACS fluorescence-activated cell sorting Fc fragment, crystallizable FcyR Fc gamma receptor FDA US Food and Drug Administration FFPE formalin-fixed paraffin embedded FIH first-in-human FSH follicle-stimulating hormone GCP good clinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HBAIC glycated hemoglobin HBV hepatitis B virus HICV hepatitis C virus HIV human immunodeficiency virus HIR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-\(\gamma\) interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IHC International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IFN-\(\gamma\) interferon-gamma Ig immunoglobulin E IHC International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IHC I | ЕОТ | end of treatment |
|---|---|---|
| Fe fragment, crystallizable FeyR Fe gamma receptor FDA US Food and Drug Administration FFPE formalin-fixed paraffin embedded FIH first-in-human FSH follicle-stimulating hormone GCP good clinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GI.P good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HbA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IFN-7 interferon-gamma Ig immunoglobulin E IHC Inmunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | Fab | antigen-binding fragment of an antibody |
| FeyR Fe gamma receptor FDA US Food and Drug Administration FFPE formalin-fixed paraffin embedded FIH first-in-human FSH follicle-stimulating hormone GCP good clinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HBAIC glycated hemoglobin HBV hepatitis B virus HIV human immunodeficiency virus HIR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IFN-\(\gamma\) interferon-gamma Ig immunoglobulin IgE immunoglobulin E HIC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | FACS | fluorescence-activated cell sorting |
| FDA US Food and Drug Administration FFPE formalin-fixed paraffin embedded FIH first-in-human FSH follicle-stimulating hormone GCP good clinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HBAIC glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IFN-\(\gamma\) interferon-gamma Ig immunoglobulin IgE immunoglobulin E HIC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | Fc | fragment, crystallizable |
| FFPE formalin-fixed paraffin embedded FIH first-in-human FSH follicle-stimulating hormone GCP good elinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HBAIC glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-y interferon-gamma Ig immunoglobulin IgE immunoglobulin E HC Immunolistochemistry IL Interleukin IMP(s) investigational New Drug Application IRAE immune-related adverse event | FcγR | Fc gamma receptor |
| FIII first-in-human FSH follicle-stimulating hormone GCP good clinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HbA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-\gamma immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational New Drug Application IRAE immune-related adverse event | FDA | US Food and Drug Administration |
| FSH follicle-stimulating hormone GCP good clinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HBAIC glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-\(\gamma\) interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | FFPE | formalin-fixed paraffin embedded |
| GCP good clinical practice GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HbA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-\gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunobistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immunoglobulin immunoglobulin immunoglobulin immunoglobulin imvestigational New Drug Application IRAE immunoglobulin immune-related adverse event | FIH | first-in-human |
| GGT gamma glutamyl transferase GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HbA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-\gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | FSH | follicle-stimulating hormone |
| GIST gastrointestinal stromal tumor GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HBA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-y interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | GCP | good clinical practice |
| GLP good laboratory practice HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HbA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-\(\gamma\) interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immuno-related adverse event | GGT | gamma glutamyl transferase |
| HBcAb hepatitis B core antibody HBsAg hepatitis B surface antigen HbA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-y interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | GIST | gastrointestinal stromal tumor |
| HBsAg hepatitis B surface antigen HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | GLP | good laboratory practice |
| HbA1C glycated hemoglobin HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-\gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | HBcAb | hepatitis B core antibody |
| HBV hepatitis B virus HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | HBsAg | hepatitis B surface antigen |
| HCV hepatitis C virus HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | HbA1C | glycated hemoglobin |
| HIV human immunodeficiency virus HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | HBV | hepatitis B virus |
| HR heart rate FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | HCV | hepatitis C virus |
| FSH follicle-stimulating hormone ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Inmunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | HIV | human immunodeficiency virus |
| ICANS immune effector cell-associated neurotoxicity syndrome ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | HR | heart rate |
| ICE Immune Effector Cell-Associated Encephalopathy ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | FSH | follicle-stimulating hormone |
| ICF informed consent from ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | ICANS | immune effector cell-associated neurotoxicity syndrome |
| ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | ICE | Immune Effector Cell-Associated Encephalopathy |
| Human Use IEC Independent Ethics Committee IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | ICF | informed consent from |
| IFN-γ interferon-gamma Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | ICH | |
| Ig immunoglobulin IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | IEC | Independent Ethics Committee |
| IgE immunoglobulin E IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | IFN-γ | interferon-gamma |
| IHC Immunohistochemistry IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | Ig | immunoglobulin |
| IL Interleukin IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | IgE | immunoglobulin E |
| IMP(s) investigational medicinal product(s) IND Investigational New Drug Application IRAE immune-related adverse event | IHC | Immunohistochemistry |
| IND Investigational New Drug Application IRAE immune-related adverse event | IL | Interleukin |
| IRAE immune-related adverse event | IMP(s) | investigational medicinal product(s) |
| | IND | Investigational New Drug Application |
| IRB Institutional Review Board | IRAE | immune-related adverse event |
| | IRB | Institutional Review Board |


| IUD | intrauterine device |
|---------|----------------------------------------------|
| IV | Intravenous |
| mAb | monoclonal antibody |
| MCC | Merkel cell carcinoma |
| MCPyV | Merkel cell polyomavirus |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMSE | Mini-mental State Examination |
| MRI | magnetic resonance imaging |
| MTD | maximum tolerated dose |
| NCCN | National Comprehensive Cancer Network |
| NCI | US National Cancer Institute |
| NET(s) | neuroendocrine tumor(s) |
| NETSPOT | Ga-68 DOTATATE PET gallium scanning |
| NOAEL | no-observed-adverse-effect-level |
| ORR | overall response rate |
| OS | overall survival |
| PBMC | peripheral blood mononuclear cells |
| PBS | phosphate-buffered saline |
| PD | pharmacodynamics; progressive disease |
| PD1 | programmed cell death protein 1 |
| PDL1 | programmed cell death ligand 1 |
| PDL2 | programmed cell death ligand 2 |
| PE | physical examination |
| PET | positron emission tomography |
| PFS | progression-free survival |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PO | Orally |
| PR | partial response |
| Q6W | every 6 weeks |
| RBC | red blood cell |
| RD | recommended dose |
| RedFlu | red fluorescent protein |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE(s) | serious adverse event(s) |


| CAD | |
|---|---|
| SAP | statistical analysis plan |
| scFv | single-chain variable fragment (immunoglobulin fusion protein) |
| SCLC | small cell lung cancer |
| SOC | System Organ Class |
| SOP(s) | standard operating procedure(s) |
| SRC | Safety Review Committee |
| SST | Somatostatin |
| SSTR | somatostatin receptor |
| t <sub>1/2</sub> | half-life |
| TEAE(s) | treatment-emergent AE(s) |
| TESAE(s) | treatment-emergent SAE(s) |
| TNF-α | tumor necrosis factor $\alpha$ |
| t <sub>max</sub> | time to reach maximum concentration |
| t <sub>min</sub> | time of minimum concentration |
| ULN | upper limit of normal |
| US | United States |
| UV | Ultraviolet |
| Vd | volume of distribution |
| Vd <sub>ss</sub> , V <sub>ss</sub> | steady-state volume of distribution |
| WBC | white blood cell |
| %Fluct | steady-state fluctuation in concentrations |


## 5. INTRODUCTION

## 5.1. Background

## 5.1.1. Somatostatin and Somatostatin Receptors

Somatostatin (SST), a peptide hormone that is secreted by endocrine and other cells throughout the body, has largely inhibitory effects that are mediated through 5 SST receptor (SSTR) subtypes (1-5). The specific effects of SSTR subtypes are largely due to different distributions and levels of expression within tissues (Barbieri, 2013). SSTR2 is widely expressed in normal tissues and upregulated in many types of tumors (Bronstein-Sitton, 2006; Taniyama, 2005). Like other neuroendocrine tumors, a high proportion of Merkel cell carcinomas (MCC) possesses receptors for somatostatin. In one series of 105 MCC tissue samples from 98 patients, SSTR2a and SSTR5 were expressed in 58 cases (59.2%) and 44 cases (44.9%), respectively. Overall, at least one SSTR subtype was expressed in 75 tumors (76.5%). Expression of SSTR2A, but not SSTR5, was associated with Merkel cell polyomavirus (MCPyV) positivity (Gardair, 2015).

Small cell lung cancer (SCLC), like MCC, often expresses SSTR2, with expression detected by immunohistochemistry (IHC) in patient tumor samples at varying frequencies. Among three different studies, SSTR2 IHC positivity was reported in 11/18 cases (61%; Reubi, 2000), 6/19 cases (32%; Lapa, 2016), and 47/98 cases (48%; Lehman, 2019).

These receptors can also be demonstrated in vivo in both MCC and SCLC by somatostatin receptor-based diagnostic imaging techniques, such as indium-111 pentetreotide single-photon emission computed tomography (SPECT; OctreoScan) or Ga-68 DOTATATE positron emission tomography (PET) gallium scanning (NETSPOT) (Kritikos, 2015; Epstude, 2013; Reisinger, 1998; Lapa, 2016; NETSPOT Package Insert, 2018).

Small series and some case reports have demonstrated success with therapeutic targeting of the SSTR in patients with MCC. This includes radionuclide therapy with yttrium-90-DOTATOC (a somatostatin analog containing the active octapeptide of somatostatin (Meier, 2004); peptide receptor radionuclide therapy with lutetium-177 isotope (Salavati, 2012), the somatostatin analogs lanreotide and octreotide (di Bartolomeo, 1996). Somatostatin analog therapy has also been tested in a limited number of SCLC patients with mixed results (Tartarone, 2016).

## 5.1.2. Merkel Cell Carcinoma

MCC is a rare, aggressive cutaneous malignancy that predominantly affects older adults and is more common in Caucasians compared with other ethnicities. Risk factors for the disease include ultraviolet exposure and advancing age. Immunosuppression, such as that associated with organ transplant, lymphoproliferative malignancies, or HIV, is also a risk factor for the diagnosis.

The tumor has a propensity for local recurrence and early regional lymph node metastasis. In 2013, the MCC incidence rate was 0.7 cases per 100,000 person-years, corresponding to 2488 cases per year. The incidence increased exponentially with age, from 0.1 to 1.0 to 9.8 (per 100,000 person-years) among age groups 40 to 44 years, 60 to 64 years, and  $\geq$  85 years, respectively (Paulson, 2018).


MCC pathogenesis is associated with either the presence of MCPyV or chronic exposure to ultraviolet light (UV), which can cause a characteristic pattern of multiple DNA mutations. In areas with high UV exposure, UV-mediated carcinogenesis is predominant; by contrast, in areas with lower UV exposure, the majority of MCC cases are of viral etiology. The 2 etiologies share similar clinical, histopathological, and prognostic characteristics. Ultraviolet light exposure is suspected to be involved in viral-mediated and non-viral-mediated carcinogenesis, by contributing to immunosuppression or DNA damage, respectively (Becker, 2017).

Approximately 30% of patients have locoregional metastases at the time of initial diagnosis. In an analysis of over 9000 MCC cases from the National Cancer Database between 1998 and 2012, patients presented with local disease in 65% of cases, while 26% had regional lymph node involvement and 8% had distant metastases (Harms, 2016).

Excision of the primary tumor is the first-line therapy for locoregional disease, and surgery is frequently combined with radiation therapy to improve locoregional control. However, recurrences of MCC are frequent, even after definitive local and regional therapy, and are associated with a relatively poor prognosis (Eng, 2004).

In general, the management of patients with distant metastases must be individually tailored. While systemic therapy and radiation therapy have until recently been the primary treatment options, surgery may be beneficial in highly selective circumstances for resection of oligometastasis or symptomatic lesions (NCCN Guidelines, 2019).

Until recently, systemic therapy for metastatic MCC consisted of various regimens of cytotoxic chemotherapy, but these treatments have been met with limited success. While a response rate of 55% was observed to a first-line chemotherapeutic regimen (most commonly platinum plus etoposide), the responses were typically not durable, and the median progression-free survival (PFS) was only 3 months (Iyer, 2016; NCCN Guidelines, 2019).

In contrast, immunotherapy with checkpoint inhibitors has shown promise in treating metastatic MCC. Avelumab, an anti-programmed cell death ligand 1 (PDL1)-targeted monoclonal antibody, is approved in the United States to treat patients with metastatic MCC, irrespective of prior therapy. In the JAVELIN Merkel 200 trial, Part A, 88 patients who had received prior cytotoxic chemotherapy were treated with avelumab. With a median follow-up of 2 years, there was a 33% overall response rate (ORR), including 10 complete responses (Kaufman, 2016; Kaufman, 2018; Nghiem, 2018). The 2-year PFS rate was 26%, and the 2-year overall survival rate was 36%. In addition, 2 anti-programmed cell death protein 1 (PD1) monoclonal antibodies, pembrolizumab and nivolumab, have shown evidence of activity in patients with metastatic MCC (Nghiem, 2019; Topalian, 2017).

There are no FDA approved therapies or standard treatments if anti PD1 or anti PDL1 checkpoint inhibitor therapy fails. MCC is an aggressive tumor with high rates of locoregional recurrence and metastatic spread; thus, development of novel therapeutic agents is a significant unmet medical need. XmAb18087 is a bispecific antibody that simultaneously targets a highly expressed somatostatin receptor and CD3, a T cell identifier, bringing together tumor cells and immune effector cells with the idea of activating the immune system to kill tumor cells. Given the medical need and the previous success of immunotherapy in this indication, XmAb18087 should be investigated for treatment of MCC.


## 5.1.3. Small Cell Lung Cancer

Small cell lung cancer shares several biological and clinical characteristics with MCC that warrant the investigation of XmAb18087 in this indication as well, including SSTR2 expression, responsiveness to immunotherapy, rapid progression, and poor prognosis. Accounting for 15% of all lung cancers, SCLC is, like MCC, a high-grade neuroendocrine tumor with poor clinical outcome. The estimated yearly incidence of small cell lung cancer in 2017 was approximately 30,000 cases in the United States; almost all cases are associated with a history of cigarette smoking (NCCN Guidelines, 2018).

Around 70% of patients with SCLC present with extensive stage, metastatic disease, for which treatment options are palliative. The standard of care for extensive stage SCLC remains combination chemotherapy with various regimens, with a platinum agent plus etoposide being the most commonly used (NCCN Guidelines, 2018, Früh, 2013). Most patients initially benefit from chemotherapy, with response rates of 60 to 70%, but then quickly relapse; the median PFS in this patient population is less than 6 months (Früh, 2013).

Recently, immune checkpoint inhibitors have shown activity in SCLC. Atezolizumab and durvalumab each received FDA approval in combination with chemotherapy for first line treatment of extensive stage SCLC; pembrolizumab and nivolumab are each approved in the US as single agents in the third-line setting. Still, improvements in clinical outcomes have been modest. For example, in the IMpower133 trial, patients who received atezolizumab plus chemotherapy had a median PFS of 5.2 months, compared to 4.3 months for those receiving chemotherapy alone (Horn, 2018). Thus, despite recent advances in the field, there remains a substantial need for better treatment options for extensive-stage SCLC. This high unmet clinical need coupled with the biological features of SCLC warrant investigation of XmAb18087 in this indication.

## **5.1.4.** Therapeutic Bispecific Antibodies

The concept of recombinant antibodies that would allow for simultaneous engagement with 2 targets was first developed in the late 1990s. Bispecific antibodies (bsAbs), it was theorized, could potentially increase binding specificity, providing simultaneous dual activation or blockade of 2 disease mediators, or in the case of cancer therapy, simultaneous binding of cytotoxic T cells and tumor antigens, thus promoting T-cell activation and killing of tumor cells. Although technical obstacles in production initially slowed development of bsAbs, recent advances in protein biology and recombinant expression techniques have resulted in several more easily producible formats for bsAbs, each of which has different properties (Spiess, 2015). While small format bispecific constructs are rapidly excreted and have short half-lives that require continuous infusion for maintenance of efficacious concentrations, XmAb18087 is built on a construct that includes a full fragment, crystallizable (Fc) region, which is designed to yield pharmacokinetics (PK) similar to humanized antibodies and should allow intermittent administration on a weekly or biweekly schedule (Przepiorka, 2015).

## 5.1.5. XmAb18087 Product Description

XmAb18087 is a humanized bsAb that binds both the tumor antigen SSTR2 and CD3 antigen to recruit cytotoxic T cells for killing of SSTR2<sup>+</sup> tumor cells.




Figure 1. Molecular Domain Format of XmAb18087



Fc = fragment, crystallizable; scFv = single-chain variable fragment (immunoglobulin fusion protein); SSTR = somatostatin receptor.

### **5.1.6.** Preclinical Studies

## 5.1.6.1. Pharmacology

XmAb18087 is a humanized and affinity-optimized bsAb that engages both SSTR2 on tumor cells as well as CD3 on T cells to recruit cytotoxic T cells to kill SSTR2<sup>+</sup> tumor cells. XmAb18087 has been designed to maintain full-length humanized monospecific antibody properties in a bispecific antibody, thus enabling the design of stable molecules with favorable in vivo half-life and allowing for standard antibody production methods.

In preclinical in vitro studies, XmAb18087 stimulated robust redirected T-cell-mediated cytotoxicity against SSTR2<sup>+</sup> cell lines





Xencor, Inc **CONFIDENTIAL** 18 August 2020 Protocol XmAb18087-02

Figure 2. **Antitumor Activity in a Mouse Xenograft Model** 





huPBMCs = human peripheral blood mononuclear cells; NSG = NOD SCID gamma; PBS = phosphate-buffered saline; FLuc = Firefly Luciferase.

On Study Day 0, young NSG mice received a subcutaneous injection of 1x106 A549 Red-FLuc cells from a human non-small cell lung tumor cell line that had been modified to express a red-shifted luciferase transgene for in vivo imaging. Seven days later, mice were engrafted intraperitoneally with 10 × 106 huPBMCs and treated with either vehicle (PBS), or 0.03, 0.1, 0.3, or 1.0 mg/kg of XmAb18087 once a week for 3 consecutive weeks. (A) Tumor burden was monitored by in vivo imaging using total flux (p/s) captured by In Vivo Imaging System. (B) Tumor volumes were determined using physical caliper measurements.




In summary, the results in human cells, in human xenograft in mice, and in cynomolgus monkeys indicate activity of XmAb18087 against SSTR2<sup>+</sup> cells and supports clinical assessment of XmAb18087 in SSTR2<sup>+</sup> cancers, including neuroendocrine tumors (NET) and gastrointestinal stromal tumor (GIST.)

## **5.1.6.2.** Pharmacokinetics and Toxicokinetics



Figure 3. XmAb18087 Mean Serum Concentration Versus Time in Cynomolgus Monkeys (Good Laboratory Practice)



The mean results of a noncompartmental analysis of this study are shown in Table 1.




# 5.1.6.3. Toxicology

The toxicology of XmAb18087 was also explored in this GLP toxicology study and in 3 non-GLP pharmacology studies.

In the GLP toxicology study,

All doses and regimens of XmAb18087 were well tolerated, with no observed effects on food consumption, electrocardiography, body temperature, ophthalmic examinations, or urinalysis







## 5.1.7. Human Experience with XmAb18087 and Related Molecules

Two bsAb products have previously been approved by FDA. In 2014, accelerated approval was granted to blinatumomab (Blincyto® PI, 2018) for the treatment of Philadelphia chromosome-negative, relapsed or refractory precursor B-cell acute lymphoblastic leukemia (Przepiorka, 2015). It has since also received approval for treatment of relapsed or refractory B-cell precursor acute lymphoblastic leukemia. Blinatumomab is an anti-CD19/anti-CD3 bsAb, constructed as a small-format recombinant protein that, due to its small size, is rapidly cleared and given as a continuous infusion. Cytokine release syndrome and neurologic events were the drug's primary toxicities (Spiess, 2015). In 2017, approval was granted to emicizumab-kxwh (Hemlibra), a bispecific factor IXa- and factor X-directed antibody for prophylaxis to prevent or reduce the frequency of bleeding episodes in adult and pediatric patients with hemophilia A. Emicizumab-kxwh is administered by subcutaneous injection. In contrast to blinatumomab, emicizumab-kxwh is not designed to engage T-cells; thus, cytokine release syndrome is not a significant risk with this drug (HEMLIBRA® Package Insert, 2018).

Although the receptor target of XmAb18087 and its distribution are different from those of blinatumomab, the 2 drugs' common mechanism of T-cell engagement and redirection, in addition to the results of Xencor's toxicology studies with XmAb18087 and the company's experience with 2 other CD3-directed bsAb products now in the clinic, indicate that CRS is expected to be a toxicity of the drug, principally after the first dose.

The first-in-human (FIH) Phase 1 clinical study of XmAb18087 in advanced low to intermediate grade NETs and advanced GISTs (XmAb18087-01) has thus far borne out this expectation, with mostly low-grade CRS events being observed. The maximum tolerated dose (MTD)-determining toxicities in the NET arm of the trial were nausea and vomiting. The trial now includes a CRS prophylactic regimen and an antiemetic prophylactic regimen for at least the first these prophylactic regimens decreased the incidence of CRS and the incidence and severity of nausea and vomiting. See also Section 5.3.

## 5.2. Pembrolizumab

Pembrolizumab (MK-3475; Keytruda<sup>®</sup>) is a potent humanized immunoglobulin G4 monoclonal antibody (mAb) with high specificity of binding to the PD1 receptor, thus inhibiting its interaction with PDL1 and programmed cell death ligand 2 (PDL2). Pembrolizumab has high affinity and potent receptor blocking activity for PD1. Pembrolizumab is in clinical development as an IV immunotherapy for advanced malignancies. Pembrolizumab is indicated for the treatment of patients across several indications, including MCC. For more details on these specific indications, refer to the approved product labeling for detailed background information (Keytruda<sup>®</sup> Package Insert, 2020).

The clinical responses to pembrolizumab highlight the utility of immunotherapeutic agents for treating cancer. However, some patients either fail to respond to pembrolizumab or relapse after an initial response. Such patients could potentially benefit from the addition of an additional immune-targeted agent with a distinct mechanism of action. This general rationale has spurred the investigation of several T-cell bispecific antibodies in combination with anti-PD1 agents, and supports the proposed combination of XmAb18087 with pembrolizumab in MCC, an indication for which the latter is already FDA-approved (Kobold, 2018; Keytruda® Package Insert, 2020).

#### 5.2.1. Pharmaceutical and Therapeutic Background

The importance of intact immune surveillance function in controlling outgrowth of neoplastic transformations has been known for decades (Disis, 2010). Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T cells and the ratio of CD8+ effector T cells/FoxP3+ regulatory T cells correlates with improved prognosis and long-term survival in solid malignancies, such as ovarian, colorectal, and pancreatic cancer; hepatocellular carcinoma; malignant melanoma; and renal cell carcinoma. Tumor-infiltrating lymphocytes can be expanded ex vivo and reinfused, inducing durable objective tumor responses in cancers such as melanoma (Dudley, 2005; Hunder, 2008).

The PD1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD1, expressed on the cell surface of activated T cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD1 (encoded by the gene *Pdcd1*) is an immunoglobulin (Ig) superfamily member related to CD28 and CTLA4 that has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PDL1 and/or PDL2; Greenwald, 2005; Okazaki, 2001).

The structure of murine PD1 has been resolved (Zhang, 2004). PD1 and its family members are type I transmembrane glycoproteins containing an Ig-variable—type domain responsible for ligand binding and a cytoplasmic tail responsible for the binding of signaling molecules. The cytoplasmic


tail of PD1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif, and an immunoreceptor tyrosine-based switch motif. Following T-cell stimulation, PD1 recruits the tyrosine phosphatases, SHP-1 and SHP-2, to the immunoreceptor tyrosine-based switch motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3 zeta (CD3 $\zeta$ ), protein kinase C-theta (PKC $\theta$ ), and zeta-chain-associated protein kinase (ZAP70), which are involved in the CD3 T-cell signaling cascade (Okazaki, 2001; Chemnitz, 2004; Sheppard, 2004; Riley, 2009). As a consequence, the PD1/PDL1 pathway is an attractive target for therapeutic intervention in a number of neoplastic diseases.

#### **5.2.2.** Nonclinical Studies

Therapeutic studies in mouse models have shown that administration of antibodies blocking PD1/PDL1 interaction enhances infiltration of tumor-specific CD8+ T cells and ultimately leads to tumor rejection, either as a monotherapy or in combination with other treatment modalities (Blank, 2004; Curran, 2010; Hirano, 2005; Pilon-Thomas, 2010; Strome, 2003; Spranger, 2014; Weber, 2010). Antimouse PD1 or antimouse PDL1 antibodies have demonstrated antitumor responses in models of squamous cell carcinoma, pancreatic carcinoma, melanoma, acute myeloid leukemia, and colorectal carcinoma (Curran, 2010; Nomi, 2007; Pilon-Thomas, 2010; Strome, 2003; Zhang, 2004). In such studies, tumor infiltration by CD8+ T cells and increased IFN-γ, granzyme B, and perforin expression were observed, indicating that the mechanism underlying the antitumor activity of PD1 checkpoint inhibition involved local infiltration and activation of effector T-cell function in vivo (Curran, 2010). Experiments have confirmed the in vivo efficacy of antimouse PD1 antibody as a monotherapy, as well as in combination with chemotherapy, in syngeneic mouse tumor models.

#### 5.2.3. Justification for Pembrolizumah Dose

The planned dose of pembrolizumab for this study is 400 mg every 6 weeks (Q6W), which is a current FDA-approved dose for adults with recurrent locally advanced or metastatic MCC (Keytruda® Package Insert, 2020).

# 5.3. Rationale for Dose Selection of XmAb18087-01 FIH, XmAb18087-02, and Study Design







#### 6. STUDY OBJECTIVES

## 6.1. Primary Objectives

The primary objectives of the study are as follows:

- 1. To determine the safety and efficacy (by ORR, complete response [CR], and partial response [PR] per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) of XmAb18087 monotherapy in subjects with advanced MCC that has progressed after treatment with standard therapies
- 2. To determine the safety and efficacy (by ORR, CR, and PR per RECIST 1.1 criteria) of XmAb18087 in combination with pembrolizumab in subjects with advanced MCC who have not received prior anti-PD1 or anti-PDL1 therapies, and for whom pembrolizumab as a single agent is indicated
- 3. To determine the safety and efficacy (by ORR, CR, and PR per RECIST 1.1 criteria) of XmAb18087 monotherapy in subjects with extensive-stage SCLC that has progressed after treatment with standard therapies

## 6.2. Secondary Objectives

The secondary objectives of the study are as follows:

- 1. To assess antitumor activity of XmAb18087 by PFS per RECIST 1.1 criteria, as well as overall survival (OS) and duration of response, when administered with and without pembrolizumab in subjects with advanced MCC, and as monotherapy in subjects with extensive-stage SCLC
- 2. To characterize the PK and immunogenicity of XmAb18087 administered with and without pembrolizumab in subjects with advanced MCC, and as monotherapy in subjects with extensive-stage SCLC
- 3. To assess the PK profile ( $C_{max}$  and trough concentration,  $C_{min[trough]}$ ) of pembrolizumab when co-administered with XmAb18087

# 6.3. Exploratory Objectives

The exploratory objectives of the study are as follows:

- 1. To assess the incidence, timing, and severity of CRS by the following:
  - a. CRS-related AEs (incidence and grade of AEs and incidence of serious adverse events [SAEs])
  - b. Biomarkers of CRS
- 2. To characterize the biological activity associated with administration of XmAb18087 with and without pembrolizumab by assessment of cell surface markers on selected immune system cells in peripheral blood, including changes in lymphocyte subsets and in T-cell activation/exhaustion by flow cytometry and similar bioanalytical methods


- 3. To characterize PD by correlation of clinical response with NETSPOT® (gallium 68 dotatate) positron emission tomography/computed tomography (PET/CT) scan results after XmAb18087 administration with and without pembrolizumab
- 4. To evaluate by immunohistochemistry tumor-cell expression of SSTR2 and PDL1 and tumor-infiltrating T cells expression of proliferation markers and PD1/PDL1 after XmAb18087 administration with and without pembrolizumab, as well as changes in other immune cell subsets
- 5. To characterize the pharmacodynamic (PD) changes in the intratumoral inflammatory response using immunostaining of immune cells and analysis of RNA signatures
- 6. To correlate clinical response in MCC subjects to MCPyV status as determined by serology and immunohistochemistry


#### 7. INVESTIGATIONAL PLAN

## 7.1. Overall Study Design and Plan

This is a Phase 1b/2, multiple-dose study of XmAb18087, both as a monotherapy and in combination with pembrolizumab in MCC subjects, and as monotherapy only in SCLC subjects. The study is designed in 3 parts, Part A, Part B, and Part C shown in Figure 4.

Figure 4: Study Design



MCC = Merkel cell carcinoma; PD1 = programmed cell death protein 1; PDL1 = programmed cell death ligand 1; SCLC = small cell lung cancer.

**Part A** is designed to describe safety and efficacy, and to assess PK and immunogenicity of XmAb18087 monotherapy in subjects with advanced MCC. All eligible subjects will have relapsed or refractory disease that has previously been treated with all standard therapies for which they are eligible.

Part A will enroll safety run-in cohorts to confirm the safety and tolerability of XmAb18087 monotherapy administered IV with weekly step-up dosing for 42-day cycles. Additional subjects will then be enrolled into an expansion cohort and will receive XmAb18087 monotherapy using the recommended dose (RD) identified following the safety run-in cohorts.

**Part B** is designed to describe safety and efficacy, and to assess PK and immunogenicity of XmAb18087 in combination with pembrolizumab in subjects with advanced MCC. All eligible subjects may be treatment naïve or have relapsed or refractory disease after prior treatment; however, subjects who have received prior treatment with anti-PD1 or anti-PDL1 therapeutics will not be eligible to participate in Part B.

Part B will enroll additional safety run-in cohorts to confirm the safety and tolerability of XmAb18087 in combination with pembrolizumab. Subjects will receive step-up IV dosing of XmAb18087 (except for Cohort 1B, in which subjects will receive the same dose level on each


dosing day) on Days 1, 8, 22, 29, and 36, and IV dosing of pembrolizumab on Day 15 of each 42-day cycle. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 plus pembrolizumab combination therapy using the RD identified following the safety run-in.

Enrollment into Part B safety run-in cohorts (starting with Cohort 1B) may begin after the first safety run-in cohort in Part A (Cohort 1A, one dose level higher than Cohort 1B) has completed the first cycle and the regimen has been demonstrated to be tolerable.

**Part** C is designed to describe safety and efficacy, and to assess PK and immunogenicity of XmAb18087 monotherapy in subjects with extensive-stage SCLC. All eligible subjects will have relapsed or refractory disease that has previously been treated with all standard therapies for which they are eligible.

Part C of the study will enroll additional safety run-in cohorts to confirm the safety and tolerability of XmAb18087 monotherapy in this indication. The safety run-in will follow the same cohort schema as described for Part A to identify a RD for expansion in SCLC. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 monotherapy using the RD identified following the safety run-in.

Enrollment into Part C may begin concurrently with Part A.

**Part A, Part B, and Part C:** The decision to advance to higher dose levels after each safety run-in cohort will be made by an SRC based on review of the aggregate safety data for all subjects in that cohort as well as cumulative safety data for the study overall. The SRC will be allowed to make adaptations to the dosing schema, if needed, in accordance with evolving trial safety and tolerability findings, as long as adaptations do not significantly increase subject risk. Any such adaptations would require a protocol amendment and IRB approval.

In each safety run-in cohort, no more than 1 subject will receive the first infusion of XmAb18087 on any given day.

Subjects may be admitted and monitored on Day -1 (hospitalization is optional), and will be admitted on study days 1, 2, and 3 for their first dose of XmAb18087 and for at least 48 hours following the second dose. In addition, any subject who has shown symptoms of CRS during inpatient admission will continue to be monitored as an inpatient for at least 24 hours after the symptoms have subsided.

The Schedules of Assessments is provided in Section 7.9, Table 7.


## 7.2. Study Flowcharts

Figure 5 shows the dosing schedule for each 42-day cycle in the Part A and Part C monotherapy portions of the trial, while Figure 6 shows Part B combination therapy portions of the trial. Inpatient stays are only required in Cycle 1.

Figure 5: Part A and Part C: XmAb18087 Monotherapy Treatment



Figure 6: Part B: XmAb18087/Pembrolizumab Combination Therapy Treatment



# 7.3. Dosing Schedule

Each subject will be administered XmAb18087 IV at a constant infusion rate over


The initial treatment period for each subject in this study is 1 cycle. Each cycle is 42 days long. In Part A and Part C, each cycle will consist of 6 weekly doses of XmAb18087 (on Days 1, 8, 15, 22, 29, and 36).

In Part B, each cycle will consist of 5 XmAb18087 doses on Days 1, 8, 22, 29, and 36. Pembrolizumab will be administered as 1 dose during each 42-day cycle, on Day 15.

Part A dose levels are defined in Table 2. Part B dose levels are defined in Table 3. Part C dose levels are defined in Table 4.

The dose is based on the subject's actual baseline weight measurement in kilograms (rounded to the nearest integer) on Day -1. Following the first dose at any dose level, the weight used for calculation of subsequent doses will be modified only if the subject's weight changes by more than 10% from the baseline weight, at which point the dose will be recalculated using the current weight (rounded to the nearest integer).


Table 2: Part A (MCC) Monotherapy Safety Run-in and Expansion Cohorts

| | | | | | Cycle | e 1 | | | | | | Cycle | 2+ | | | Subjects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cycle<br>and Day | D1 | D8 | D15 | D22 | D29 | D36 | D40 | D1 | D8 | D15 | D22 | D29 | D36 | <b>D40</b> | |
| | • | | | | | | | ± 2 | | | | | | | ± 2 | |
| | Drug | | | XmA | b1808 | 7 | | EA | | | XmAb | 18087 | | | EA | |
| | | | | (με | g/kg) | | | | | | (μg/ | kg) | | | | |
| | 1 | 8 | 15 | 22 | 29 | 36 | 40 | 43 | 50 | 57 | 64 | 71 | 78 | 82 | | |
| Part A | 1A | 0.3 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 3 - 6 |
| (Safety | 2A | 0.3 | 1.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 3 - 6 |
| Run-in) | 3A | 0.3 | 1.0 | 2.0 | 4.0 | 4.0 | 4.0 | | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | | 3 - 6 |
| Part A (Expansion) | Expansion A | | | | | | | At | RD coho | rt | | | | | | Up to 22 |

D = day; EA = efficacy assessment (no drug administered); MCC = Merkel cell carcinoma; RD = recommended dose. Maximum escalated dose for each cohort in bold.


Table 3: Part B (MCC) Combination Therapy Safety Run-in and Expansion Cohorts

| | Cycle | | | ( | Cycle 1 | | | | | | ( | Cycle 2 | + | | | Subjects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | and Day | D1 | D8 | D15 | D22 | <b>D29</b> | D36 | <b>D40</b> | D1 | D8 | D15 | D22 | <b>D29</b> | D36 | D40 | |
| | | | | | | | | ± 2 | | | | | | | ± 2 | |
| | Drug | XmAb<br>(μg/ | | Pem (mg) | X | mAb18<br>(μg/kg | | EA | XmAb<br>(μg/ | | Pem (mg) | X | mAb18<br>(μg/kg | | EA | |
| | Study<br>Day | 1 | 8 | 15 | 22 | 29 | 36 | 40 | 43 | 50 | 57 | 64 | 71 | 78 | 82 | |
| | 1B | 0.3 | 0.3 | 400 | 0.3 | 0.3 | 0.3 | | 0.3 | 0.3 | 400 | 0.3 | 0.3 | 0.3 | | 3 - 6 |
| Part B | 2B | 0.3 | 1.0 | 400 | 1.0 | 1.0 | 1.0 | | 1.0 | 1.0 | 400 | 1.0 | 1.0 | 1.0 | | 3 - 6 |
| (Safety<br>Run-in) | 3B | 0.3 | 1.0 | 400 | 1.0 | 2.0 | 2.0 | | 2.0 | 2.0 | 400 | 2.0 | 2.0 | 2.0 | | 3 - 6 |
| | 4B | 0.3 | 1.0 | 400 | 1.0 | 2.0 | 2.0 | | 2.0 | 4.0 | 400 | 4.0 | 4.0 | 4.0 | | 3 - 6 |
| Part B (Expansion) | Expansion B | | | | | | | At RE | ochort cohort | | | | | | | Up to 30 |

18 August 2020

D = day; EA = efficacy assessment (no drug administered); MCC = Merkel cell carcinoma; Pem = pembrolizumab; RD = recommended dose. Maximum escalated dose for each cohort in bold.


Table 4: Part C (SCLC) Monotherapy Safety Run-in and Expansion Cohorts

| | | | | | Cycle | e 1 | | | | | | Cycle | 2+ | | | Subjects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cycle<br>and Day | D1 | <b>D8</b> | D15 | D22 | D29 | D36 | D40 | D1 | D8 | D15 | D22 | D29 | D36 | D40 | |
| | | | | | | | | ± 2 | | | | | | | ± 2 | |
| | Drug | | | XmA | b1808 | 7 | | EA | | | XmAb | 18087 | | | EA | |
| | (μg/kg) (μg/kg) | | | | | | | | | | | | | | | |
| | Study<br>Day | 1 | 8 | 15 | 22 | 29 | 36 | 40 | 43 | 50 | 57 | 64 | 71 | 78 | 82 | |
| Part C | 1C | 0.3 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 | | 3 - 6 |
| (Safety | 2C | 0.3 | 1.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | | 3 - 6 |
| Run-in) | 3C | 0.3 | 1.0 | 2.0 | 4.0 | 4.0 | 4.0 | | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | 4.0 | | 3 - 6 |
| Part C<br>(Expansion) | Expansion C | | | | | | | At l | RD coho | rt | | | | | | Up to 30 |

18 August 2020


D = day; EA = efficacy assessment (no drug administered); RD = recommended dose; SCLC = small cell lung cancer. Maximum escalated dose for each cohort in bold.

## 7.4. Continuation/Discontinuation of Therapy

There will be a pretreatment tumor assessment, followed by a reassessment after each treatment cycle (Table 7).

#### 7.4.1. Continuation Prior to Progression

Subjects who appear to benefit from XmAb18087 or XmAb18087/pembrolizumab combination therapy may continue to receive additional drug treatment until unacceptable toxicity develops, progression occurs, or the Investigator thinks there is no longer clinical benefit to the subject.

To receive study drug past the first cycle, a subject in Part A or Part C must also satisfy the following criteria:

- Does not meet any criteria for stopping dosing (Section 7.8 and Section 10.3)
- Has recovered from any toxicity to  $\leq$  Grade 2 or to baseline
- Has experienced clinical benefit, as assessed by the Investigator

To receive combination therapy past the first cycle, a subject in Part B must satisfy all continuation criteria for Part A and Part C, and, in addition, must have recovered sufficiently from any immune-related adverse event so that he/she is eligible for continuation/re-initiation of study treatment. Refer to Section 7.4 and the pembrolizumab label (Keytruda® Package Insert, 2020) for dose modification and toxicity management guidelines.

For subjects who continue to receive XmAb18087 or XmAb18087 and pembrolizumab combination therapy past the first cycle, tumor assessments will be repeated after every cycle of therapy.

## 7.4.2. Continuation/Discontinuation at Progression

Treatment with XmAb18087 as monotherapy (in Part A and Part C) or as part of the combination regimen (in Part B) will be discontinued upon assessment of progressive disease (PD) per RECIST 1.1 (Appendix A).

A subject on combination therapy who is assessed as having PD per RECIST 1.1 may choose to continue pembrolizumab monotherapy in this clinical trial until confirmatory RECIST 1.1 assessment not less than one month and not more than six weeks after the initial determination of PD if he/she

- Meets all the criteria for continuation of dosing listed above in Section 7.4.1
- Has not experienced a decline in Eastern Cooperative Oncology Group (ECOG) performance status since the baseline assessment
- Does not have signs or symptoms of unequivocal PD or PD at disease sites that pose a medical risk to the subject.

Subjects who are assessed as having initial RECIST 1.1 PD but who wish to continue receiving pembrolizumab monotherapy until confirmatory RECIST 1.1 assessment will be reconsented with a separate consent form to ensure they are aware of all treatment options and therapies that they may be foregoing.


If PD is confirmed on follow-up RECIST 1.1 assessment, the subject must discontinue receiving pembrolizumab in this clinical trial.

If PD is not confirmed by follow-up RECIST 1.1 assessment, the subject must discontinue receiving pembrolizumab in this clinical trial but will continue to be followed for progression and survival.

Subjects will be followed as per Table 7, or until death or the initiation of other anticancer therapy (whichever comes first). Information regarding disease status will be collected by the investigational sites for up to an additional 12 months, or until death or disease progression requiring other anticancer therapy (whichever comes first).

## 7.4.3. Intrasubject Dose Escalation

Intrasubject dose escalation of XmAb18087 is permitted in the study. The subject must meet the following criteria in order to be eligible for treatment at the higher dose level:

- The subject tolerates his/her dose level of XmAb18087
- The subject meets criteria for continuation of therapy prior to progression (Section 7.4.1)
- All subjects in the safety run-in cohort at the next higher dose level have completed the
  first cycle of treatment, and the SRC has made the decision that the higher dose level
  is tolerable

No dose escalation will be permitted for pembrolizumab.

For MCC subjects, crossover from monotherapy (Part A) to combination therapy (Part B) is not permitted. Subjects in Part B may not escalate more than once.

# 7.5. Number of Subjects

Up to 142 subjects will be enrolled; the total number required will depend on the number of safety run-in cohorts required to define each RD for expansion in Part A, Part B, and Part C. Up to 25 clinical investigation sites in the US will enroll subjects in this study.

# 7.6. Treatment Assignment

Subject Screening Number: Subjects who consent for the study will be assigned a Subject Screening Number.

Subject Enrollment Number: Subjects eligible to receive study treatment will be assigned a Subject Enrollment Number.

Enrolled subjects will be assigned to a cohort as follows:

- Subjects with advanced MCC who have received prior treatment with or are ineligible for treatment with anti-PD1 and/or anti-PDL1 will be assigned to a monotherapy cohort in Part A
- Subjects with advanced MCC who are anti-PD1 and anti-PDL1 therapy naïve and who do
  not have a contraindication to anti-PD1 therapy will be assigned to a combination therapy
  cohort in Part B.


• Subjects with extensive stage SCLC who have received prior treatment with standard therapies will be assigned to a monotherapy cohort in Part C.

## 7.7. Safety Run-in Cohorts

In each safety run-in cohort, no more than 1 subject will be initiated on treatment with XmAb18087 on any given day.

The planned initial XmAb18087 dose for all cohorts is  $0.3 \,\mu\text{g/kg}$ . Subsequent doses will then be escalated in steps (except for Cohort 1B, which will use  $0.3 \,\mu\text{g/kg}$  for all doses) as indicated in Table 2, Table 3, and Table 4 in an effort to reduce the incidence and severity of CRS.

For all safety run-in cohorts in Part A, Part B, and Part C, the SRC will decide whether to advance to the next higher dose level cohort based on review of all available safety data. For each cohort, 3 subjects will be initially enrolled. If no subject experiences an adverse event of specific concern (AESC, as defined in Section 7.8 below), the SRC will be convened after all 3 subjects have completed one treatment cycle or discontinued treatment, whichever comes first. If 1 of the initial 3 subjects experiences an AESC, 3 additional subjects will be enrolled in that cohort (up to a total of 6 subjects) prior to convening the SRC. If 2 subjects experience an AESC, no additional subjects will be enrolled until the SRC has convened and made a recommendation based on the available safety data. Based on the type and severity of toxicities observed, the SRC may modify the safety run-in scheme (eg, decreases in dose level, smaller escalation steps, or other changes in the regimen), as long as the changes do not significantly affect the risk profile of the study.

If a subject discontinues treatment prior to completion of the first cycle due to an AE, that subject will not be replaced. If a subject discontinues treatment prior to completion of the first cycle for any other reason, an additional subject may be enrolled as a replacement.

Part A will begin by enrolling 3 to 6 subjects in Cohort 1A. After Cohort 1A dosing is demonstrated to be tolerable and is approved by the SRC, Part B will begin by enrolling Cohort 1B, which is one dose level lower than Cohort 1A.

Part C may begin concurrently with Part A.

The safety run-in portion will continue until establishment of an RD for expansion or until the repeated dose level reaches the highest dose planned in this study.

Enrolling additional subjects beyond 142 will require a protocol amendment.

# 7.8. Criteria for Adverse Events of Specific Concern and Dose Adjustment

The National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0, will be used for grading toxicities, except for CRS, which will be graded using the CRS revised grading system (Section 11.2 or Appendix C; Lee, 2014).

An AESC is defined as an AE or clinically significant abnormal laboratory value (unless clearly attributable to underlying malignancy or concurrent disease) occurring after the initiation of dosing and meeting the criteria listed below:

#### For Parts A, B, and C:

1. Any Grade 5 toxicity


- 2. Grade  $\geq$  3 thrombocytopenia lasting  $\geq$  7 days or  $\geq$  Grade 3 thrombocytopenia of any duration if associated with  $\geq$  Grade 3 bleeding
- 3. Grade 4 neutropenia or Grade 3 febrile neutropenia lasting ≥ 7 days, or Grade 4 febrile neutropenia
- 4. Any  $\geq$  Grade 3 nonhematological toxicity, **except**:
  - a. Grade 3 fatigue, asthenia, fever, anorexia, or constipation
  - b. Grade 3 nausea, vomiting, diarrhea, or abdominal pain controlled by medical management that decreases to  $\leq$  Grade 2 within  $\leq$  7 days
  - c. Grade 3 alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) that decrease to  $\leq$  Grade 2 within  $\leq$  5 days
  - d. Grade ≥ 3 gamma glutamyl transferase (GGT), unless it occurs with AST, ALT, and/or total bilirubin values that meet AESC criteria
  - e. Grade 3 electrolyte abnormalities that are clinically insignificant, or treatable, and that resolve, with or without intervention, to < Grade 2 in < 72 hours
  - f. Grade 3 or 4 lipase values that are not accompanied by ≥ Grade 3 amylase values or clinical symptoms or radiographic evidence of pancreatitis

#### Additional Criterion for Part B (combination therapy) only:

1. Any immune related adverse event (IRAE) that requires permanent discontinuation of study drug according to the guidelines in Table 18

Subjects who experience any toxicity should be followed until the toxicity stabilizes or has returned to their baseline level, or until the commencement of a new anticancer treatment.

Refer to Section 10.3 for safety criteria for adjustment or stopping XmAb18087 and pembrolizumab.

## 7.8.1. Replacement of Subjects

A subject enrolled in a safety run-in cohort who withdraws from study before completing the first cycle for reasons other than an AE will be considered to have inadequate data for evaluation by the SRC. In such cases, a replacement subject may be enrolled to receive the same dose of XmAb18087 (and pembrolizumab, when applicable) as the subject who withdrew prematurely. Subjects enrolled in the safety run-in cohorts who are discontinued from the study for any reason after the first cycle will not be replaced.

#### 7.8.2. Criteria for Study Termination

Sequential boundaries will be used to monitor AESC rates over the monotherapy expansion cohorts and combination therapy expansion cohorts, separately. If excessive numbers of AESC are seen; that is, if the number of AESC that occur in either expansion cohort is equal to or exceeds a boundary,  $b_n$ , out of n subjects (n = all safety-evaluable subjects in the disease-specific expansion cohort [Table 5]), then enrollment will be suspended until the SRC has met.


**Table 5:** Boundaries for AESC Incidence: Cohort A

| Subjects, n<br>of 22 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Boundary, b <sub>n</sub> | - | - | 3 | 3 | 3 | 4 | 5 | 5 | 6 | 6 | 6 | 7 | 7 | 7 | 8 | 8 | 8 | 8 | 9 | 9 | 9 | 10 |

AESC = adverse event of specific concern.

This is a Pocock-type stopping boundary that yields the probability of crossing the boundary of at most 7.5% when the rate of AESC is equal to the acceptable rate of 20% (Ivanova, 2005). If instead the rate of AESC is an excessive 40%, then on average only 14 of the 22 patients will complete the toxicity follow up period before the boundary is crossed.

Table 6: Boundaries for AESC Incidence: Cohorts B and C

| Subjects, n<br>of 30 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Boundary, b <sub>n</sub> | - | - | 3 | 3 | 3 | 4 | 5 | 5 | 6 | 6 | 6 | 7 | 7 | 7 | 8 | 8 | 8 | 6 | 9 | 9 |
| Subjects, n of 30 | 21 | 22 | 23 | 24 | 25 | 26 | 27 | 28 | 29 | 30 | | | | | | | | | | |
| Boundary,<br>b <sub>n</sub> | 9 | 10 | 10 | 10 | 11 | 11 | 11 | 11 | 12 | 12 | | | | | | | | | | |

AESC = adverse event of specific concern.

This is a Pocock-type stopping boundary that yields the probability of crossing the boundary of at most 8% when the rate of AESC is equal to the acceptable rate of 20% (Ivanova, 2005). If instead the rate of AESC is an excessive 40%, then on average only 17 of the 30 patients will complete the toxicity follow up period before the boundary is crossed.

If the enrollment of a disease-specific expansion cohort has been suspended in accordance with this section, it may not be reopened until the SRC has met, considered the available data, and made a decision to continue, with or without modifications to the trial.

# 7.9. Study Assessments

The Schedule of Assessments is shown in Table 7. Pretreatment, treatment, and follow-up procedures are detailed in Sections 7.9.1 through 7.9.5.


**Table 7:** Schedule of Assessments

| Evaluation or Procedure | Pretrea | tment | | | | | | | Cycle | e 1 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screen<br>(-28 to<br>-2) | Day<br>-1 | 1 | 2 | 3 | 8 | 9 | 10 | 15 | 22 | 29 | 36 | 37 | 38 | 39 | 40<br>± 2 |
| Informed consent | X | | | | | | | | | | | | | | | |
| NETSPOT Gallium 68 dotatate PET/CT scan <sup>a,b</sup> | X | | | | | | | | | | | | | | | X |
| Review of inclusion/exclusion criteria | X | | | | | | | | | | | | | | | |
| Collection of FFPE tumor sample/slides | X | | | | | | | | | | | | | | | |
| Record tumor genetic information | X | | | | | | | | | | | | | | | |
| Inpatient status <sup>c,d</sup> | | X | X | X | X | X | X | X | | | | X | X | X | X | |
| XmAb18087 administration <sup>e,f</sup> | | | X | | | X | | | X | X | X | X | | | | |
| Pembrolizumab administration <sup>f</sup> | | | | | | | | | X | | | | | | | |
| Medical history <sup>g</sup> | X | X | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| Physical examination <sup>g,h</sup> | X | X | | X | X | X | X | X | X | X | X | X | | | | X |
| Neurologic examination <sup>i</sup> | | X | | | | | | | | | | | | | | |
| Vital signs <sup>c,j,k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Height | | X | | | | | | | | | | | | | | |
| Weight | | X | X | | | X | | | X | X | X | X | | | | |
| ECOG performance statush | X | X | X | | | X | | | X | X | X | X | | | | |
| 12-lead electrocardiogram (supine) <sup>l,m</sup> | X | X | X | | | X | X | | X | X | X | X | | | | |
| CBC w/ differential (absolute and percentage), platelet count <sup>h</sup> | X | | X | X | X | X | X | X | X | X | X | X | | | | |
| Chemistry panel <sup>h</sup> | X | | X | X | X | X | X | X | X | X | X | X | | | | |
| Coagulation panelh | X | | X | X | | X | | X | X | X | X | X | | | | |
| Urinalysis | X | X | | X | | X | | X | X | X | X | X | | | | |
| HBsAg, HBcAb, HCV, HIV | X | | | | | | | | | | | | | | | |


**Table 7:** Schedule of Assessments (Continued)

| Evaluation or Procedure | Pretrea | itment | | | | | | | Cycle | : 1 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screen<br>(-28 to<br>-2) | Day<br>-1 | 1 | 2 | 3 | 8 | 9 | 10 | 15 | 22 | 29 | 36 | 37 | 38 | 39 | 40<br>± 2 |
| Serum β–hCG (females of childbearing potential) FSH (postmenopausal) <sup>n</sup> | X | X | | | | | | | | X | | | | | | |
| Flow cytometry (blood) <sup>o</sup> | | | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Cytokine/inflammation panel <sup>p</sup> | | | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Polyoma virus assay (serum) <sup>q</sup> | | X | | | | | | | | | | | | | | |
| Biobanking sample (blood) <sup>r,s</sup> | | X | | X | | X | | | | | | | | | | X |
| PK blood sampling <sup>t</sup> | | X | X | X | X | X | | X | X | X | X | X | X | X | X | |
| Immunogenicity (ADA) blood sampling <sup>u</sup> | | X | X | | | X | | | X | X | X | X | | | | |
| RECIST 1.1 tumor assessment <sup>v</sup> | X | | | | | | | | | | | | | | | X |
| Monitor/record adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Fresh tumor biopsy (optional) <sup>s,w</sup> | X | | | | | | | X | | | | | | | | |


**Table 7:** Schedule of Assessments (Continued)

| Evaluation or Procedure | | | C | ycle 2 and | Higher | | |
|---|---|---|---|---|---|---|---|
| Study Day | 1 | 8 | 15 | 22 | 29 | 36 | 40 ± 2 |
| NETSPOT Gallium 68 dotatate PET/CT scan <sup>a,b</sup> | | | | | | | X |
| XmAb18087 administration <sup>e,f</sup> | X | X | X | X | X | X | |
| Pembrolizumab administration <sup>f</sup> | | | X | | | | |
| Physical examination | X | X | X | X | X | X | |
| Vital signs <sup>j, k</sup> | X | X | X | X | X | X | |
| Weight | X | X | X | X | X | X | |
| ECOG performance status <sup>h</sup> | X | X | X | X | X | X | |
| 12-lead electrocardiogram (supine) <sup>l,m</sup> | X | X | X | X | X | X | |
| CBC w/ differential (absolute and percentage), platelet count <sup>h</sup> | X | X | X | X | X | X | |
| Chemistry panel <sup>h</sup> | X | X | X | X | X | X | |
| Coagulation panel <sup>hl</sup> | X | X | X | X | X | X | |
| Urinalysis | X | | | X | | | |
| Serum $\beta$ -hCG (females of childbearing potential) FSH (postmenopausal) <sup>n</sup> | X | | | X | | | |
| Flow cytometry (blood) <sup>o</sup> | | | | X | | X | |
| Cytokine/inflammation panel <sup>p</sup> | X | | | X | | | |
| PK blood sampling <sup>t</sup> | X | | X | | | | |
| Immunogenicity (ADA) blood sampling <sup>u,x</sup> | X | | X | X | | X | |
| RECIST 1.1 tumor assessment <sup>v</sup> | | | | | | | X |
| Monitor/record adverse events | X | X | X | X | X | X | |
| Concomitant medications | X | X | X | X | X | X | |


Table 7: **Schedule of Assessments (Continued)** 

| Evaluation or Procedure | | | Post-treatment | |
|---|---|---|---|---|
| Study Day | ЕОТ | 14 d post-EOT | 28 d post-EOT | Long-term Follow-up (6 & 12<br>mo after EOT) |
| NETSPOT Gallium 68 dotatate PET/CT scan <sup>a,b</sup> | X | | | |
| Medical history | | | X | |
| Physical examination | X | X | X | |
| Vital signs <sup>i, k</sup> | X | X | X | |
| Weight | X | X | X | |
| ECOG performance statush | X | X | X | |
| 12-lead electrocardiogram (supine) l,m | | | X | |
| CBC w/ differential (absolute and percentage), platelet count <sup>h</sup> | X | X | X | |
| Chemistry panel <sup>h</sup> | X | X | X | |
| Coagulation panel <sup>h</sup> | X | X | X | |
| Urinalysis | X | X | X | |
| HBsAg, HBcAb, HCV, HIV | X | | | |
| Serum β–hCG (females of childbearing potential) FSH (postmenopausal) <sup>n</sup> | X | | X | |
| Flow cytometry (blood) <sup>o</sup> | X | X | X | |
| Cytokine/inflammation panel <sup>p</sup> | | | | |
| Polyoma virus assay (serum) <sup>q</sup> | X | | X | |
| PK blood sampling <sup>t</sup> | X | X | X | |
| Immunogenicity (ADA) blood sampling <sup>u,x</sup> | X | X | X | |
| RECIST 1.1 tumor assessment <sup>v</sup> | X | | | |
| Monitor/record adverse events | X | X | X | |
| Concomitant medications | X | X | X | |
| Phone/email/mail contact for progression | | | | X |

Version 1.0  Abbreviations: ADA = anti-drug antibody; β–hCG = beta unit of human chorionic gonadotrophin; CBC = complete blood counts; CT = computed tomography; EOI = end of infusion. EOT = end of treatment; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; FACS = fluorescence-activated cell sorting; FFPE = fresh frozen paraffin-embedded; FSH = follicle-stimulating hormone; HBsAg = hepatitis B surface antigen; HBcAb = hepatitis B core antibody; HCV = hepatitis C virus; HIV = human immunodeficiency virus; mo = month; MRI = magnetic resonance imaging; NET = neuroendocrine tumors; PE = physical examination; PET = positron emission tomography; PK = pharmacokinetic; RECIST = Response Evaluation Criteria In Solid Tumors; SSTR2 = somatostatin

- <sup>a</sup> If subject has undergone NETSPOT gallium 68 dotatate PET/CT scan within 6 weeks prior to enrollment and the images and a report of results are available for collection, the scan need not be repeated at baseline. If SSTR2 radionuclide scanning and RECIST 1.1 tumor assessment by CT/MRI are planned within 2 days of each other. RECIST imaging should be conducted first.
- b NETSPOT gallium 68 dotatate PET/CT scan will be performed on Day 40 ± 2 of Cycle 1 and of every second cycle thereafter; that is, at the end of Cycle 3, Cycle 5, etc. The EOT scan will be performed only if the subject has not undergone scan within the past 2 months.
- <sup>c</sup> On Day -1, hospitalization is optional. Hospitalization on Days 36 through 39 in Cycle 1 is optional if PK sampling cannot be accommodated as an outpatient. Vital sign assessments on Days 36 through 39 in Cycle 1 will be performed only if the subject is hospitalized.
- d Any subject who has shown symptoms of CRS during a required inpatient hospitalization will be monitored as an inpatient for at least 24 hours after the symptoms have subsided.
- EXMAb18087 will be administered as be observed as inpatients for the first 2 doses. For all other infusions of XmAb18087, the subject will be observed for at least 4 hours following subsequent infusions, except that the observation period may be decreased to 2 hours if no infusion reactions have occurred for at least 3 consecutive infusions and the subject has completed 4 infusions at the highest dose for that subject.
- f XmAb18087 is administered on Day 15 in Parts A and C only. Pembrolizumab is administered on Day 15 of each cycle in Part B only. XmAb18087 is NOT to be administered on Day 15 in Part B. Pembrolizumab will be provided by sites as standard of care.
- g Complete medical history and PE is to be performed at Screening. For all the other time points, only an abbreviated, symptom-directed PE is to be performed.
- May be performed up to 24 hours prior to infusion. The following procedures that are completed on Day -1 within 24 hours of Cycle 1 Day 1 dosing do not need to be repeated on Cycle 1 Day 1: PE, ECOG, and local safety laboratories (eg, CBC with differential and platelets, chemistry panel, coagulation panel, and urinalysis). These safety laboratory assessments will be performed by the central laboratory and should also be performed by local clinical site laboratories so that clinical site personnel can review results before administering XmAb18087.
- Baseline neurologic examination to be performed on Day -1. If a subject appears to be experiencing neurologic toxicity, the neurologic examination should be repeated as necessary to evaluate the subject's condition. Guidelines on management of neurologic toxicity are included in both Section 11.3.3.4 and Appendix C.
- Supine blood pressure and pulse rate, body temperature, respiratory rate, and blood oxygen saturation by pulse oximetry. On days of XmAb18087 infusions, vital signs should be taken within 60 minutes of predose; 15, 30, and 60 minutes after start of infusion (± 5 minutes for each time point); immediately (within 5 minutes) before EOI; 15, 30, and 60 minutes after EOI (± 5 minutes for each time point); and then hourly (± 5 minutes) for 3 hours. When possible, vitals should be measured before blood sampling. Oxygen saturation levels will be captured with each vital sign collection; however, pulse oximetry monitoring must be maintained continuously throughout the entire admission or observation period for each administration of XmAb18087. For information on management of oxygen saturation of 90% or lower, see Section 11.3.3.1. All vital signs during infusion should be taken with the subject in the same position. On nondosing days, vitals should be measured before blood sampling.
- Non days of pembrolizumab infusions, vital signs should be taken immediately prior (within 10 minutes before blood sampling) to the start of infusion; during the infusion at 5 and 15 minutes (± 2 minutes); immediately (within 2 minutes) before the EOI; and at 15 minutes (± 2 minutes) after EOI.
- On days when XmAb18087 is infused, electrocardiograms should be taken prior to infusion, 2 to 4 hours after EOI, and if clinically indicated.
- $^{\rm m}$   $\,$  Part B only: ECGs are not performed on days when pembrolizumab is administered.

receptor 2.

- <sup>n</sup> Once postmenopausal status has been established by FSH, this test need not be repeated during the clinical trial.
- In Cycle 1, whole blood for flow cytometry (FACS) analysis will be obtained predose on Day 1 (± 1 hour); on Day 2 (24 hours post-EOI ± 3 hours); on Day 3 (48 hours post-EOI ± 3 hours); predose on Day 8 ± 1 hour; on Day 9 (24 hours post-EOI ± 3 hours); on Day 10 (48 hours post-EOI ± 3 hours); predose on Day 15 ± 1 hour; predose on Day 22 ± 1 hour; predose on Day 29 ± 1 hour; predose on Day 36 ± 1 hour; on Day 37 (24 hours post-EOI ± 3 hours); on


- Day 38 (48 hours post-EOI  $\pm$  3 hours); and on Day 39 (72 hours post-EOI  $\pm$  3 hours). In **Cycles 2 and higher**, whole blood for FACS will be obtained predose on Day 22  $\pm$  2 days and on Day 36  $\pm$  2 days. **Upon discontinuation from the study**, whole blood for FACS analysis should be obtained at EOT ( $\pm$  2 days), at 14 days post-EOT ( $\pm$  2 days), and at the 28 days post-EOT visit( $\pm$  2 days.)
- In **Cycle 1**, serum for cytokine profile analysis will be obtained predose on Day 1, 8, and 36 and at 5 minutes (± 1 minute), 1 hour (± 10 minutes), 2 hours (± 10 minutes), 4 hours (± 10 minutes), 7 hours (± 10 minutes), and 10 hours (± 10 minutes) post-EOI; on Days 2, 9, and 37 (24 hours post-EOI ± 3 hours), Day 3, 10, and 38 (48 hours post-EOI ± 3 hours), and on Day 39 (72 hours post-EOI ± 3 hours). Additionally, samples will be collected predose on Days 15, 22, and 29 and at 5 minutes (± 1 minute), 1 hour (± 10 minutes), 2 hours (± 10 minutes), 4 hours (± 10 minutes), and 7 hours (± 10 minutes) post EOI. In **Cycle 2 and higher**, serum for cytokine profile analysis will be obtained on Day 1 and Day 22 (± 2 days) of each cycle predose and at 1 hour (± 10 minutes), 2 hours (± 10 minutes), and 4 hours (± 10 minutes) post EOI. Serum should also be drawn at any time there is clinical suspicion of cytokine release syndrome and repeated 4 hours later.
- <sup>q</sup> Polyoma virus assay serum collection is for Part A and Part B only.
- <sup>r</sup> Including serum, peripheral blood, and nucleic acid samples.
- s Optional; by specific subject consent.
- In **Cycle 1**, serum for PK analysis will be obtained at Day -1; on Days 1 and 36 predose and at 5 minutes (± 1 minute), 1 hour (± 10 minutes), 2 hours (± 10 minutes), 4 hours (± 10 minutes), 7 hours (± 10 minutes), and 10 hours post-EOI (± 10 minutes, Day 1 only); on Days 2 and 37 (24 hours post-EOI ± 3 hours), and Days 3 and 38 (48 hours post-EOI ± 3 hours), and Day 39 (72 hours post-EOI ± 3 hours); on Day 8 predose and at 5 minutes (± 1 minute) post-EOI; on Day 10 (48 hours post-EOI); and on Days 15, 22, and 29 predose and at 5 minutes post-EOI (± 1 minute). In **Cycles 2 and higher**, serum for PK analysis will be collected on the first day of each cycle (± 2 days) predose and 5 minutes (± 1 minute) post-EOI (all subjects). Subjects in Part B only (combination therapy) will also have serum collected for PK analysis on Day 15 at predose and 5 minutes (± 1 minute) post-EOI. Upon **discontinuation from the study**, serum for PK analysis should be obtained at the EOT visit (± 2 days), the 14-day post-EOT visit (± 2 days), and the 28 day post-EOT visit (± 2 days).
- In Cycle 1, serum for ADA will be collected on Day -1 and predose (± 1 hour) on Days 1, 8, 15, 22, 29, and 36. In Cycles 2 and higher, serum for ADA analysis will be collected predose on Days 1, 15, 22 and 36 (± 2 days). Upon discontinuation from the study, serum for ADA will be collected at EOT (± 2 days), at 14 days post-EOT (± 2 days), and at 28 days post-EOT (± 2 days).
- Radiographic tumor evaluation will be performed by CT/MRI at baseline and at all other disease assessment time points. All studies for the baseline RECIST assessment should be performed within 14 days prior to the first dose of drug. The EOT tumor assessment will not be performed if the subject has had an assessment within the past 30 days.
- <sup>w</sup> The post-treatment fresh tumor biopsy should be performed between 12 and 21 days after first dose of XmAb18087.
- Subjects with a positive ADA at termination will be followed every 28 days (± 3 days) until ADA reverts to baseline or until the next intervening treatment.


#### 7.9.1. Pretreatment Evaluations

Only those subjects who meet all inclusion (Sections 8.1 and 8.2) and no exclusion (Sections 8.6 and 8.7) criteria specified may be enrolled into this study. Prior to the initiation of any on-study testing, including screening testing, the subject must have signed the ICF and received a Subject Screening Number (Section 7.6). The pretreatment period lasts for up to 28 days and includes screening evaluations (Day -28 to -2) and baseline assessments (defined as the assessment immediately prior to the first dose).

Prior to administration of XmAb18087, each subject must have completed all screening activities and received approval via the eligibility checklist from the Medical Monitor.

#### **7.9.1.1.** Screening Period (Day -28 to -2)

Subjects will undergo a Screening Visit 2 to 28 days prior to the planned first day of study treatment. Screening assessments are as follows:

- Obtain signed informed consent (Section 17.3)
- Review inclusion and exclusion criteria (Sections 8.1, 8.2, 8.6, and 8.7)
- Medical history
- Demographics
- Physical examination (PE; Section 11.7)
- Collect formalin-fixed paraffin embedded (FFPE) tumor sample or slides for immunohistochemical assessment of MCPyV status (MCC subjects only), tumor cell SSTR2 expression and immune cell expression of proliferation and exhaustion markers
- Perform tumor assessment by CT/magnetic resonance imaging (MRI) per RECIST 1.1 criteria and guidelines (Appendix A) within 14 days prior to the first dose of drug
- Perform NETSPOT gallium 68 dotatate PET/CT if not performed within 3 months prior to enrollment (refer to study manual for details on performing NETSPOT gallium 68 dotatate PET/CT). If the subject has undergone NETSPOT gallium 68 dotatate PET/CT scan within 3 months prior to enrollment and the images and reports of results are available, the scan need not be repeated at baseline; however, a copy of images and the report of scan results must be collected.
- Record any available genetic information on the tumor, including sequencing data
- ECOG performance status (Appendix B)
- Vital signs (Section 11.8)
- Electrocardiogram (ECG) standard 12-lead, supine position (Section 11.6)
- Complete blood count (CBC; Section 11.5)
- Chemistry panel (Section 11.5)
- Coagulation panel (Section 11.5)


- Screening test for hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb; a subject whose HBsAg is negative and HBcAb is positive may be enrolled if a hepatitis B virus [HBV] DNA test is negative and either the subject is treated with potent antiviral therapy or is retested for HBsAg and HBV DNA every month while on study drug treatment).
- Screening tests for human immunodeficiency virus (HIV) and hepatitis C virus (HCV)
- Serum beta human chorionic gonadotropin (β-hCG) pregnancy test for women of childbearing potential or follicle-stimulating hormone (FSH) for postmenopausal women (Section 11.5)
- Urinalysis (Section 11.5)
- Record concomitant medications (Section 9.2)
- Record adverse events (using CTCAE and CRS revised grading system for grading; Section 11.1)
- Pretreatment fresh tumor biopsy (optional; by specific subject consent) to be examined
  by fluorescent immunohistochemical assay for tumor-cell expression of SSTR2 and
  tumor and immune-cell expression of proliferation and exhaustion markers, and by
  Nanostring analysis of nucleic acid and protein content

## 7.9.1.2. Baseline Assessments (Day -1 or 1)

If a test or assessment is performed on both Day -1 and Day 1, the Day 1 (predose) test is considered the baseline:

- Medical history
- Abbreviated PE (Section 11.7)
- Neurological examination
- ECOG performance status (Appendix B)
- Vital signs (Section 11.8)
- Height, weight
- ECG: standard 12-lead, supine position (Section 11.6)
- CBC (Section 11.5)
- Chemistry panel (Section 11.5)
- Coagulation panel (Section 11.5)
- Urinalysis (Section 11.5)
- Urine β-hCG pregnancy test for women of childbearing potential (Section 11.5)
- Blood for cell surface markers by flow cytometry or other similar bioanalytical methods (Section 13.3)
- Serum for MCPyV assay (Part A and Part B only)


- PK, cytokine/inflammation panel blood sample (Section 13.1)
- Immunogenicity (ADA) blood sample (Section 13.1)
- Blood for biobanking (Section 13.4)
- Record concomitant medications (Section 9.2) and AEs

## 7.9.2. Subject Enrollment

Subjects who have completed screening activities and whose eligibility has been confirmed by the Medical Monitor will be considered enrolled in the study.

## 7.9.3. Treatment Cycle Assessments

The schedule of required procedures and clinical site study days for each cycle are detailed in the Schedule of Assessments (Table 7). The day prior to Cycle 1 Day 1 is Day -1.

Subjects will be followed for PFS and overall survival at 6 and 12 months after end of treatment (EOT) by telephone, email, or mail contact from the clinical site (Section 7.9.5).

Procedures during the treatment cycles to 4 weeks after EOT are detailed in Sections 7.9.3.1 to 7.9.3.2. Study days for required procedures are specified in the Schedule of Assessments (Table 7).

#### 7.9.3.1. Clinical Assessments

PEs and laboratory evaluations may be performed within 24 hours prior to XmAb18087 infusion:

- Record concomitant medications and AEs (CTCAE and CRS revised grading system, Section 11.1).
- Abbreviated, symptom-directed PE, including weight
- ECOG performance status (Appendix B)
- Vital signs (Section 11.8):
  - On infusion days, time points include: within 60 minutes of predose; approximately 15, 30, and 60 minutes after start of infusion (± 5 minutes for each time point); immediately (within 5 minutes) before end of infusion (EOI; if different than 60 minutes from start of infusion); approximately 15, 30, and 60 minutes after EOI (± 5 minutes for each time point); and then hourly (± 5 minutes) for 3 hours. The pulse oximetry for blood oxygen saturation level needs to be captured with each vital sign collection; however, pulse oximetry monitoring must be maintained continuously throughout the entire admission or observation period for each administration of XmAb18087. For information on management of oxygen saturation of 90% or lower, see Section 11.3.3.1.
  - On non-dosing days, vitals should be measured before blood is drawn.
  - For subjects who tolerate 3 XmAb18087 consecutive infusions without an infusion reaction during the infusion or postinfusion observation period and who have completed 4 infusions at the highest dose for that subject, the postinfusion


observation period and vital signs assessment may be reduced from 4 hours to 2 hours.

#### 7.9.3.2. Laboratory Assessments

Unless otherwise specified, assessments during Cycle 1, Days 1, 8, 15, 22, 29, and 36 should be completed  $\pm$  1 hour of the scheduled time; for other days during Cycle 1,  $\pm$  3 hours; and for subsequent cycles and disease assessments,  $\pm$  2 days. Details for laboratory assessments are provided in Section 11.5 and Section 11.6; details for PK, PD, flow cytometry, and biobanking are provided in Section 13.

Laboratory assessments include the following:

- CBC
- Chemistry panel
- Coagulation panel
- Urinalysis
- Serum pregnancy test for women of childbearing potential
- Blood for cell surface markers by flow cytometry or similar bioanalytical methods (see the Laboratory Manual for detailed instructions)
- PK (see the Laboratory Manual for detailed instructions)
- Cytokine/inflammation panel (see the Laboratory Manual for detailed instructions)
- ADA blood sample (see the Laboratory Manual for detailed instructions)
- Biobanking blood sample (optional; by specific subject consent)
- ECG, standard 12-lead
- RECIST 1.1 tumor assessment by CT/MRI (See Appendix A)
- Post-treatment fresh tumor biopsy (optional; by specific subject consent) to be examined by various immunohistochemistry assays for tumor-cell expression of SSTR2 and tumor- and immune-cell expression of proliferation and exhaustion markers, and transcriptomic analysis by Nanostring. The optional post-treatment fresh tumor biopsy should be performed between 12 and 21 days after the first dose of XmAb18087.
- NETSPOT gallium 68 dotatate PET/CT after the first cycle of treatment and, for subjects continuing to receive study drug, after every second cycle thereafter NETSPOT gallium 68 dotatate PET/CT should be performed after RECIST tumor assessment by CT/MRI has been completed. Refer to study manual for details on performing NETSPOT gallium 68 dotatate PET/CT.


#### 7.9.3.3. End-of-Treatment Visit

Subjects will have their EOT visit at the end of the last cycle of treatment. If a subject terminates before the end of a cycle, the EOT assessments (Table 7, Schedule of Assessments) will be performed on the day of study termination.

Subjects with a positive ADA at study termination will be followed every 28 days ( $\pm$  3 days), if feasible, until administration of another anticancer therapy, or until ADA levels return to baseline if results are available.

#### 7.9.4. Post-treatment Follow-up Period (2 Weeks and 4 Weeks After EOT)

Subjects will have visits 14 days post-EOT and 28 days post-EOT. Assessments are as indicated in Table 7. Once these two visits have been completed, the subject will be considered as having completed participation in the clinical trial. If a subject enrolls into another trial or requires treatment before either of these scheduled visits, the visits may be performed earlier. If a subject is unable to return for any scheduled visits after the end of treatment, he/she will be considered as having completed study requirements at the end of treatment.

#### 7.9.5. Long-Term Follow-up Period (6 and 12 Months After EOT)

Subjects will be contacted by site staff by telephone, email, or mail at 6 and 12 months after their active participation in the study ends to gather information about disease progression and survival. Completion of the long-term follow-up period is not required for a subject to be considered as having completed the clinical trial.

## 7.10. Discussion of Study Design

This is a Phase 1b/2, multiple-dose study designed to describe safety and efficacy, and to assess PK and immunogenicity of XmAb18087 monotherapy and in combination with pembrolizumab in subjects with metastatic MCC or locoregional MCC that has recurred after locoregional therapy with surgery and/or radiation therapy, and XmAb18087 monotherapy in subjects with extensive-stage SCLC that has progressed after standard therapies.

Part A of the study will enroll safety run-in cohorts of subjects with advanced MCC that has progressed after treatment with standard therapies to confirm the safety and tolerability of XmAb18087 monotherapy administered IV with weekly step-up dosing for 42-day cycles. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 monotherapy using the RD identified following the safety run-in.

Part B of the study will enroll safety run-in cohorts of subjects with advanced MCC not previously treated with anti-PD1 or anti-PDL1 agents, and for whom pembrolizumab as a single agent is indicated, to confirm the safety and tolerability of XmAb18087 in combination with pembrolizumab. Subjects will receive step-up IV dosing of XmAb18087 on Days 1, 8, 22, 29, and 36, and IV dosing of pembrolizumab on Day 15 of each 42-day cycle. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 plus pembrolizumab combination therapy using the RD identified following the safety run-in.

Enrollment into the first safety run-in cohort of Part B (Cohort 1B) may begin after the first safety run-in cohort in Part A (Cohort 1A, one dose level higher than Cohort 1B) has completed the first cycle and the regimen has been demonstrated to be tolerable.


Part C of the study will enroll safety run-in cohorts of subjects with extensive-stage SCLC that has progressed after treatment with standard therapies to confirm the safety and tolerability XmAb18087 monotherapy. The safety run-in will follow the same cohort schema as described for Part A to identify a RD for expansion in SCLC. Additional subjects will be enrolled into an expansion cohort and will receive XmAb18087 monotherapy using the RD identified following the safety run-in.

Enrollment into Part C may begin concurrently with Part A.

#### 7.10.1. Risk/Benefit and Ethical Assessment

XmAb18087 has been characterized through an extensive program of in vitro and in vivo testing which demonstrates that the drug binds CD3 and SSTR2 and is active against SSTR2<sup>+</sup> cells and tumors. The pharmacology and toxicology of the drug have also been studied in numerous experiments using cynomolgus monkeys, the relevant species for a CD3-directed bsAb. Pharmacology results show that XmAb18087 activates T cells, and toxicology results, as well as results from the first 42 subjects dosed in the XmAb18087-01 trial, indicate that the drug can be administered safely within the careful program of prophylactic medication, frequent subject assessment, and close observation that the XmAb18087-02 clinical trial protocol describes. Given that Part A and Part C of the XmAb18087-02 trial are being conducted in subjects with advanced cancer for which there is no effective available therapy, the sponsor believes that the administration of monotherapy under the auspices of this clinical study is ethical.

Pembrolizumab (Keytruda<sup>®</sup>) is approved for the treatment of adult and pediatric patients with recurrent locally advanced or metastatic MCC. Given that the combination of XmAb18087 and pembrolizumab will be administered to this patient population within a careful program of frequent subject assessment and close observation, the Sponsor believes that the proposed combination therapy portion of the clinical study is ethical.

## 7.10.2. Termination of Study

If the Investigator or the Sponsor becomes aware of conditions or events that suggest a possible hazard to subjects should the clinical study continue, the clinical study may be terminated after appropriate consultation among the involved parties. The clinical study also may be terminated at the Sponsor's discretion, also in the absence of such a finding.

Conditions that may warrant termination of the clinical study include, but are not limited to:

- The discovery of an unexpected, relevant, or unacceptable risk to the subjects enrolled in the clinical study.
- Failure to enroll subjects at the required rate.
- A decision of the Sponsor to suspend or discontinue development of the IMP.

Should the study be terminated and/or the site closed for whatever reason, all documentation pertaining to the study and IMP must be returned to the Sponsor. Any actions required for assessing or maintaining study-subject safety will continue as required, despite termination of the study by the Sponsor.

Details for study termination due to AESC are provided in Section 7.8.2.


#### 8. SELECTION AND WITHDRAWAL OF SUBJECTS

## 8.1. Inclusion Criteria for All Cohorts

Each subject must meet all of the following inclusion criteria to be enrolled in the study:

- Able to provide written informed consent
- Adult subjects  $\geq$  18 years
- Disease measurable by RECIST 1.1 criteria using either CT or MRI scan
- ECOG performance status of 0 or 1
- All subjects must have adequate archival tumor sample (slides or archival FFPE block[s] containing tumor that has not been previously irradiated; FFPE blocks are preferred to slides, and newly obtained biopsies are preferred to archived tissue. Refer to the laboratory manual for further instructions). Excepted are subjects who consent to having a fresh tumor biopsy to provide a fresh tumor sample instead of the archival tumor sample.
- Female subjects of childbearing potential must agree to use a highly effective method of birth control during and for 4 weeks after completion of study. Women are considered to be of childbearing potential unless it is documented that they are over the age of 60 OR postmenopausal by history with no menses for 1 year and confirmed by FSH (using local reference ranges) OR have a history of hysterectomy and/or bilateral oophorectomy OR have a history of bilateral tubal ligation. Highly effective methods of birth control include combined hormonal birth control (oral, intravaginal, or transdermal), or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or intrauterine), intrauterine devices (IUDs), intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner (provided partner is the sole sexual partner and there has been a medical assessment of surgical success), or sexual abstinence as defined in Section 8.9.1.
- Fertile male subjects must be willing to practice a highly effective method of birth control for the duration of the study and continuing for 4 weeks after the last dose of XmAb18087 or pembrolizumab (when applicable). Highly effective methods of birth control include vasectomy or a condom in combination with double-barrier methods, spermicide, hormonal birth control, or IUD (nonhormonal) used by the woman.
- Able and willing to complete the entire study according to the study schedule

## 8.2. Additional Inclusion Criteria for Part A and Part B Cohorts:

In addition to the inclusion criteria above, the following criteria are required for Parts A and B safety run-in and expansion cohorts:

Histologically or cytologically confirmed metastatic MCC or locoregional MCC that
has recurred following standard locoregional therapy with surgery and/or radiation
therapy.


## 8.3. Additional Inclusion Criteria for Part A Cohorts:

In addition to the inclusion criteria above, the following criteria are required for Part A safety run-in and expansion cohorts:

• Subjects must have progressed on or been ineligible for treatment with anti-PD1 or anti-PDL1 therapy.

#### 8.4. Additional Inclusion Criteria for Part B Cohorts:

In addition to the inclusion criteria above, the following criteria are required for Part B safety run-in and expansion cohorts:

• Subjects must be eligible to receive pembrolizumab as standard of care.

#### 8.5. Additional Inclusion Criteria for Part C Cohorts:

In addition to the inclusion criteria above, the following criteria are required for Part C safety run-in and expansion cohorts:

• Histologically or cytologically confirmed extensive-stage SCLC that has progressed following standard therapies

#### 8.6. Exclusion Criteria for All Cohorts

Subjects who meet any of the following criteria will be excluded from the study:

- History of prior organ or bone marrow transplant
- History of chronic lymphocytic leukemia
- Subjects currently receiving anticancer therapies
- Subjects who have received anticancer therapies within 2 weeks of the start of study drug (including chemotherapy, radiation therapy, immunotherapy, etc.)
- Prior therapy with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA4, OX40, CD137) AND were permanently discontinued from that treatment due to an IRAE
- Failure to recover from any IRAE from prior cancer therapy to ≤ Grade 1 (participants with ≤ Grade 2 neuropathy or endocrinopathies controlled by hormone replacement are eligible)
- Failure to recover from any other toxicity (other than immune-related toxicity) from previous anticancer treatment to ≤ Grade 2
- Known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days prior to trial treatment.


- Have a history of (noninfectious) pneumonitis that required steroids or have current pneumonitis (history of radiographically visible but asymptomatic radiation pneumonitis is allowed)
- Platelet count  $< 50 \times 10^9/L$
- Absolute neutrophil count  $< 1.0 \times 10^9/L$
- AST  $\geq$  3 × upper limit of normal (ULN), or if subject has known liver metastases, AST > 7 × ULN
- ALT  $\geq$  3 × ULN, or if subject has known liver metastases, ALT  $\geq$  7 × ULN
- Estimated creatinine clearance < 50 mL/min calculated by the Cockcroft Gault or Modification of Diet in Renal Disease formulas at screening
- Treatment with immunosuppressive therapy within 28 days of first dose of study drug
- History or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary, renal, metabolic, hematologic, or psychiatric) other than their primary malignancy that in the opinion of the Investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
- Treatment for any serious bacterial, viral, parasitic, or systemic fungal infections within the 30 days prior to study entry
- Active known or suspected COVID-19 disease
- Active known or suspected autoimmune disease (except that subjects are permitted to
  enroll if they have vitiligo; type 1 diabetes mellitus; residual hypothyroidism due to an
  autoimmune condition that is treatable with hormone replacement therapy only;
  psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed
  without systemic therapy; or arthritis that is managed without systemic therapy beyond
  oral acetaminophen and nonsteroidal anti-inflammatory drugs [NSAIDS])
- Positive test for HIV or hepatitis C antibodies
- Positive test for HBsAg or HBcAb (a subject whose HBsAg is negative and HBcAb is positive may be enrolled if an HBV DNA test is negative and either the subject is treated with potent antiviral therapy or is retested for HBsAg and HBV DNA every month)
- Subject is pregnant or breastfeeding, planning to become pregnant, or expecting to conceive or father children while enrolled in the study, up to the end of study (EOS) visit.
- Positive serum pregnancy test (ie, urine human chorionic gonadotropin) at screening


# 8.7. Additional Exclusion Criteria for Part B Cohorts: XmAb18087 in Combination with Pembrolizumab

In addition to the exclusion criteria in Section 8.6, subjects will be excluded from Part B safety run-in and expansion cohorts administered XmAb18087 in combination with pembrolizumab if they meet the following criteria:

- Prior treatment with therapeutics directed at anti-programmed cell death 1 (anti-PD1) or anti-programmed cell death ligand 1 (anti-PDL1)
- Have severe hypersensitivity ( $\geq$  Grade 3) to pembrolizumab and/or any of its excipients

## 8.8. Withdrawal of Subjects

Subjects must be withdrawn if the  $\beta$ -HCG pregnancy test is consistent with pregnancy. Before permanent discontinuation, the treatment may be interrupted to confirm the positive pregnancy test. Pregnancy should be reported as described in Section 11.1.4.2.

The Principal Investigator (PI) also has the right to withdraw subjects from the study at his/her discretion for any of the following reasons:

- Disease progression
- Occurrence of an unacceptable serious or non-serious AE
- Failure to return for follow-up
- Uncontrolled intercurrent illness unrelated to the disease under study that renders continuing treatment with XmAb18087 unsafe or regular study visits impossible
- Investigator decision
- Subject decision
- Death
- Administrative reasons

Subjects will be considered to have completed/ended participation in the study at the time that a subsequent anticancer therapy is administered.

Whenever possible, the Sponsor must be notified within 24 hours if a subject is withdrawn from the study. The reason(s) for a subject's discontinuation from the study are to be recorded in the source documents and the subject's electronic case report form (eCRF).

The EOT eCRF must be completed for all subjects who discontinue XmAb18087 permanently.

For subjects who discontinue prematurely, all assessments described for the EOT visit should be performed at the scheduled visit date, if at all possible. If this is not possible, all assessments should be performed as close to the scheduled dates as is practicable. Post-treatment evaluations should be completed no later than 4 weeks after the final administration of XmAb18087 and prior to initiation of a new treatment for malignancy.

Subjects who are withdrawn for any reason may not reenter this study. The Study Sponsor, Xencor, reserves the right to terminate this clinical study at any time and for any reason.


## 8.9. Other Subject Restrictions

#### 8.9.1. Avoidance of Pregnancy

Women are considered to be of childbearing potential unless there is a documented reason (ie, postmenopausal by history with no menses for 1 year and confirmed by FSH [using local reference ranges], OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy).

Women of childbearing potential must have a negative pregnancy test during screening and at Day 1 prior to study drug infusion and must use 1 highly effective method of birth control during the study and for 4 weeks following last dose of XmAb18087 or pembrolizumab (when applicable). Highly effective methods of birth control include combined hormonal birth control (oral, intravaginal, or transdermal), or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or intrauterine), IUDs, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner (provided partner is the sole sexual partner and there has been a medical assessment of surgical success), or sexual abstinence. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. Total abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. The Investigator is responsible for evaluating the reliability of the subject's ability to maintain sexual abstinence throughout the duration of the clinical trial.

Fertile male subjects must be willing to practice a highly effective method of birth control for the duration of the study and continuing for 4 weeks after the last dose of XmAb18087 or pembrolizumab (when applicable). Highly effective methods of birth control include vasectomy or a condom in combination with double-barrier methods, spermicide, hormonal birth control, or IUD (nonhormonal) used by the woman.

#### 8.9.2. Use in Nursing Women

It is unknown whether XmAb18087 or pembrolizumab are excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, participants who are breastfeeding are not eligible for enrollment.


#### 9. TREATMENT OF SUBJECTS

## 9.1. Identity of Study Treatments

XmAb18087 is a humanized bsAb that binds both CD3 and the tumor antigen SSTR2 to recruit cytotoxic T cells that will kill SSTR2<sup>+</sup> tumor cells. Intravenous Stabilization Solution is a concentrated form of the XmAb18087 buffer that minimizes protein binding to the administration equipment.



Prior to dilution, the vial containing parenteral drug product should be inspected visually. If particulate matter and/or discoloration are noted, drug should not be administered, and the Sponsor should be notified.

Pembrolizumab (Keytruda<sup>®</sup>) is an approved humanized mAb targeting the cell surface antigen PD1. It will be administered at the dose and schedule of 400 mg IV over 30 minutes every 6 weeks. It is supplied as a 100 mg per 4 mL (25 mg/mL) solution in a single-dose vial. Pembrolizumab is provided by sites as standard of care for advanced MCC.

# 9.2. Concomitant Therapy

All medications (including over-the-counter medications and herbals) and blood products that are administered within the 30 days prior to start of study treatment and throughout a subject's participation in the study until the post-treatment follow-up visit must be recorded in the source document and on the eCRF. Concomitant medications for other medical conditions are permitted as clinically indicated, subject to the specific requirements outlined in Section 7.9.1 and 7.9.2.

#### 9.2.1. Permitted Medications

Subjects who experience CRS should receive aggressive intervention and supportive measures as indicated. These may include, but are not limited to, epinephrine, antihistamines, corticosteroids, IV fluids, vasopressors, oxygen, bronchodilators, diphenhydramine, acetaminophen, and tocilizumab (see Section 11.3.3 or Appendix C for suggested management of infusion reactions, CRS, and neurologic toxicities).

Subjects who experience IRAE after pembrolizumab exposure should receive specific therapy in accordance with the guidelines in Table 18 and/or the NCCN guidelines for management of IRAEs (Appendix E)

In addition to required prophylactic medications, subjects may also receive the following additional therapy during the clinical trial:


 Antiemetics, antidiarrheals, anticholinergics, antispasmodics, antipyretics, antihistamines, analgesics, antibiotics, antihyperglycemics, and other medications intended to treat symptoms related to cancer, cancer therapy, or concurrent conditions. Other antitumor treatments may not be received.


- Antiviral treatments for subjects with a positive HBcAb (and negative HBV DNA test) at screening
- Transfusions of blood products such as red blood cells (RBCs) and platelets, if medically indicated
- Histamine receptor type 2 antagonists, or proton-pump inhibitors for treatment of indigestion, nausea, and/or vomiting
- Multivitamins, provided they be documented on the concomitant medications eCRF.
   No other vitamins or supplements will be permitted during this study without prior notification and approval of the Medical Monitor.

#### 9.2.2. Excluded Medications

Subjects may not concurrently receive other therapeutics for treatment of their malignancy. It is suggested that subjects not receive live prophylactic vaccinations while enrolled in the study.

## 9.3. Subject Compliance

The Sponsor or its designee will monitor the study according to GCP guidelines. All investigational therapy will be prepared and administered at the study site, and complete records of administration doses, times, durations, and supportive therapies will be kept.

Dosing will be performed by trained, qualified personnel designated by the PI. The date and time of dosing will be documented on each dosing day. Comments will be recorded if there are any deviations from the planned dosing procedures.

# 9.4. Blinding and Randomization of Study Treatment

No randomization or blinding is required for this open-label trial.

# 9.5. Procedure for Breaking the Randomization Code

Not applicable.

#### 10. STUDY DRUG MATERIALS AND MANAGEMENT

#### 10.1. XmAb18087

As of 27 April 2020, XmAb18087 has been given to 42 human subjects; hence, the safety profile associated with this agent is not well known and caution should be exercised as infusion reactions, CRS, allergic reactions, or other unexpected reactions may occur.

#### 10.1.1. Pretreatment of XmAb18087

Because administration of XmAb18087 has been associated with nausea and vomiting and has also been associated with symptoms of infusion reaction/CRS in subjects and a severe CRS reaction in 1 subject, prophylactic medications are to be administered to all subjects before at least the first

# 10.1.2. Prophylaxis of Nausea and Vomiting





are recommended for treatment of the symptoms.

Sites may also choose to use other or additional antinausea/vomiting medications for prophylaxis or treatment of symptoms, according to their practice and assessment of the subject's responses.

#### 10.1.3. Prophylaxis of Infusion Reactions/Cytokine Release Syndrome:

It is also required that all subjects receive the following medications before at least the first 4 doses the of study drug:

- a. Acetaminophen (Tylenol®): 650 mg PO once before dosing with XmAb18087
- b. Diphenhydramine (Benadryl®): 50 mg PO once before dosing with XmAb18087
- c. 10 to 20 mg IV dexamethasone (Decadron®) before dosing with XmAb18087

If a subject receives 4 consecutive doses of XmAb18087 without  $\geq$  Grade 1 infusion reaction or CRS, the prophylaxis described above may be modified, including elimination and/or reduced doses of some required medications.

For guidelines on the treatment of infusion reactions and CRS, see Section 11.2 or Appendix C of this protocol.

If at all possible, infusions of XmAb18087 should start before 2 PM local time. This is especially important for the C1D1 and any first dose at an escalated level to ensure that adequate staffing and services are available to manage a severe episode of CRS. In addition, either a Principal


Protocol XmAb18087-02

Investigator or subinvestigator (MD) must be readily available during, and for a minimum of 24 hours after, administration of an XmAb18087 dose.

#### 10.1.4. Administration of XmAb18087

XmAb18087 administration should begin as soon as possible after the dosing solution is made. If there is a delay in administration, it

The full-calculated dose will be

administered based on the subject's actual baseline weight measurement in kilograms. Following the first dose, subsequent doses will only be modified if the subject's weight changes by more than 10% from the Day -1 weight at which point it will be recalculated using the current weight.

# XmAb18087 should not be administered as an IV push or bolus.

Study drug will be administered as an open-label solution at a constant rate period. Precautions for CRS or infusion reactions or anaphylaxis should be observed during XmAb18087 administration. Due to the possibility that CRS, allergic reactions, or infusion reactions may occur, emergency resuscitation equipment (a "crash cart") and medications including steroids and tocilizumab should be present in the immediate area where subjects are receiving their infusions. Additional supportive measures should be available and may include, but are not limited to: acetaminophen, antihistamines, corticosteroids, IV fluids, bronchodilators, epinephrine, vasopressors, oxygen, and tocilizumab. Please refer to Section 11.3 or Appendix C for management of infusion reactions, CRS, and neurologic toxicities.

Vital signs will be measured and recorded as follows: immediately (within 60 minutes) prior to the infusion; during the infusion at 15, 30, and 60 minutes (± 5 minutes for each time point) from start time of the infusion; immediately (within 5 minutes) before EOI; and at 15, 30, and 60 minutes (± 5 minutes for each time point), then hourly (± 5 minutes) for a 3-hour period, after EOI. Oxygen saturation levels will be captured with each vital sign collection; however, pulse oximetry monitoring must be maintained continuously throughout the entire admission or observation period for each administration of XmAb18087. All supportive measures consistent with optimal subject care will be provided throughout the study according to institution standards. For subjects who a) tolerate 3 consecutive infusions without an infusion reaction during the observation period and b) have completed 4 infusions at the highest dose for that subject, the postinfusion observation period and vital signs assessment may be reduced from 4 hours to 2 hours.

# 10.2. Pembrolizumab (Keytruda®)

Pembrolizumab is an FDA-approved humanized monoclonal antibody that blocks the interaction between PD1 and its ligands, PDL1 and PDL2.

#### 10.2.1. Administration of Pembrolizumab

In dosing cohorts incorporating pembrolizumab (Part B only), pembrolizumab will be administered by IV infusion on Days 15 and 36 of each 42-day cycle. Pembrolizumab will be provided by sites as standard of care for advanced MCC.


Vital signs associated with the pembrolizumab infusion will be measured and recorded as follows: immediately prior (within 10 minutes before blood sampling) to the start of the infusion; during the infusion at 5 and 15 minutes ( $\pm$  2 minutes) from the start time of the infusion; immediately (within 2 minutes) before the EOI; and at 15 minutes ( $\pm$  2 minutes) after EOI. During Cycle 1, the subject will be observed for 4 hours after the infusion. On subsequent pembrolizumab administration days, the subject may be discharged 15 minutes postinfusion, if stable.

Pembrolizumab will be administered at a dose of 400 mg using a 30-minute IV infusion. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window between -5 minutes and +15 minutes is permitted (ie, infusion time is 30 minutes [-5 minutes/+15 minutes]). For additional information, refer to the pharmacy manual and the pembrolizumab prescribing information (Keytruda<sup>®</sup> Package Insert, 2020).

Pembrolizumab injection is a sterile, preservative-free, clear to slightly opalescent, colorless to slightly yellow solution that requires dilution for IV infusion. Each vial contains 100 mg of pembrolizumab in 4 mL of solution. Each 1 mL of solution contains 25 mg of pembrolizumab and is formulated in: L-histidine (1.55 mg), polysorbate 80 (0.2 mg), sucrose (70 mg), and Water for Injection, USP.

#### **10.2.2.** Treatment of Overdose

For this study, an overdose of pembrolizumab will be defined as any dose of 2000 mg or  $\geq 5 \times$  the indicated dose.

No specific information is available on the treatment of overdose of XmAb18087, or of pembrolizumab. In the event of overdose of either drug, the participant should be observed closely for signs of toxicity. Appropriate supportive treatment should be provided if clinically indicated.

# 10.3. Safety Criteria for Dose Adjustment or Stopping Dose

#### 10.3.1. Criteria for Adjustment or Stopping Dose of XmAb18087

Subjects experiencing a significant toxicity should be treated with standard medical interventions (eg, acetaminophen for fever) as appropriate.

For guidelines on management of infusion reactions/CRS/neurologic toxicity, and rules regarding study drug adjustment/discontinuation after an infusion reaction/CRS/neurologic toxicity, see Section 11.3.3 or Appendix C.

Subjects experiencing an AE that meets AESC criteria (as defined in Section 7.8 above) will have subsequent dosing held until recovery to baseline or ≤ Grade 2 following the AE. In the event that a > Grade 2 drug-related toxicity persists > 14 days and/or 2 consecutive doses are missed, the subject will be permanently discontinued from the study drug treatment. Subjects who experience the same AE that meets AESC criteria on 2 consecutive infusions will be subsequently treated at one dose level lower than the dose at which the AE occurred. Rechallenge with study drug is not permitted for any Grade 4 toxicity.


#### 10.3.2. Criteria for Adjustment or Stopping Dose of Pembrolizumab

Refer to Table 18 for dose modification and management guidelines for IRAEs related to pembrolizumab. Additional guidelines from the NCCN on the diagnosis and management of IRAEs can be found in Appendix E. Rechallenge with pembrolizumab is not permitted for the following:

- Any IRAE that requires permanent discontinuation of study drug according to the guidelines in Table 18.
- Any severe (Grade 3) or life-threatening (Grade 4) infusion-related reaction.

If it is determined that pembrolizumab must be permanently discontinued based on the above criteria, dosing with XmAb18087 must also be discontinued.

# 10.4. Study Treatment Packaging and Labelling

#### 10.4.1. Packaging and Labelling of XmAb18087

XmAb18087 and the IV Solution Stabilizer will be supplied in single-use glass vials.

XmAb18087 and the IV Solution Stabilizer will be supplied by Almac. IMPs will be packaged and labeled according to applicable local and regulatory requirements.

#### **10.4.2.** Storage of XmAb18087

Vials containing XmAb18087 and IV Solution Stabilizer must be stored under refrigeration at in an appropriately secured area accessible only to the pharmacist, the PI, or a duly designated person. Since XmAb18087 does not contain preservatives, opened vials of XmAb18087 must be used within 24 hours.

#### 10.4.3. Preparation of XmAb18087

Note that XmAb18087 has PD effects in vivo at very low concentrations and therefore each product vial must be highly diluted before administration.

Prior to administration, XmAb18087 will be diluted to the required final concentration in 1 or more ethylene/polypropylene copolymer infusion bags

. Prior to dilution, the vial containing parenteral drug product should be inspected visually. If particulate matter and/or discoloration are noted, drug should not be administered, and the Sponsor should be notified. After dilution, the bag containing XmAb18087 should be gently inverted 2 to 3 times to mix the solution. **THE BAG MUST NOT BE SHAKEN**; excess agitation may cause aggregate formation. See the XmAb18087 Pharmacy Manual for additional details.

#### 10.4.4. Packaging and Labeling of Pembrolizumab

Pembrolizumab will be obtained from commercial sources and administered to subjects in the combination therapy cohorts on Day 15 of each 42-day cycle as directed by the package insert (Keytruda® Package Insert, 2020).


Xencor, Inc

#### 10.4.5. Storage of Pembrolizumab

Store under refrigeration at 2 °C to 8 °C, do not freeze, do not shake, and protect from light, as per the pembrolizumab prescribing information (Keytruda® Package Insert, 2020).

# 10.5. Study Treatment Accountability, Handling, and Disposal

Detailed instructions and procedures for study-drug dispensing are included in the Pharmacy Manual.

Accurate accounting of all study drug must be maintained. The PI agrees to keep an inventory of study drugs using local investigational pharmacy drug accountability logs. Drug disposition records must be kept in compliance with applicable guidelines and regulations.

These records shall include dates, quantities, batch numbers, expiry dates, and the unique code numbers assigned to the study drug and to the study subjects.

The Investigator shall be responsible for ensuring records adequately document that the subjects were provided the doses specified in the protocol and that all study drug received from the Sponsor is reconciled.

Upon completion or termination of the study, any used or partially used vials, unused study medication, diluted drug dosing solutions, or IV Solution Stabilizer should be destroyed in compliance with local investigational pharmacy policies or returned to the Sponsor or its designee.


#### 11. ASSESSMENT OF SAFETY

Adverse event reporting will begin with the signing of the informed consent document (Screening) and will continue until the end of the subject's participation in the study: ie, until a subject has discontinued or completed the study.

Safety and tolerability assessments will include the following:

- AEs
- Vital signs
- PE findings
- Clinical laboratory safety assessments
- ECG parameters

Biomarkers of CRS (IL-2, IL-6, IL-8, IL-10, IFN- $\gamma$ , IL-13, IL-1B, and TNF- $\alpha$ ) will also be collected as additional safety information.

Details for management of hypersensitivity reactions, CRS, and neurologic toxicities are provided in Section 11.3.2, 11.3.3.3, and 11.3.3.4, respectively, as well as in Section 11.3.3 and Appendix C of this protocol.

#### 11.1. Adverse Events

#### 11.1.1. Definitions

#### 11.1.1.1. Adverse Event

An AE is any untoward medical occurrence in a study-subject administered IMP. The AE does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP. Adverse events may include the onset of new illness and the exacerbation of preexisting conditions.

Other untoward events occurring in the framework of a clinical study will be recorded as AEs, eg, those occurring during treatment-free periods (including Screening or post-treatment follow-up periods), in association with study-related procedures and assessments, or under placebo. For IMPs, lack of efficacy may be an expected potential outcome and should not be reported as an AE, unless the event is unusual in some way, eg, greater in severity.

Concomitant illnesses, which existed prior to entry into the clinical study, will not be considered AEs unless they worsen during the treatment period. Preexisting conditions will be recorded as part of the subject's medical history.

#### 11.1.1.1.2. Serious Adverse Event

AEs are classified as "serious" and "non-serious" for regulatory reporting purposes. The classification determines the procedures used to document and report the AE.


An SAE is an AE occurring during any study phase (ie, baseline, treatment, washout, or follow-up), and at any dose of the investigational product or comparator, that fulfills one or more of the following:

- Results in death
- Is life-threatening; this means that the subject was at immediate risk of death at the time of the event. It does not mean that the event hypothetically might have caused death if it were more severe.
- Requires inpatient hospitalization or prolongation in existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly or birth defect
- Is an important medical event. Important medical events are events that may not be immediately life threatening but are clearly of major clinical significance. They may jeopardize the patient and may require intervention to prevent one of the other serious outcomes listed above.

Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or in a physician's office, blood dyscrasias or seizures that do not result in subject hospitalization, and the development of drug dependency or drug abuse. Hospitalizations for planned surgical/medical elective procedures will not be reported as SAEs. In addition, hospitalizations of  $\leq$  24 hours will not be reported as SAEs. A death due to disease progress will not be considered an expedited report.

The following will **not** be reported as an SAE:

- Hospitalization for planned surgical/medical elective procedures per protocol for study drug administration, any admission required for disease assessments, or any admissions planned prior to enrollment (eg, planned surgical/medical elective procedures) will not be recorded/reported as an SAE.
- Hospitalization or death due to disease progression. Signs/symptoms and conditions related to disease progression of the primary condition under the investigation (eg, tumor-related pain, metastasis, new lesions, etc).

A distinction should be drawn between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria above. For example, a mild degree of gastrointestinal bleeding requiring hospitalization for monitoring purposes would be considered an SAE but is not necessarily severe. Similarly, an AE that is severe in intensity is not necessarily an SAE. For example, alopecia may be assessed as severe in intensity but would not be considered an SAE.

Medical and scientific judgment should be exercised in deciding if an AE is serious and if expedited reporting is appropriate.

#### 11.1.1.3. Abnormal Laboratory Values

Clinically significant abnormal laboratory results which are not caused by the underlying disease or are not consistent with the subject's medications will be recorded as AEs and the relationship


Protocol XmAb18087-02

Xencor, Inc

to the study drug will be indicated as below. Laboratory values outside the normal range will be assigned one of the following categories by the Investigator or designee:

- 1. Not clinically significant, minor out of range value or finding. AE No
- 2. Not clinically significant, out of range value or finding explainable by anticipated or known effect of study drug or concomitant drugs. AE No
- 3. Clinically significant but consistent with the subject's underlying disease. AE No
- 4. Clinically significant out of range value or finding. AE Yes

In general, a clinically significant laboratory value or finding would require some diagnostic or therapeutic intervention other than repeating the test.

# 11.1.2. Recording of Adverse Events

AEs should be collected and recorded for each subject from the date the ICF was signed until the end of their participation in the study, ie, the subject has discontinued or completed the study. All AEs experienced by a subject, irrespective of the suspected causality, will be monitored until the event has resolved or stabilized, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the Investigator and Sponsor medical representative, until there is a satisfactory explanation for the changes observed, or until the subject is lost to follow-up.

Any new SAEs that are suspected to be related to study drug occurring up to 28 days after the last administration of study drug should be reported to ICON according to Section 11.1.5. Adverse events may be volunteered spontaneously by the study subject, discovered by the study staff during physical examinations, or by asking an open, nonleading question such as "How have you been feeling since you were last asked?" All AEs and any required remedial action will be recorded. The nature of AE, date (and time, if known) of AE onset, date (and time, if known) of AE outcome to date, severity, and action taken with the study drug because of the AE will be documented together with the Investigator's assessment of the seriousness on the AE and causal relationship to study drug and/or study procedure.

All AEs should be recorded individually unless, in the opinion of the Investigator, the AEs constitute components of a recognized condition, disease, or syndrome. In the latter case, the condition, disease, or syndrome should be named rather than each individual symptom. The date (and time, if known) that the Investigator or study site is first made aware of the AE (or any subsequent follow-up information is received) will be documented. The AEs will be coded using the current version of the Medical Dictionary for Regulatory Activities (MedDRA).

Each AE will be assessed by the Investigator with regard to the categories discussed in the sections below.

#### 11.1.2.1. Intensity

The Investigator will assess all AEs for severity utilizing the NCI-CTCAE grading scale (Version 5.0). AEs not contained within CTCAE Version 5.0 will be rated on a five-point scale (Table 8):


**Table 8:** Severity Grading Scale

| Mild (Grade 1) | Mild events are those which are easily tolerated with no disruption of normal daily activity. |
|---|---|
| Moderate (Grade 2) | Moderate events are those which cause sufficient discomfort to interfere with daily activity. |
| Severe (Grade 3) | Severe events are those which incapacitate and prevent usual activity. |
| Life-threatening (Grade 4) | An adverse event that has life-threatening consequences, for which urgent intervention is indicated, that puts the subject at risk of death at the time of the event if immediate intervention is not undertaken, or that causes blindness or deafness. |
| Fatal (Grade 5) | The termination of life as a result of an adverse event. |


When changes in the intensity of an AE occur more frequently than once a day, the maximum intensity for the event should be noted for that day. Any change in severity of signs and symptoms over a number of days will be captured by recording a new AE, with the amended severity grade and the date (and time, if known) of the change.

## 11.1.2.2. Causality

The Investigator will assess the causality/relationship between the IMP and the AE. One of the following categories should be selected based on good medical and scientific judgment, considering the definitions in Table 9 and all contributing factors.


**Table 9: Causality Grading Scale** 

| Related | A clinical event, including laboratory test abnormality that occurs in a plausible time relationship to treatment administration, and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (dechallenge <sup>a</sup> ) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge <sup>b</sup> procedure if necessary. |
|---|---|
| Probably Related | A clinical event, including laboratory test abnormality, with a reasonable time sequence to administration of the treatment, unlikely to be attributed to concurrent disease or other drugs or chemicals, and which follows a clinically reasonable response on withdrawal (dechallenge). Rechallenge information is not required to fulfill this definition. |
| Possibly Related | A clinical event, including laboratory test abnormality, with a reasonable time sequence to administration of the treatment, but which could also be explained by concurrent disease or other drugs or chemicals. Information on treatment withdrawal may be lacking or unclear. |
| Unlikely Related | A clinical event, including laboratory test abnormality, with a temporal relationship to treatment administration that makes a causal relationship improbable, and in which other drugs, chemicals, or underlying disease provide plausible explanations. |
| Not Related | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative dechallenge and rechallenge information. Typically explained by extraneous factors (eg, concomitant disease, environmental factors, or other drugs or chemicals). |

AE = adverse event.

# 11.1.2.3. Action Taken with Study Treatment

Action taken with XmAb18087 (and pembrolizumab, when applicable) will be reported as one of the following:

- Dose not changed
- Dose reduced
- Drug interrupted
- Drug withdrawn
- Not applicable

#### 11.1.2.4. Outcome

Outcome will be defined as follows:

- Death related to adverse event
- Not recovered or not resolved


<sup>&</sup>lt;sup>a</sup> Dechallenge is when a drug suspected of causing an AE is discontinued. If the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation, this is termed a <u>positive dechallenge</u>. If the symptoms continue despite withdrawal of the drug, this is termed a <u>negative dechallenge</u>. Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug-relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).

b Rechallenge is when a drug suspected of causing an AE in a specific subject in the past is readministered to that subject. If the AE recurs upon exposure, this is termed a <u>positive rechallenge</u>. If the AE does not recur, this is termed a <u>negative rechallenge</u>.

- Recovered or resolved
- Recovered or resolved with sequelae
- Recovering or resolving
- Unknown

#### 11.1.3. Preidentified Immune-Mediated Adverse Events

See the pembrolizumab package insert (Keytruda<sup>®</sup> Package Insert, 2020) for a description of potential IRAEs. Guidelines for the management of IRAEs can be found in Table 18 and Appendix E.

#### 11.1.4. Adverse Events of Special Interest

IRAEs (Part B only) and infusion reactions (hypersensitivity reactions and CRS) are designated events of special interest in this protocol. Refer to Section 11.3.

#### 11.1.4.1. Deaths

Should a death occur within the study period or within 28 days after the last administration of study drug (or until the subject initiates other anticancer therapy, whichever comes first), an AE form and an SAE form should be completed, detailing the AE that resulted in the death (death is an outcome, not an event). The SAE must be reported to the Medical Monitor within 24 hours. The report should contain a comment regarding the coinvolvement of progression of disease, if appropriate, and should assign main and contributory causes of death.

#### **11.1.4.2. Pregnancy**

The teratogenic potential of XmAb18087 is unknown. Based on its mechanism of action, pembrolizumab can cause fetal harm when administered to a pregnant woman; however, there are no available human data informing the risk of embryo-fetal toxicity (Keytruda® Package Insert, 2020). The Investigator and Sponsor have a responsibility to monitor the outcome of all pregnancies, including pregnancies in female partners of male participants, reported during the clinical study.

Pregnancy alone is not regarded as an AE unless there is a suspicion that the IMP may have interfered with the effectiveness of a contraceptive medication. Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions (see below). Hospitalization for normal delivery of a healthy newborn should not be considered an SAE. All notifications of pregnancy should be documented and reported through 120 days following cessation of study treatment (or through 30 days following cessation of study treatment if the subject initiates new anticancer therapy), whether or not there is an associated AE or SAE.

Each pregnancy notification must be reported by the Investigator to the Sponsor and ICON within 24 hours after becoming aware of the pregnancy. The Investigator must follow-up and document the course and the outcome of all pregnancies even if the subject was withdrawn from the clinical study or if the clinical study has finished. The follow-up period will be deemed to have ended when the health status of the child has been determined on its birth.


All outcomes of pregnancy must be reported by the Investigator to the Sponsor and ICON on the pregnancy outcome report form within 24 hours after he/she has gained knowledge of the normal delivery or elective abortion, or other outcome.

Any SAE that occurs during pregnancy must be recorded on the SAE report form (eg, maternal serious complications, therapeutic abortion, ectopic pregnancy, stillbirth, neonatal death, congenital anomaly, birth defect) and reported within 24 hours of awareness in accordance with the procedure for reporting SAEs.

#### 11.1.5. Reporting Serious Adverse Events

The Investigator will review each potential SAE and evaluate the intensity and the causal relationship of the event to IMP. All potential SAEs will be recorded from signing of informed consent until the end of the subject's participation in the study: ie, the subject has discontinued or completed the study, except for the long-term follow-up period. During the long-term follow-up period, only SAEs that come to the attention of the Investigator and that the Investigator believes to have a reasonable causal relationship to the IMP will be reported.

The Investigator is responsible for reporting SAEs related to pembrolizumab to regulatory authorities per reporting guidelines.

The Investigator is responsible for providing notification to ICON of any potential SAE, whether deemed IMP-related or not, that a subject experiences during his/her participation in study within 24 hours of becoming aware of the event. ICON will provide the information to the Sponsor.

The initial SAE form should be completed and emailed to with the following information:

- Study number
- Subject number
- Gender
- Year of birth
- Name of PI and full clinical site address
- Name of the reporter
- SAE event term
- Details of SAE
- Criterion for classification as "serious"
- Study drug name, dose, and treatment start date
- Date of SAE onset
- Date of SAE first awareness (by Investigator or study site staff)
- Causality assessment


18 August 2020

ICON will request clarification of omitted or discrepant information from the initial notification. The Investigator or an authorized delegate is responsible for providing the requested information to ICON within 24 hours of the request.

Initial reports of SAEs must be followed up as soon as possible with detailed descriptions; this may include clear photocopies of other documents as necessary (eg, hospital reports, consultant reports, autopsy reports, etc.) with the study subject's personal identifiers removed. All relevant information obtained by the Investigator through review of these documents will be recorded and forwarded to ICON within 24 hours of receipt of the information.

If a new SAE report form for the same SAE is completed, then the Investigator must sign and date the SAE form and mark the form as "follow-up." ICON and/or the Sponsor may also request additional information on the SAE in order to obtain the full clinical picture, to which the PI or an authorized delegate must respond to ICON within 24 hours of the request.



- 1. E-mail your SAE form to the study specific e-mail address above.
- 2. Provide ICON with the name of the PI, your name, the telephone number where you can be reached and the protocol number and title.
- 3. Immediately forward the SAE form and any supporting documentation to ICON; this <u>must</u> be done within 24 hours of becoming aware of the event.

#### 11.1.6. Follow-up of Adverse Events

All AEs experienced by a subject, irrespective of the suspected causality, will be monitored until the event has resolved or stabilized, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the Investigator and Sponsor medical representative, until there is a satisfactory explanation for the changes observed, or until the subject is lost to follow-up.

#### 11.1.7. Treatment/Reporting of Overdose

In the event of an overdose, the physician should:

- Contact the Medical Monitor immediately
- Closely monitor the subject for any AE/SAE and laboratory abnormalities
- Obtain a plasma PK sample if requested by the Medical Monitor (determined on a case-by-case basis)
- Document the quantity and duration of the excess dose

Decisions regarding dose interruptions or modifications will be made by the Investigator in consultation with the Medical Monitor based on the clinical evaluation of the subject.


All overdose cases should be reported as SAEs.

# 11.2. Investigational New Drug Safety Reports

During the course of the study, the Sponsor may determine that certain safety reports are required to comply with regulations. The PI may receive a letter called an "Investigational New Drug (IND) Safety Report." These reports must be submitted to the IRB per local requirements as soon as possible, and documentation of this submission should be available to the Sponsor or ICON.

# 11.3. Guidelines for Prophylaxis and Management of Hypersensitivity Reactions, Cytokine Release Syndrome, and Neurological Toxicity Attributed to XmAb18087

Because administration of XmAb18087 has been associated with symptoms of infusion reaction/CRS in some subjects, it is required that all subjects receive the following medications before at least the first 4 doses of XmAb18087:

- a. Acetaminophen (Tylenol®): 650 mg PO once before dosing with XmAb18087
- b. Diphenhydramine (Benadryl®): 50 mg PO once before dosing with XmAb18087
- c. 10 to 20 mg IV dexamethasone (Decadron®) before dosing with XmAb18087

If a subject receives 4 consecutive doses of XmAb18087 without ≥ Grade 1 infusion reaction/CRS, the prophylaxis described above may be modified, prophylactic medications are to be administered to all subjects before at least the first 4 doses of the study drug.

#### 11.3.1. Introduction and Grading

Grading of toxicity, including allergic/hypersensitivity reactions, is by CTCAE version 5.0, except for CRS, which is graded using the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading (Lee, 2019) See Table 10 for these definitions.

All sites should review and implement the general guidelines for the use of tocilizumab and IV fluids discussed below in Sections 11.3.3.1 and 11.3.3.2. Otherwise, management of CRS and other infusion-related reactions should be per standard investigational site procedures. Or, if there are no local standards or if they are incomplete, the approaches discussed here may be used.




Table 10: American Society for Transplantation and Cellular Therapy Cytokine Release Syndrome Consensus Grading

| CRS Parameter | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Fever <sup>a</sup> | Temperature ≥ 38 °C | Temperature ≥ 38 °C | Temperature ≥ 38 °C | Temperature ≥ 38 °C |
| | | | With | |
| Hypotension | None | Not requiring vasopressors | Requiring a vasopressor with or without vasopressin | Requiring multiple<br>vasopressors<br>(excluding<br>vasopressin) |
| | | | And/or <sup>b</sup> | |
| Нурохіа | None | Requiring low-flow nasal cannula <sup>c</sup> or blow-by | Requiring high-flow<br>nasal cannula c,<br>facemask,<br>nonrebreather mask,<br>or Venturi mask | Requiring positive<br>pressure (eg, CPAP,<br>BiPAP, intubation<br>and mechanical<br>ventilation) |

BiPAP = bilevel positive airway pressure; CPAP = continuous positive airway pressure; CRS = cytokine release syndrome; CTCAE = Common Terminology Criteria for Adverse Events.

Organ toxicities associated with CRS may be graded according to CTCAE v5.0, but they do not influence CRS grading.

#### 11.3.2. Cytokine Release Syndrome Versus Allergic or Hypersensitivity Reactions

Cytokine release syndrome is mechanistically different from allergic/hypersensitive reactions (Lee, 2019), although some of the manifestations are common to both AEs and both have been reported to occur with therapeutic antibodies. An acute infusion reaction is often caused by a type 1 hypersensitivity mechanism due to immunoglobulin-E (IgE)-mediated release of histamines and prostaglandins, although a direct interaction with mast cells and basophils can also occur. It is less clear how cytokine release is triggered, although it is likely to be associated with immune cell activation; in this case, there is evidence that immunologic cascade is initiated by triggering of CD3-expressing T lymphocytes, resulting in TNF- $\alpha$  mediated monocyte/macrophage activation and systemic toxic cytokine release (Li, 2019).

Signs and symptoms usually develop during or shortly after drug infusion in hypersensitivity reactions, are more likely to occur after several doses of the drug and are largely related to histamine release. Typical signs and symptoms of hypersensitivity reaction include rash/urticaria, flushing, pruritus, fever, dyspnea, cough, and hypotension, although the following may also occur (Lenz, 2007):

Arthralgia


<sup>&</sup>lt;sup>a</sup> Fever is defined as temperature ≥ 38 °C not attributable to any other cause. In patients who have CRS then receive antipyretic or anticytokine therapy such as tocilizumab or steroids, fever is no longer required to grade subsequent CRS severity. In this case, CRS grading is driven by hypotension and/or hypoxia.

<sup>&</sup>lt;sup>b</sup> CRS grade is determined by the more severe event: hypotension or hypoxia not attributable to any other cause. For example, a patient with temperature of 39.5 °C, hypotension requiring 1 vasopressor, and hypoxia requiring low-flow nasal cannula is classified as grade 3 CRS.

<sup>&</sup>lt;sup>c</sup> Low-flow nasal cannula is defined as oxygen delivered at  $\leq$  6 L/minute. Low flow also includes blow-by oxygen delivery, sometimes used in pediatrics. High-flow nasal cannula is defined as oxygen delivered at  $\geq$  6 L/minute.

- Bronchospasm
- Confusion, mental status changes, and/or delirium
- Dizziness
- Fatigue (asthenia, lethargy, malaise)
- Hallucinations
- Headache
- Hypertension
- Myalgia
- Nausea and/or vomiting
- Rigors/chills
- Diaphoresis
- Tachycardia

Cytokine release syndrome, on the other hand, is more likely to occur after the first dose or first escalated dose of drug than after subsequent doses. It may begin somewhat later and is more likely to be associated with hepatic and neurologic complications, including the following:

- Any of the hypersensitivity signs or symptoms listed above
- Aphasia or word-finding difficulty
- Elevated d-dimer and/or hypofibrinogenemia
- Fatigue (asthenia, lethargy, malaise)
- Gait disturbance/dysmetria
- Hallucinations
- Seizures
- Transaminitis and/or hyperbilirubinemia
- Tremor

The Xencor Medical Monitor should be contacted immediately if questions arise concerning the grade and/or treatment of the infusion reaction.

#### 11.3.3. Treatment Guidelines for Cytokine Release Syndrome

#### 11.3.3.1. Use of Tocilizumab for Cytokine Release Syndrome

Tocilizumab is a therapeutic antibody that interferes with binding of IL-6 to the IL-6 receptor. It has been used to decrease the severity and possibly mortality of severe CRS (Frey, 2017), and early administration may be useful in improving outcomes. Below are suggested guidelines for its use:


- Sufficient tocilizumab (dose of 8 mg/kg) should be readily available to the area where subjects are receiving their infusions and being observed post infusion.
- Prompt tocilizumab therapy should be strongly considered if:
  - Oxygen saturation falls below 90% on room air, **OR**
  - Systolic blood pressure falls 20 mm Hg below predose measurements and below 100 mm Hg, **OR**
  - Temperature of > 38 °C (100.4 °F) in the presence of new or worsening dyspnea and/or tachypnea and/or rigors and/or tachycardia (heart rate [HR] > 110 bpm), OR
  - Early discovery of hepatic transaminase elevation. (Note that peak transaminase elevation appears to occur within 24 hours, so that it is unlikely that tocilizumab treatment on the day after study drug administration would affect the course or outcome in the absence of concurrent symptoms or signs of CRS).
- Repeat dosing of tocilizumab may be necessary if signs and symptoms persist or return after initial treatment.

#### 11.3.3.2. Fluid Management

Cytokine release syndrome is sometimes associated with myocardial dysfunction, pulmonary edema, or capillary leak syndrome (Shimabukuro-Vornhagen, 2018). Although there are little or no data regarding use of anti-CD3 antibodies and the need for fluid management, it seems prudent to monitor subjects for weight gain and limit IV fluid administration in the acute setting.

- If a subject is noted to have had a ≥ 10% increase in body weight over the previous 2 weeks in association with new or significantly increased bilateral lower extremity edema, dosing should be delayed until this finding is evaluated and, if indicated, treated.
- For acute hypotension, an IV fluid bolus should be limited to 500 mL of normal saline or the equivalent.
- If there is not an adequate response to fluids, treatment with tocilizumab (and vasopressors, if necessary) should be considered rather than additional fluid boluses.

#### 11.3.3.3. Cytokine Release Syndrome Treatment Guidelines by Grade

The following are treatment guidelines for XmAb18087 treatment-related infusion reactions (Lee, 2019); since it can be difficult to differentiate between different infusion reaction etiologies, both are included here.

#### Grade 1:

- Administer acetaminophen and/or diphenhydramine or dexamethasone to treat signs and symptoms if clinically indicated.
- Vital signs should be measured every 15 minutes or less as clinically indicated.
- Obtain a blood sample for cytokine analysis during the event and approximately 4 hours later, unless to scheduled cytokine monitoring is already in progress.


- Monitor the subject for worsening of condition; if severity of event increases to a higher grade, stop the infusion, administer appropriate treatment, and refer to guidelines below for more severe infusion reactions.
- It may be useful to premedicate the subject with acetaminophen and antihistamines prior to the next infusion.

#### Grade 2:

- Hypotension responsive to fluids or a low dose of a single pressor, or mild respiratory symptoms treatable with low-flow oxygen are signs of Grade 2 toxicity. Older subjects or those with significant comorbidities may be at higher risk of decompensation in this situation.
- **Discontinue the infusion** and administer acetaminophen and/or diphenhydramine or dexamethasone to treat signs and symptoms if clinically indicated. Once symptoms have resolved, slow the infusion rate by 50% of the baseline rate. If after 1 hour, the subject's symptoms do not return and vital signs are stable, the infusion rate may be increased every 30 minutes, as tolerated, to the baseline rate.
- Note that older subjects or those with significant comorbidities may be at higher risk of decompensation in this situation. When reactions occur in these vulnerable subjects, or in the case of rapidly escalating reactions, consider treatment with **tocilizumab** 4 to 8 mg/kg IV over 1 hour, with or without dexamethasone 10 to 20 mg IV (or equivalent).
- Vital signs should be measured every 15 minutes or less as clinically indicated. For subjects who are able to tolerate an increase in the infusion rate back to baseline and maintain normal blood pressure for 30 minutes after the rate increase then, at the discretion of the Investigator, the frequency of vital sign assessment may be reduced to every 30 minutes during the infusion.
- Obtain a blood sample for cytokine analysis during the event and approximately 4 hours later, in addition to scheduled cytokine monitoring if already in progress.
- Monitor the subject for worsening of condition; if severity of event increases to a higher grade, stop the infusion, administer appropriate treatment, and refer to guidelines below for Grades 3 and 4 infusion reactions.
- Subjects with maximum Grade 2 infusion reaction may continue on study and should receive prophylactic premedication with acetaminophen 650 mg PO and diphenhydramine hydrochloride 25 to 50 mg IV or PO prior to all subsequent XmAb18087 infusions.

#### Grade 3 and 4:

- Stop the infusion and disconnect the infusion tubing from the subject.
- Aggressive supportive care should be given immediately. Vasopressors, fluids, oxygen, epinephrine or bronchodilators, ventilatory support, antipyretics, and analgesics should be used as indicated.


- Treatment with tocilizumab 4 to 8 mg/kg IV over 1 hour with or without dexamethasone 10 mg IV (or equivalent) is strongly encouraged for CRS due to the high risk of progression and permanent organ dysfunction.
- Hospital admission for observations is almost always indicated, usually to an intensive care unit, since an initial appearance of improvement may quickly yield to rapid decompensation.
- Subjects with Grade 3 CRS or infusion reaction may be rechallenged once resolved. Subjects with recurrent Grade 3 or any Grade 4 infusion reaction should not receive further XmAb18087 treatment but will continue to be followed on the protocol (ie, for 4 weeks after last dose).
- Obtain a blood sample for cytokine analysis during the event and approximately 4 hours later, in addition to scheduled cytokine monitoring if already in progress.
- Obtain a sample for ADA testing as close to the onset of the event as possible, at the resolution of the event, and 28 days following the event.
- Notify the Xencor Safety Monitor or Xencor Medical Monitor, (Telephone: ; Email: ), immediately.

#### 11.3.3.4. Neurotoxicity

In addition to CRS, another toxicity observed after chimeric antigen receptor T cell (CAR-T) therapy and CD3 bispecific antibodies is neurotoxicity. Immune effector cell-associated neurotoxicity syndrome (ICANS) may manifest as delirium, encephalopathy, aphasia, lethargy, difficulty concentrating, agitation, tremor, seizures, and, rarely, cerebral edema (Lee, 2019). Neurotoxicity was previously considered in aggregate with CRS, but is now treated separately, due to its timing and response to treatment.

Neurologic symptoms may occur during or after CRS symptoms, but rarely precede CRS symptoms. The earliest manifestations of ICANS are tremor, dysgraphia, mild difficulty with expressive speech (especially in naming objects), impaired attention, apraxia, and mild lethargy. Headache is a nonspecific symptom, frequently occurring during fever or after chemotherapy in patients without other neurologic dysfunction. Thus, headache alone is not a useful marker of ICANS. Expressive aphasia, on the other hand, appears to be a very specific symptom of ICANS (Lee, 2019).

A consensus grading scheme, which is a slightly modified version of the CARTOX-10 screening tool, which incorporated key elements of the Mini-mental State Examination (MMSE), the Immune Effector Cell-Associated Encephalopathy (ICE) score, will be used for the grading of ICANS (Table 9). It is important to note that the 10-point ICE screening tool is helpful for assessing patients for encephalopathy; however, the grading of ICANS requires assessment of the 10-point ICE score as well as evaluation of other neurologic domains, such as level of consciousness, motor symptoms, seizures, and signs of elevated ICP/cerebral edema, which may occur with or without encephalopathy. The ASTCT ICANS toxicity grading system is shown in Table 10. This grading scale will be used to assess neurotoxicity, rather than the CTCAE 5.0.


#### Table 11: Immune Effector Cell-associated Encephalopathy Scoring

#### **ICE**

Orientation: orientation to year, month, city, hospital: 4 points

Naming: ability to name 3 objects (eg, point to clock, pen, button): 3 points

**Following commands:** ability to follow simple commands (eg, "Show me 2 fingers" or "Close your eyes and stick out your tongue"): 1 point

Writing: ability to write a standard sentence (eg, "Our national bird is the bald eagle"): 1 point

Attention: ability to count backwards from 100 by 10: 1 point

ICANS = immune effector cell-associated neurotoxicity syndrome; ICE = Immune Effector Cell-Associated Encephalopathy (score).

Scoring: 10, no impairment;

- 7 9, Grade 1 ICANS;
- 3 6, Grade 2 ICANS;
- 0 2, Grade 3 ICANS;

0 due to patient unarousable and unable to perform ICE assessment, Grade 4 ICANS (Lee, 2019).


| Neurotoxicity<br>Domain | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| ICE score <sup>a</sup> | 7 - 9 | 3 - 6 | 0-2 | 0 (patient is<br>unarousable and<br>unable to perform<br>ICE) |
| Depressed level of consciousness <sup>b</sup> | Awakens<br>spontaneously | Awakens to voice | Awakens only to tactile stimulus | Patient is<br>unarousable or<br>requires vigorous or<br>repetitive tactile<br>stimuli to arouse.<br>Stupor or coma |
| Seizure | N/A | N/A | Any clinical seizure focal or generalized that resolves rapidly or nonconvulsive seizures on EEG that resolve with intervention | Life-threatening prolonged seizure (> 5 min); or Repetitive clinical or electrical seizures without return to baseline in between |
| Motor findings <sup>c</sup> | N/A | N/A | N/A | Deep focal motor<br>weakness such as<br>hemiparesis or<br>paraparesis |
| Elevated<br>ICP/cerebral edema | N/A | N/A | Focal/local edema on neuroimaging <sup>d</sup> | Diffuse cerebral edema on neuroimaging; decerebrate or decorticate posturing; or cranial nerve VI palsy; or papilledema; or Cushing's triad |

EEG = electroencephalogram; ICANS = immune effector cell-associated neurotoxicity syndrome; ICE = Immune Effector Cell-Associated Encephalopathy (score); ICP = intracranial pressure; N/A = not applicable; VI = sixth.

ICANS grade is determined by the most severe event (ICE score, level of consciousness, seizure, motor findings, raised ICP/cerebral edema) not attributable to any other cause; for example, a patient with an ICE score of 3 who has a generalized seizure is classified as grade 3 ICANS.

It has been speculated that high levels of IL-6 may directly mediate neurotoxicity in this situation (Lee, 2014).


<sup>&</sup>lt;sup>a</sup> A patient with an ICE score of 0 may be classified as Grade 3 ICANS if awake with global aphasia, but a patient with an ICE score of 0 may be classified as Grade 4.

<sup>&</sup>lt;sup>b</sup> Depressed level of consciousness should be attributable to no other cause (eg, no sedating medication).

<sup>&</sup>lt;sup>c</sup> Tremors and myoclonus associated with immune effector cell therapies may be graded according to CTCAE v5.0, but they do not influence ICANS grading.

<sup>&</sup>lt;sup>d</sup> Intracranial hemorrhage with or without associated edema is not considered a neurotoxicity feature and is excluded from ICANS grading. It may be graded according to CTCAE v5.0 (Lee, 2019).

Clinical management of neurotoxicity consists of the following:

- Monitor subjects closely for signs and symptoms of these events (including administration of mental status and neurologic examinations when these seem clinically warranted).
- If neurotoxicity becomes evident, a blood sample for cytokine analysis should be drawn at that time, and again 4 hours later, in addition to scheduled cytokine monitoring if already in progress.
- If neurologic toxicity is Grade 4, discontinue XmAb18087, if still infusing.
- For Grade 3 neurologic toxicity, withhold both drugs until the toxicity has recovered to ≤ Grade 1 (mild) and has remained at ≤ Grade 1 for at least 3 days before restarting therapy. Restart XmAb18087 at 75% of the previous dose. Restart pembrolizumab at the full dose. Escalate back to full dose at the time of the next dose if ≥ Grade 2 toxicity does not recur. If ≥ Grade 2 toxicity reoccurs at 75% dose, or if < Grade 2 toxicity takes more than 7 days to resolve, discontinue permanently.
- For severe neurologic symptoms, administer additional dexamethasone 10 mg intravenously and repeat every 12 hours if symptoms do not abate rapidly, or treat according to the clinical site's institutional protocol for such reactions.
- For recurrent seizures, anticonvulsant therapy may be necessary.

# 11.4. Guidelines for Prophylaxis and Management of Infusion Reactions Attributed to Pembrolizumab

Pembrolizumab may cause severe or life-threatening infusion reactions, including severe hypersensitivity or anaphylaxis. Refer to the pembrolizumab prescribing information (Keytruda® Package Insert, 2020) for diagnosis, management, prophylaxis, and dose modification for infusion-related reactions related to pembrolizumab administration.

# 11.5. Laboratory Assessments

Safety clinical laboratory assessments will be performed by ICON Central Labs. Specified predosing safety laboratory assessments will also be performed by clinical site local laboratories so that site personnel are able to review the results before administering XmAb18087. In addition, investigators may also perform locally any laboratory assessments that they feel are necessary to protect subject safety.

Blood samples should be taken using standard venipuncture techniques. Blood sampling will be performed according to site or laboratory standard operating procedures (SOPs).

Unless otherwise prescribed within this clinical protocol, assessments during Cycle 1 Days 1, 8, and 15 should be completed  $\pm$  1 hour of the scheduled time; for other days during Cycle 1  $\pm$  3 hours; and for subsequent cycles and within  $\pm$  2 days of the scheduled day. Disease assessments by RECIST and by radionuclide imaging should be performed within  $\pm$  2 days of the scheduled day. Imaging will be collected and stored for potential central assessment at a later date. Details for laboratory assessments, PK, PD, flow cytometry, and biobanking are provided in the Laboratory Manual.


The following laboratory variables will be determined as outlined below:

**Hematology:** RBC, hemoglobin, erythrocyte mean corpuscular volume, RBC distribution width, white blood cell (WBC) with differential (percent and absolute; neutrophils, lymphocytes, monocytes, eosinophils, basophils, and nucleated RBCs), and platelet count.

**Coagulation panel**: prothrombin time/international normalized ratio and activated partial thromboplastin time.

Clinical chemistry: Chemistry panel (sodium, chloride, potassium, bicarbonate, blood urea nitrogen, creatinine, glucose, uric acid, calcium, phosphorous, total bilirubin, ALT, AST, total protein, albumin, alkaline phosphatase, and lactate dehydrogenase), serum gamma-glutamyl transpeptidase, amylase, and lipase.

**Urinalysis**: pH, specific gravity, ketones, leukocyte esterase, bilirubin, blood protein, RBCs, WBCs, hyaline casts, RBC casts, WBC casts, granular casts, waxy casts, broad casts, and fatty casts.

**Pregnancy test**: Serum β-hCG pregnancy test for women of childbearing potential or FSH for postmenopausal women.

# 11.6. Electrocardiogram Assessments

The timing of ECGs is noted in Table 7. On all dosing days in Cycle 1 and selected dosing days in cycles after Cycle 1, supine ECGs will be performed predose.

The 12-lead ECGs will be performed after the subject has been resting supine for  $\geq 5$  minutes. The ECG will include all 12 standard leads. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QTc interval.

All ECGs must be evaluated by a qualified physician for the presence of abnormalities.

# 11.7. Physical Examination

Complete or abbreviated (symptom-directed) PEs will be performed as indicated in Table 7.

The complete PE includes an assessment of general appearance and a review of systems (dermatologic, head, eyes, ears, nose, mouth/throat/neck, thyroid, lymph nodes, respiratory, cardiovascular, gastrointestinal, extremities, musculoskeletal, neurologic, and psychiatric systems).

An abbreviated PE is symptom-directed and need not include detailed examination of all systems.

# 11.8. Vital Signs

Vital signs will be assessed at as indicated in Table 7. All vital signs should be taken with the subject in the same position. On nondosing days, vital signs should be measured prior to blood sampling. The following vital signs will be measured:

- Blood pressure (systolic and diastolic [mmHg])
- Heart rate (beats per minute [bpm])
- Respiratory rate (breaths per minute)


- Body temperature (°C)
- Supine BP and heart rate recordings will be made after the study subject has been recumbent and at rest  $\geq 5$  minutes
- Blood oxygen saturation by pulse oximetry. Oxygen saturation levels will be captured at each vital sign collection; however, pulse oximetry monitoring must be maintained continuously throughout the entire admission or observation period for each administration of XmAb18087.


#### 12. ASSESSMENT OF EFFICACY

Radiographic tumor evaluation will be performed at baseline and at all other disease assessment time points per RECIST 1.1 criteria (Appendix A). If additional clarification or detail is needed, please consult the literature referenced or the Sponsor's Medical Monitor.

The timing for these evaluations will be uniform. Initial evaluation will occur within 14 days (60 days for NETSPOT® gallium 68 dotatate PET/CT) before administration of the first dose of XmAb18087, and follow-up evaluation will be performed on Cycle 1 Day  $40 \pm 2$  days. Reevaluation will be performed after every cycle, as long as the subject continues on study, and at EOT. NETSPOT® gallium 68 dotatate PET/CT scan will be performed and interpreted locally. Copies of images and reports will be collected and sent to Xencor, Inc., for interpretation and archiving. Scans used for RECIST assessments will be performed and interpreted locally. Copies of these images will be collected and stored for potential central assessment at a later date.

#### 13. PHARMACOKINETIC/PHARMACODYNAMIC ASSESSMENTS

# 13.1. Serum Sampling for Pharmacokinetic Analyses, Anti-drug Antibodies, Cytokines, and Inflammatory Factors

The Sponsor or designee will provide cryotubes, labels, and requisition forms. Serum cryotubes will be labeled at the clinical site with the subject number, date, visit day and time point, and time of sampling. Samples will be stored on site at -70 °C until the Sponsor notifies the sites to ship the samples on dry ice to the designated laboratory for sample analysis. Detailed instructions for processing and shipping serum samples are provided in the Laboratory Manual. Venous blood samples for serum analyses of PK, ADA, and the cytokine and inflammation panel will be obtained according to the Schedule of Assessments (Table 7).

#### 13.2. Pharmacokinetics

Samples for PK analysis will be collected at the times specified in the Schedule of Assessments (Table 7). The exact time and date of the blood draw must be accurately recorded using an unambiguous format such as DD MON YYYY and HH:MM on a 24-hour clock. Missed samples will be considered protocol deviations.

# 13.3. Pharmacodynamics

Baseline and serial assessment of B-cell, NK-cell, and T-cell numbers and T-cell activation will be assessed in peripheral venous blood. The Sponsor/designated vendor will provide blood sampling tubes, label, requisition forms, and shipping containers. Samples for flow cytometry should be shipped immediately at ambient temperature. Detailed instructions for processing and shipping flow cytometry samples are provided in the Laboratory Manual. For the sampling schedules, see the Schedule of Assessments (Table 7).

Antibodies to MCPyV tumor antigens will be measured at baseline and end of treatment. Refer to the Laboratory Manual for instructions on sample procurement, processing, and shipping.


Formalin-fixed paraffinized archival tumor samples and optional fresh tumor biopsies will be assessed by immunohistochemistry for tumor cell SSTR2 expression and immune cell expression of proliferation, exhaustion, and other markers and for transcriptomics by Nanostring.

# 13.4. Biobanking Samples

Additional exploratory genetic, cellular, and/or serum markers of potential future interest may be explored if evidence of therapeutic activity is seen with XmAb18087. For biobanking, blood obtained for flow cytometry will be sent to Navigate BioPharma, where serum, PBMCs, and extracted nucleic acid will be aliquoted and stored at -70 °C. Biobanking is voluntary and requires specific subject consent.


#### 14. STATISTICAL EVALUATION

# 14.1. Sample Size and Power

This study is being performed in 3 parts: MCC monotherapy (Part A), MCC combination therapy (Part B), and SCLC monotherapy (Part C). No formal power analyses were performed for efficacy endpoints for the initial dose escalation cohorts. After identification of each RD, Part A, Part B, and Part C will enroll expansion cohorts using a 2-stage design (Schultz, 1973).

In Part A, up to 9 subjects will be enrolled at the RD. If at least 1 subject shows a response by RECIST 1.1 criteria, then enrollment will continue up to a total of 22 subjects. A true response rate of 40% has statistical power of 84% to rule out a lower inactivity rate of 16% with a one-sided Type I error rate of 5%.

In Part B, up to 12 subjects will be enrolled at the RD. If at least 4 subjects show a response by RECIST 1.1 criteria, enrollment will continue up to a total of 30 subjects. A true response rate of 67% has statistical power of 84% to rule out a lower inactivity rate of 43% with a one-sided Type I error rate of 5%.

In Part C, up to 9 subjects will be enrolled at the RD. If at least 1 subject shows a response by RECIST 1.1 criteria, then enrollment will continue up to a total of 30 subjects.

Subjects who are not evaluable may be replaced. Up to 142 subjects will be enrolled. The total number of subjects enrolled will depend upon the number of safety run-in cohorts required to identify the RD for each Part. A true response rate of 30% has statistical power of 82% to rule out a lower inactivity rate of 11% with a one-sided Type I error rate of 5%.

#### 14.2. Statistical Methods

Before database lock, a statistical analysis plan (SAP) will be issued as a separate document, providing detailed methods for the analyses outlined below. Any deviations from the planned analyses will be described and justified in the final integrated clinical study report.

Unless otherwise specified, continuous variables will be summarized with N (ie, sample size), mean, median, standard deviation, minimum and maximum, and discrete variables will be summarized with frequencies and percentages. Safety and efficacy summaries will be performed for Parts A, B, and C separately and, for safety, also for the combined arms. For each Part, summary tables will be provided for each dose cohort and for the dose cohorts combined.

# 14.3. Study Endpoints

#### 14.3.1. Primary Endpoints

The primary endpoints are as follows:

- Safety of (1) XmAb18087 monotherapy in MCC and SCLC, and (2) XmAb18087 and pembrolizumab combination therapy in MCC, as assessed by the following:
  - Incidence of treatment-emergent AEs (TEAEs)
  - Incidence of clinically significant changes in safety laboratory tests, PE findings, vital signs, and ECGs


- Incidence and severity of CRS
- Efficacy of (1) XmAb18087 monotherapy in MCC and SCLC, and (2) XmAb18087 and pembrolizumab combination therapy in MCC using RECIST 1.1 assessment of CT/MRI imaging, as well as aggregate data, for the following:
  - ORR
  - CR rate
  - PR rate

#### 14.3.2. Secondary Endpoints

The secondary endpoints are as follows:

- Efficacy of (1) XmAb18087 monotherapy in MCC and SCLC, and (2) XmAb18087 and pembrolizumab combination therapy in MCC using RECIST 1.1 assessment of CT/MRI imaging, as well as aggregate data, for the following:
  - Duration of response
  - PFS
  - OS
- PK characterization of XmAb18087, when administered as monotherapy and in combination with pembrolizumab, based on the parameters of C<sub>max</sub>, time to reach maximum concentration (t<sub>max</sub>), half-life (t<sub>1/2</sub>), area under the serum concentration-time curve from time zero to infinity (AUC<sub>0-∞</sub>), clearance (CL), volume of distribution (Vd), and volume of distribution at steady state (Vd<sub>ss</sub>). Further details will be defined in a PK analysis plan.
- Assessment of immunogenicity by incidence of anti-XmAb18087 antibodies and qualitative assessment of safety outcomes
- PK characterization of pembrolizumab, when administered in combination with XmAb18087, based on parameters similar to those for XmAb18087, with further details to be provided in a PK analysis plan.

#### 14.3.3. Exploratory Endpoints

The exploratory endpoints are as follows:

- Assessment of peripheral blood for cell surface markers by flow cytometry and similar bioanalytical methods that evaluate the response of selected immune system cells following administration of XmAb18087 as a monotherapy and in combination with pembrolizumab, including changes in lymphocyte subsets and in T-cell activation and exhaustion markers
- PD characterized by NETSPOT (gallium 68 dotatate) PET/CT results and by tumor-cell expression of SSTR2 and PDL1 and tumor-infiltrating immune-cell expression of PD1/PDL1 and other markers by immunohistochemistry, in response to administration of XmAb18087 monotherapy and in combination with pembrolizumab


- PD: IHC SSTR2 panel
- PD: MCC and SCLC IHC panels
- Correlation of clinical/radiographic response with MCPyV serology (MCC subjects only)
- Additional exploratory genetic, cellular, and/or serum markers of potential future interest. If evidence of therapeutic activity is seen with XmAb18087, biobanked samples may be assessed for genetic and immunologic factors that might predict response or nonresponse (optional part of study and may be reported separately from the clinical study report). Samples will not be retained for more than 15 years.

# 14.4. Analysis Populations

The populations defined below will be used for analysis:

- **Safety population**: All subjects who are enrolled and receive at least 1 infusion of XmAb18087.
- Evaluable population: All subjects who are enrolled, receive at least 1 cycle (Parts A and C: 6 doses XmAb18087, Part B: 5 doses XmAb18087 and 1 dose pembrolizumab) of XmAb18087 and have at least 1 postbaseline RECIST 1.1 assessment of tumor imaging available.
- **PD population**: All subjects who are enrolled, receive at least 1 dose of XmAb18087 (and 1 infusion of pembrolizumab, when relevant for a particular PD assessment), and have at least 1 preinfusion and 1 postinfusion set of biomarker data available for analysis.
- **PK populations**: All subjects who are enrolled and receive at least 1 dose of XmAb18087 (ie, the XmAb18087 PK population) or 1 infusion of pembrolizumab (ie, the pembrolizumab PK population), and have at least 1 set of postinfusion PK data available for analysis.

Continuous data will be presented using descriptive statistics: number of subjects (N), mean, standard deviation, median, minimum, and maximum. Categorical data will be summarized by the number and percentage, where the percentage is presented in brackets to 1 decimal place. Safety and efficacy summaries will be provided for the monotherapy and combination therapy arms separately, as well as for the combined arms.

# 14.5. Subject Characteristics and Disposition

The SAP will define analysis parameters for the study and takes precedence over this protocol section.

Demographic (age, gender, ethnic origin, race) and baseline characteristics (eg, height, weight, body mass index, ECOG performance status, etc.) will be summarized, as will disease-related characteristics (including any available genetic data), prior anticancer therapy, and relevant supportive care therapies.

A summary of subject disposition will include the following:


- Number of subjects enrolled
- Number of subjects who received treatment
- Number of subjects who complete the study treatment (1 cycle)
- Number of subjects who terminated treatment and reason for discontinuation of treatment
- Number of subjects who complete 6-month and 12-month follow-up period
- Number of subjects who terminated study and reasons for study terminations

# 14.6. Safety Assessment

Safety variables will include AEs, PE findings, vital signs, ECGs, and laboratory values.

The extent of exposure to XmAb18087 monotherapy, as well as exposure in combination with pembrolizumab, will be summarized by dose cohort based on the number of infusions administered and the number of treatment cycles completed, as well as the total dose received. Additional summaries of drug exposure will be provided based on the PK parameters described in Section 13. Reasons for missed infusions or early permanent discontinuation of XmAb18087 will be reported.

Summary tables and listings will be provided for all reported AESC.

Adverse events will be coded using the latest version of MedDRA. The verbatim term recorded by the Investigator will be mapped to System Organ Class (SOC) and Preferred Term using MedDRA.

Treatment-emergent AEs are defined as events with onset dates on or after the start of study treatment or events that are present before the first infusion of XmAb18087 and subsequently worsen in severity.

Adverse-event-related endpoints include the following:

- TEAEs
- Treatment-emergent SAEs (TESAEs)
- Treatment-related TEAEs (for XmAb18087 or for pembrolizumab, if they can be distinguished)
- Treatment-related TESAEs (for XmAb18087 or for pembrolizumab, if they can be distinguished)
- TEAEs by severity that are defined by NCI-CTCAE, Version 5.0
- TEAEs resulting in the permanent discontinuation of XmAb18087 and/or pembrolizumab.

All AE-related endpoints will be summarized by MedDRA SOC and preferred term. At each level of summation, subject will be counted once under the greatest severity and strongest study drug relationship. All AEs will be included in the listings.

The hematology, chemistry, and other laboratory values and change from baseline values will be summarized descriptively for each scheduled assessment time point and grouped by dosing cohort. The baseline value for each laboratory value is defined as the last assessment performed on or prior


to the date of first dose of study treatment. The toxicity grades for laboratory tests will be based on NCI-CTCAE Version 5.0 criteria. The use of blood transfusions (platelets, RBCs) and/or growth factor support will be reported. Similar analyses will be done for chemistry tests (including liver and renal function tests). Subject listings of all laboratory data collected during the study will be presented. Laboratory values outside normal limits will be identified in the subject listings and will include flags for high and low values.

Vital sign results (blood pressure, pulse, respirations, temperature, and blood oxygen saturation by pulse oximetry) and change from baseline values will be summarized descriptively for each scheduled time point. The baseline value for each vital sign measurement is defined as the last assessment performed on or prior to the date of first dose of study treatment. Additionally, the vital signs measured immediately (within 60 minutes) before each infusion of XmAb18087; at 15, 30, and 60 minutes from the start of the infusion (± 5 minutes for each time point); immediately (within 5 minutes) before EOI; at 15, 30, and 60 minutes after the EOI (± 5 minutes for each time point); and then hourly (± 5 minutes) for 3 hours postinfusion will be summarized. The change of vital signs values from preinfusion will be summarized for each postinfusion point. Preinfusion assessments are defined as last vital assessment prior to the same infusion. Subject listings of all vital data collected during the study will be presented.

Electrocardiogram values and change from baseline values will be summarized descriptively for each scheduled time point. Subject listings of all ECG data collected during the study will be presented.

# 14.7. Efficacy Assessment

The objective of these analyses is to explore the effects of XmAb18087 when administered repeatedly as a single agent across a range of dose levels, in combination with pembrolizumab, and at RD for each Part of the study.

The assessment of antitumor effects of XmAb18087 will be based on response criteria defined in RECIST 1.1 (Appendix A).

The number and percentage of subjects achieving a best overall response of complete response (CR; confirmed and unconfirmed), partial response (PR; confirmed and unconfirmed), stable disease, progressive disease, and not evaluable will be presented.

Overall response rate is defined as subject's best response of PR or better. The number and percent of subjects who achieved ORR will be summarized. Two-sided exact 95% confidence intervals for the ORR will be determined using the binomial distribution. The duration of objective response will be calculated from the time of initial response (PR or better) to the first documentation of relapse (recurrence after CR) or progression (after PR).

The evaluable population defined in Section 14.4 will be used for summary of ORRs and duration of response.

Depending on the completeness of the available follow-up data, an analysis of PFS, measured relative to Day 1, will be performed based on the Kaplan-Meier method. Median time and its 95% confidence interval, as well as the 25<sup>th</sup> and 75<sup>th</sup> quartiles with their 95% confidence intervals, will be summarized. Progression will be determined using the criteria described in RECIST 1.1 (Appendix A). The date of progression is defined as the date of progression or death.


The date of censoring for subjects who end the study without documented progression will correspond to the date the last tumor assessment was performed. Subjects who terminated from study without postbaseline tumor assessment will be censored at Day 1.

Progression-free survival will be presented based on the safety population for the overall study.

The potential antitumor effects of XmAb18087 may also be evaluated in other subgroups of subjects. The specifications for these and other similar analyses will be described in the SAP and supersedes any protocol specifications.

# 14.8. Pharmacokinetic Analysis

Pharmacokinetic parameters including  $C_{max}$ ,  $t_{max}$ ,  $t_{1/2}$ ,  $AUC_{0-\infty}$ , CL, Vd, and  $Vd_{ss}$  will be estimated using either noncompartmental or compartmental methods, whichever best describes the observed data. Pharmacokinetic parameters for XmAb18087 will be compared with and without pembrolizumab administration.

Pharmacokinetic parameters at presumed steady-state will include area under the serum concentration-time curve during a dosing interval (t;  $AUC_t$ ; where t is 1 week), steady-state concentration ( $C_{ss}$ ), minimum steady-state concentration ( $C_{min,ss}$ ), steady-state fluctuation in concentrations (%Fluct), time of minimum concentration ( $t_{min}$ ) and predicted accumulation (accumulation index, AI). The observed accumulation will be computed as the ratio of  $C_{max}$  and  $AUC_t$  at presumed steady state versus  $C_{max}$  and  $AUC_t$  after the first dose. Trough concentrations ( $C_{trough}$ ) at predose will be used to evaluate the approach to steady state.

All PK parameters will be computed using actual elapsed time to PK sampling event and to dose event start and stop, calculated relative to the first dose start of infusion and the dose start for each infusion. Dose used to compute PK parameters will be the actual dose delivered during the infusion duration.

Dose proportionality across dose levels will be characterized by plotting  $C_{max}$  and  $AUC_{0-\infty}$  and  $AUC_{t}$  versus dose. Similarly, the kinetic parameters  $t_{1/2}$ ,  $t_{max}$ , CL, Vd, and  $Vd_{ss}$  across dose levels will be characterized by plots of these parameters versus dose.

Exploratory analyses may be performed to evaluate the relationship between 1 or more of the estimated PK parameters and selected safety, efficacy, and other serum protein assessment parameters described previously. The serum profile of XmAb18087 versus time will be evaluated with respect to any antibodies to XmAb18087 that may accelerate clearance.

A similar analysis of Pembrolizumab PK will be performed and details of both analyses will be described in a PK Analysis Plan.

# 14.9. Immunogenicity Assays

The incidence and titer of anti-XmAb18087 ADA will be reported by dose cohort and sample collection time point.


#### 15. DIRECT ACCESS TO SOURCE DATA/NOTES

The Investigator or institution shall provide direct access to source data and documents for study-related monitoring, audits, IRB/Independent Ethics Committee (IEC) review, and regulatory inspection.


The Sponsor or its designee will monitor the study according to GCP guidelines. The PI and study center will permit the Sponsor, its representatives, FDA, and other regulatory agencies direct access to all original source data and documents for study monitoring audits and inspections. All requested information must be entered into the eCRF in the EDC database. The completed eCRF must be promptly reviewed and electronically signed and dated by the PI.

The PI may be subjected to a field audit by the Sponsor, ICON, and/or FDA inspectors in order to validate the participation of subjects in the study and to verify the data reported in the clinical database. The Sponsor should be notified immediately of any audits scheduled by any regulatory authorities. Copies of audit reports from regulatory authorities should be promptly forwarded to the Sponsor.

The Sponsor and PI uphold the principle of the subject's right to protection against invasion of privacy. Throughout this study, all data collected and analyzed by the Sponsor will be identified only by an identification number.

ICON will provide the study sites access to the EDC database that will be used to collect the required subject eCRF data for this trial. The eCRF must be supported by the corresponding information in the source document.


# 16. QUALITY CONTROL AND QUALITY ASSURANCE

# 16.1. Conduct of the Study

To ensure compliance with GCP and all applicable regulatory requirements, the Sponsor or its representatives may conduct a quality assurance audit.

The study shall be performed in a manner that will implement and maintain quality control and quality assurance procedures with written SOPs to ensure that the study is conducted and data are generated, documented, and reported in compliance with the protocol, International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) GCP, and applicable regulatory requirements.

The study will be conducted in compliance with the following:

- The protocol
- Ethical principles of the Declaration of Helsinki (Version 2013) and its amendments
- The principles of the GCP provided in the ICH Harmonized Tripartite Guidelines for GCP 1996
- FDA regulations (Code of Federal Regulations [CFR], Sections 312.50 and 312.56)
- All applicable national laws and regulations including but not limited to country-specific GCP

Any significant protocol deviations must be documented on the eCRF.

# 16.2. Study Monitoring

The Sponsor or its designee will monitor the study according to GCP guidelines. The PI and study center will permit the Sponsor, its representatives, FDA, and other regulatory agencies direct access to all original source data and documents for study monitoring audits and inspections. All requested information must be entered into the eCRF in the EDC database. The completed eCRF must be promptly reviewed and electronically signed and dated by the PI.

During the study, a Xencor monitor or representative will have regular contacts with the investigational site for the following:

- Provide information and support to the investigators.
- Confirm that facilities remain acceptable.
- Confirm that the investigational team is adhering to the protocol, that data are being accurately recorded in the CRFs, and that investigational product accountability checks are being performed.
- Perform source data verification. This includes a comparison of the data in the CRFs with the subject's medical records at the hospital or practice, and other records relevant to the study. This will require direct access to all original records for each subject (eg, clinic charts).
- Record and report any protocol deviations not previously sent to ICON or Xencor.


 Confirm AEs and SAEs have been properly documented on CRFs, that any SAEs have been forwarded to ICON, and that those SAEs that met criteria for reporting have been forwarded to the IRB/IEC.

The Monitor will be available between visits if the Investigator(s) or other staff need information or advice.

The PI may be subjected to a field audit by the Sponsor, ICON, and/or FDA inspectors in order to validate the participation of subjects in the study and to verify the data reported in the clinical database. The Sponsor should be notified immediately of any audits scheduled by any regulatory authorities. Copies of audit reports from regulatory authorities should be promptly forwarded to the Sponsor.

The Sponsor and PI uphold the principle of the subject's right to protection against invasion of privacy. Throughout this study, all data collected and analyzed by the Sponsor will be identified only by an identification number.

ICON will provide the study sites access to the EDC database that will be used to collect the required subject eCRF data for this trial. The eCRF must be supported by the corresponding information in the source document.


#### 17. ETHICS

# 17.1. Institutional Review Board/Independent Ethics Committee

The PI will submit the protocol, protocol amendments, ICF, Investigator's Brochure, and any subject recruitment materials to the IRB/IEC for approval, as required by 21 CFR, Part 56.

It is required that a valid IRB/IEC approve, in writing, the conduct of this clinical study, together with the Investigator's ICF, prior to study initiation. Until written approval by the IRB/IEC has been received by the Sponsor, no subject may undergo any procedures solely for the purpose of determining eligibility for this study.

The PI must provide study progress reports to the IRB/IEC at least annually for all IND studies or more frequently if required by applicable guidelines, regulations, or institutional procedures.

The PI must promptly notify the IRB/IEC of any SAEs occurring at the site, as well as any IND safety reports reported to the FDA, regardless of the reporting site location.

The Sponsor reserves the right to amend the protocol during the course of the study. It is the PI's responsibility to obtain IRB/IEC approval of any protocol amendments and to implement them in a timely manner. Protocol amendments in the form of an administrative letter signed by the PI should be submitted to the IRB/IEC for review. All protocol amendments must have IRB/IEC review and approval prior to implementation.

If a protocol amendment substantially alters the study design or increases the potential risk to subjects, the ICF must be revised and submitted to the IRB/IEC for review and approval. The revised ICF must be used to obtain consent from subjects currently enrolled in the study if they are affected by the amendment and for all subsequent subjects prior to enrollment.

Documentation of IRB/IEC approval of the protocol, ICF, and other applicable study documents must be provided to the Sponsor or its agent, ICON, before commencement of this study. Copies of all study-related correspondence between the PI and IRB/IEC must be maintained in the site regulatory binder.

#### 17.2. Good Clinical Practice

The procedures set out in this clinical study protocol are designed to ensure that the Sponsor and the Investigator abide by the principles of the ICH guidelines on GCP as outlined in CPMP/ICH/135/95 and the Declaration of Helsinki (Version 2013). The clinical study also will be carried out in keeping with national and local legal requirements (in accordance with US IND regulations [21 CFR Parts 50, 56, and 312]).

The Investigator will be responsible for the care of the subjects throughout the study. If the Investigator is not present at the study site, he/she will leave instructions for the staff and a telephone number where he/she can be reached.

#### 17.3. Written Informed Consent

The PI(s) at each center will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study. Subjects must also

be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided.

The PI is responsible for ensuring that subjects sign an appropriately approved ICF prior to enrolling the subject in the study. Any required signatures must be obtained before conducting any study procedures.

Each subject must sign a statement that he/she has given consent for the subject's participation in the study that complies with the requirements of 21 CFR Part 50. A copy of the signed ICF must be provided to the subject, another copy kept with the study records, and the original kept with the subject's medical records. In addition, the medical records will include documentation of the informed consent process.

A sample of any ICF to be used in this study that has been approved by the IRB/IEC must be forwarded to the Sponsor or its agent, ICON.

## 17.4. Protocol Approval and Amendment(s)

Before the start of the clinical study, the clinical study protocol and other relevant documents will be approved by the IRB/IEC, in accordance with local legal requirements. The Sponsor must ensure that all ethical and legal requirements have been met before the first subject is enrolled in the clinical study.

This protocol is to be followed exactly. Any deviations should be agreed on by both the Sponsor and the Investigator, with the appropriate written and approved protocol amendments made to reflect the changes agreed upon. Protocol amendments must be released by the responsible staff and receive IRB/IEC approval prior to implementation (as appropriate). Where the deviation occurs for the well-being of the subject, the Sponsor must be informed of the action agreed upon.

Administrative changes may be made without the need for a formal amendment but will also be mentioned in the integrated clinical study report. All amendments will be distributed to all study protocol recipients with appropriate instructions.

## 17.5. Subject Confidentiality

Adequate records have to be maintained for the study, including but not limited to subject medical records, eCRFs, laboratory reports, worksheets, nursing notes, signed ICFs, product forms, SAE forms, and information regarding subject discontinuation and reasons for discontinuation. The confidentiality of each record with subject identification is to be guaranteed by the clinical Investigator.

## 18. DATA HANDLING AND RECORD KEEPING

## 18.1. Case Report Forms/Source Data Handling

The Investigator shall be provided with standardized case report forms (CRFs) and shall ensure that all data from subject visits are promptly entered into the CRFs in accordance with the specific instructions given. The Investigator must sign each CRF to verify the integrity of the data recorded.


A list of the normal ranges for all laboratory tests to be undertaken forms part of the documentation to be collated prior to study start. If a central laboratory has been selected to conduct any or all tests, it is essential that all samples be analyzed at that laboratory.

The Investigator must maintain source documents, such as laboratory reports, X-rays, ECGs, consultation reports, and complete medical history and PE reports.

Data to be recorded directly on the CRFs (ie, no prior written or electronic record of data) and considered to be source data must be identified in the protocol.

### 18.2. Retention of Essential Documents

The Investigator or institution should maintain the study documents as specified in the ICH guidelines on GCP and as required by the applicable regulatory requirements. The Investigator or institution should take measures to prevent accidental or premature destruction of these documents.

## 18.3. Principal Investigator's Record Requirements

The PI shall retain study drug disposition records, copies of CRFs (or electronic files), and all source documentation (such as original ECG tracings, laboratory reports, and inpatient or office patient records) for the maximum period required by the country and Institution in which the study will be conducted or for the period specified by the Sponsor, whichever is longer. The PI must contact the Sponsor prior to destroying any records associated with the study. If the PI withdraws from the study (due to relocation, retirement, etc.), the records shall be transferred to a mutually agreed upon designee, such as another PI or the IRB/IEC. Notice of such transfer will be provided in writing to the Sponsor.


## 19. PUBLICATION POLICY

By signing the clinical study protocol, the Investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the Investigator's name, address, qualifications, and extent of involvement.

An Investigator shall not publish any data (poster, abstract, paper, etc.) without receiving approval from the Sponsor in advance. Authorship criteria for all publications of Xencor-sponsored clinical trials are based on the International Committee of Medical Journal Editors guidelines, "Uniform Requirements for Manuscripts Submitted to Biomedical Journals" (Uniform Requirements for Manuscripts Submitted to Biomedical Journals, 2010). Authorship credit can be granted only to those who make substantial contributions to the publication.

At a minimum, study results will be published on www.clinicaltrials.gov on all primary and secondary outcomes, no later than 1 year after completion of the study (including completion of the study if it has been terminated early).

This protocol and other study documents contain trade secrets and commercial information that is privileged and confidential. Such information is not to be disclosed unless required by laws or regulations. The PI agrees to use this information only in conducting this study and is not allowed to use it for other purposes without written consent from the Sponsor. Results obtained from this study are the property of the Sponsor.


## 20. LIST OF REFERENCES

- 1. Barbieri F, Bajetto A, Pattarozzi A, Gatti M, Würth R, Thellung S, et al. Peptide receptor targeting in cancer: The somatostatin paradigm. International Journal of Peptides. 2013(2013):1-20.
- 2. Becker JC, Stang A, DeCaprio JA, Cerroni L, Lebbé C, Veness M, et al. Merkel cell carcinoma. Nat REv Dis Primers. 2017; 26(3):17077. doi:10.1038/nrdp.2017.77.
- 3. Blank C, Brown I, Peterson AC, Spiotto M, Iwai Y, Honjo T, et al. PD-L1/B7H-1 inhibits the effector phase of tumor rejection by T cell receptor (TCR) transgenic CD8+ T cells. Cancer Res. 2004;64(3):1140-5.
- 4. Blincyto® (blinatumomab) [package insert]. Thousand Oaks, CA: Amgen, Inc.; 2018. https://www.accessdata.fda.gov/drugsatfda\_docs/label/2018/125557s013lbl.pdf.
- 5. Bronstein-Sitton N. Somatostatin and the somatostatin receptors: Versatile regulators of biological activity. GPCR Pathways. 2006;2:25-27.
- 6. Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004;173(2):945–54.
- 7. Curran MA, Montalvo W, Yagita H, Allison JP. PD1 and CTLA4 combination blockade expands infiltrating T cells and reduces regulatory T and myeloid cells within B16 melanoma tumors. Proc Natl Acad Sci U S A. 2010;107(9):4275-80.
- 8. Di Bartolomeo M, Bajetta E, Buzzoni R, Mariani L, Carnaghi C, Somma L, et al. Clinical efficacy of octreotide in the treatment of metastatic neuroendocrine tumors. A study by the Italian Trials in medical Oncology Group. Cancer 1996; 77(2):402-08.
- 9. Disis, ML. Immune regulation of cancer. J Clin Oncol. 2010;28(29):4531-38.
- 10. Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, et al. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005;23(10):2346-57.
- 11. Eng T, Naquib M, Fuller CD, Jones WE 3<sup>rd</sup>, Herman TS. Treatment of recurrent Merkel cell carcinoma: an analysis of 46 cases. Am J Clin Oncol. 2004; 27(6):576-83.
- 12. Epstude M, Tornquist K, Riklin C, di Leonardo F, Winterhalder R, Hug U, et al. Comparison of (18)F-FDG PET/CT and (68)Ga-DOTATATE PET/CT imaging in metastasized Merkel cell carcinoma. Clin Nucl Med. 2013; 38(4):283-4.
- 13. Frey N. Cytokine release syndrome: who is at risk and how to treat. Best Pract Res Clin Haematol. 2017;30:336–40.
- 14. Früh M, De Ruysscher D, Popat S, Crinò L, Peters S, Felip E. Small-cell lung cancer (SCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013;24 Suppl 6:vi99-105.


- 15. Gardair C, Samimi M, Touze A, Coursaget P, Lorette G, Caille A, et al. Somatostatin receptors 2A and 5 are expressed in Merkel cell carcinoma with no association with disease severity. Neuroendocrinology. 2015;101(3):223-35.
- 16. Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48.
- 17. Harms K, Healy M, Nghiem P, Sober A, Johnson T, Bichakjian C, et al. Analysis of prognostic factors from 9387 Merkel cell carcinoma cases forms the basis for the new 8<sup>th</sup> Edition AJCC Staging System. Ann Surg Oncol. 2016; 23(11):3564-71.
- HEMLIBRA® (emicizumab-kxwh) [package insert]. South San Francisco, CA: Genentech, Inc.; 2018.
   https://www.accessdata.fda.gov/drugsatfda\_docs/label/2018/761083s002s004lbl.pdf
- 19. Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, et al. Blockade of B7-H1 and PD1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005;65(3):1089 96.
- 20. Horn L, Mansfield AS, Szczęsna A, Havel L, Krzakowski M, Hochmair MJ, et al. First-Line atezolizumab plus chemotherapy in extensive-stage small-cell lung cancer. N Engl J Med. 2018;379(23):2220-2229.
- 21. Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, et al. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008;358(25):2698 703.
- 22. Ivanova A, Qaqish BF, Schell MJ: Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005;61:540-545.
- 23. Iyer J, Blom A, Doumani R, Lewis C, Tarabadkar E, Anderson A, et al. Response rates and durability of chemotherapy among 62 patients with metastatic Merkel cell carcinoma. Cancer Med. 2016; 5(9):2294-301.
- 24. Kalemkerian G, Loo B, Akerley W, Attia A, Bassetti M, Boumber Y, et al. NCCN Guidelines Version 2.2018 Small Cell Lung Cancer. January 2018.
- 25. Kaufman H, Russell J, Hamid O, Bhatia S, D'Angelo SP, Shih KC, et al. Avelumab in patients with chemotherapy-refractory metastatic Merkel cell carcinoma: a multicentre, single-group, open-label, phase 2 trial. Lancet Oncol. 2016; 17(10):1374-1385.
- 26. Kaufman H, Russell J, Hamid O, Bhatia S, Terheyden P, D'Angelo SP, et al. Updated efficacy of avelumab in patients with previously treated metastatic Merkel cell carcinoma after ≥1 year of follow-up: JAVELIN Merkel 200, a phase 2 clinical trial. J Immunother Cancer. 2018; 6(1):7.
- 27. Keytruda® (pembrolizumab) [package insert]. Whitehouse Station, NJ: Merck & Co., Inc.; 2020. https://www.accessdata.fda.gov/drugsatfda\_docs/label/2020/125514s067lbl.pdf
- 28. Kobold S, Pantelyushin S, Rataj F, Vom Berg J. Rationale for combining bispecific T cell activating antibodies with checkpoint blockade for cancer therapy. Front Oncol. 2018;25;8:285.


- 29. Kritikos N, Priftakis D, Stavrinides S, Kleanthous S, Sarafianou E. Nuclear medicine techniques in Merkel cell carcinoma: A case report and review of the literature. Oncol Lett. 2015;10(3):1610-16.
- 30. Lapa C, Hänscheid H, Wild V, Pelzer T, Schirbel A, Werner RA, et al. Somatostatin receptor expression in small cell lung cancer as a prognostic marker and a target for peptide receptor radionuclide therapy. Oncotarget. 2016;7(15):20033-40.
- 31. Lee D, Gardner R, Porter DL, et al. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014;124(2):188-195.
- 32. Lee D, Santomasso B, Locke F, Ghobadi A, Turtle C, Brudno J, et al. ASTCT consensus grading for cytokine release syndrome and neurologic toxicity associated with immune effector cells. Biol Blood Marrow Transplant. 2019;25(4):625-638.
- 33. Lehman JM, Hoeksema MD, Staub J, Qian J, Harris B, Callison JC, et al. Somatostatin receptor 2 signaling promotes growth and tumor survival in small-cell lung cancer. Int J Cancer. 2019;144(5):1104–1114.
- 34. Lenz H-J. Management and preparedness for infusion and hypersensitivity reactions. The Oncologist. 2007;12(5):601–9.
- 35. Li J, Piskol R, Ybarra R, Ying-Jiun JC, Li J, Slaga D, et al. CD3 bispecific antibody-induced cytokine release is dispensable for cytotoxic T cell activity. Sci Transl Med. 2019; 11(eaax8861):1-12.
- 36. Meier G, Waldherr C, Herrmann R, Maecke H, Mueller-Brand J, Pless M. Successful targeted radiotherapy with 90Y-DOTATOC in a patient with Merkel cell carcinoma. A case report. Oncology. 2004; 66(2):160-163.
- 37. NETSPOT (kit for the preparation of gallium GA 68 dotate injection) [package insert]. Saluggia (Vc), Italy: Gipharma S.r.l; 2018. https://www.accessdata.fda.gov/drugsatfda\_docs/label/2018/208547s011lbl.pdf
- 38. Nghiem P, Bhatia S, Brohl AS, Hamid O, Mehnert J, Terheyden P, et al. Two-year efficacy and safety update from JAVELIN Merkel 200 part A: A registrational study of avelumab in metastatic Merkel cell carcinoma progressed on chemotherapy. J Clin Oncol. 2018; 36S: ASCO #9507.
- 39. Nghiem P, Bhatia S, Lipson E, Sharfman W, Kudchadkar R, Brohl S, et al. Durable tumor regression and overall survival in patients with advanced Merkel cell carcinoma receiving Pembrolizumab as first-line therapy. J Clin Oncol. 2019; 37(9):693-702.
- 40. Nomi T, Sho M, Akahori T, Hamada K, Kubo A, Kanehiro H, et al. Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic cancer. Clin Cancer Res. 2007;13(7):2151-7.
- 41. Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting SRC homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001;98(24):13866-71.


Xencor, Inc

- 42. Paulson KG, Park SY, Vandeven NA, Lachance K, Thomas H, Chapuis AG, et al. Merkel cell carcinoma: current US incidence and projected increases based on changing demographics. J Am Acad Dermatol. 2018;78(3):457-463.
- 43. Pilon-Thomas S, Mackay A, Vohra N, Mulé JJ. Blockade of programmed death ligand 1 enhances the therapeutic efficacy of combination immunotherapy against melanoma. J Immunol. 2010;184(7): 3442-9.
- 44. Przepiorka D, Ko C-W, Deisseroth A, Yancey CL, Candau-Chacon R, Chiu HJ, et al. FDA approval: Blinatumomab. Clin Cancer Res. 2015;21(18):4035-4039.
- 45. Reisinger I, Bohuslavitzki KH, Brenner W, Braune S, Dittrich I, Geide A, et al. Somatostatin receptor scintigraphy in small-cell lung cancer: results of a multicenter study. J Nucl Med. 1998;39(2):224-7.
- 46. Reubi JC, Waser B, Liu Q, Laissue JA, Schonbrunn A. Subcellular distribution of somatostatin sst2A receptors in human tumors of the nervous and neuroendocrine systems: membranous versus intracellular location. J Clin Endocrinol Metab. 2000 Oct;85(10):3882-91.
- 47. Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009; 229(1):114-25.
- 48. Salavati A, Prasad V, Schneider CP, Herbst R, Baum RP. Peptide receptor radionuclide therapy of Merkel cell carcinoma using (177)lutetium-labeled somatostatin analogs in combination with radiosensitizing chemotherapy: a potential novel treatment based on molecular pathology. Ann Nuc Med. 2012; 26(4):365-9.
- 49. Schmults C, Blitzblau R, Aasi S, Alam M, Anderson J, Bordeaux J, et al. NCCN Guidelines Version 2.2019 Merkel Cell Carcinoma. January 2019. Available from: https://merkelcell.org/wp-content/uploads/2017/10/MCC v.2.2019-2.pdf
- 50. Schultz JR, Nichol FR, Elfring GL, Weed SD. Multiple-stage procedures for drug screening. 1973;29(2):293-300.
- 51. Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, et al. PD1 inhibits T-cell receptor-induced phosphorylation of the ZAP70/CD3 signalosome and downstream signaling to PKCtheta. FEBS Letters. 2004; 574(1-3):37-41.
- 52. Shimabukuro-Vornhagen A, Gödel P, Subklewe M, Stemmler HJ, Schlößer HA, Schlaak M, et al. Cytokine release syndrome. J Immunother Cancer. 2018;6(1):56
- 53. Spiess C, Zhai Q, Carter P. Alternative molecular formats and therapeutic applications for bispecific antibodies. Mol Immunol. 2015;67(2PtA):95-106.
- 54. Spranger S, Koblish HK, Horton B, Scherle PA, Newton R, Gajewski TF. Mechanism of tumor rejection with doublets of CTLA-4, PD-1/PDL-1, or IDO blockade involves restored IL-2 production and proliferation of CD8(+) T cells directly within the tumor microenvironment. J Immunother Cancer. 2014;2:3.
- 55. Strome SE, Dong H, Tamura H, Voss SG, Flies DB, Tamada K, et al. B7-H1 blockade augments adoptive T-cell immunotherapy for squamous cell carcinoma. Cancer Res. 2003;63(19):6501-5.


Protocol XmAb18087-02

- 56. Taniyama Y, Suzuki T, Mikami Y, Moriya T, Satomi S, Sasano H. Systemic distribution of somatostatin receptor subtypes in human: An immunohistochemical study. Endocrine J. 2005;52(5):605-611.
- 57. Tartarone A, Lerose R, Aieta M. Somatostatin analog therapy in small cell lung cancer. Semin Nucl Med. 2016;46(3):239-42.
- 58. Topalian S, Bhatia S, Hollebecque A, Awada A, de Boer JP, Kudchadkar R, et al. Non-comparative, open-label, multiple cohort, phase 1/2 study to evaluate nivolumab (NIVO) in patients with virus-associated tumors (CheckMate 358): Efficacy and safety in Merkel cell carcinoma (MCC). Cancer Res. 2017; 77S: AACR #CT074.
- 59. U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research. Guidance for Industry: Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. 2005 July. Available from: https://www.fda.gov/ucm/groups/fdagov-public/@fdagov-drugs-gen/documents/document/ucm078932.pdf.
- 60. Uniform requirements for manuscripts submitted to biomedical journals: Writing and editing for biomedical publication. J Pharmacol Pharmacother. 2010;1(1):42-58.
- 61. Weber J. Immune checkpoint proteins: a new therapeutic paradigm for cancer—preclinical background: CTLA-4 and PD-1 blockade. Semin Oncol. 2010;37(5):430-9.
- 62. Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, et al. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004; 20(3):337-47.


## APPENDIX A. RECIST GUIDELINES

#### RECIST GUIDELINES

Selected Definitions and Tables from Revised RECIST Guidelines (Version 1.1)

## 1. Measurability of tumor at baseline

At baseline, tumor lesions will be categorized as measurable or nonmeasurable as follows:

## 1.1 Measurable tumor lesions

Lesions must be accurately measured in at least 1 dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of

- 10 mm by CT scan (CT scan slice thickness no greater than 5 mm)
- 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as nonmeasurable)
- 20 mm by chest X-ray

## 2. Measurability of lymph nodes at baseline

• Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be ≥ 15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

#### 3. Nonmeasurable lesions

Nonmeasurable lesions are all other lesions, including the following:

- Small lesions (longest diameter < 10 mm or pathological lymph nodes with P10 to < 15 mm short axis) as well as truly nonmeasurable lesions
- Lesions considered truly nonmeasurable include: leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.

## 4. Response criteria

- 4.1 Target lesions
- A maximum of 5 target lesions may be identified and assessed for response.
- The following definitions are used to determine objective tumor response for target lesions.
  - 1. Complete Response (CR): Disappearance of all target lesions
    - Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.</li>
  - 2. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters


- 3. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of 1 or more new lesions is also considered progression).
- 4. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.

## 4.2 Nontarget lesions

While some nontarget lesions may actually be measurable, they need not be measured and instead should be assessed only qualitatively at the time points specified in the protocol. The following tumor response definitions apply to the group of nontarget lesions:

- Complete Response (CR): Disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes must be nonpathological in size (< 10 mm short axis).
- Non-CR/Non-PD: Persistence of one or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limit
- Progressive Disease (PD): Unequivocal progression of existing nontarget lesions. (Note: the appearance of 1 or more new lesions is also considered progression.)

#### 4.3 New lesions

The appearance of new malignant lesions denotes disease progression. There are no specific criteria for the identification of new radiographic lesions; however, the finding of a new lesion should be unequivocal: ie, not attributable to differences in scanning technique, change in imaging modality, or findings thought to represent something other than tumor (for example, some 'new' bone lesions may be simply healing or flare of preexisting lesions). This is particularly important when the subject's baseline lesions show partial or complete response. For example, necrosis of a liver lesion may be reported on a CT scan report as a 'new' cystic lesion, which it is not.

A lesion identified on a follow-up study in an anatomical location that was not scanned at baseline is considered a new lesion and will indicate disease progression. An example of this is the subject who has visceral disease at baseline and while on study has a CT or MRI of the brain which reveals metastases. The subject's brain metastases are considered to be evidence of PD even if he/she did not have brain imaging at baseline.

If a new lesion is equivocal, for example because of its small size, continued therapy and follow-up evaluation will clarify if it represents truly new disease. If repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the initial scan.

## 5. Evaluation of overall response

The best overall response is the best response recorded from the start of the study treatment until the end of treatment, taking into account any requirement for confirmation. On occasion a response


Protocol XmAb18087-02

Xencor, Inc

may not be documented until after the end of therapy, so protocols should be clear if post-treatment assessments are to be considered in determination of best overall response.

The subject's overall response assignment will depend on the findings of both target and nontarget disease and will also take into consideration the appearance of new lesions.

This is captured in Table 13 (below).

**Table 13:** Assessment of Overall Response in Subjects with Target (± Nontarget Disease)

| Target Lesions | Nontarget Lesions | New Lesions | Overall Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | Not evaluable |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

CR = complete response; PD = progressive disease; PR = partial response; SD = stable disease.

#### Sources:

Eisenhauer E, Therasse P, and Bogaerts J, et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1), Eur J Can. 2009; 45: 228-247.

Chalian H, Tore H, Horowitz J, et al. Radiologic assessment of response to therapy: Comparison of RECIST versions 1.1 and 1.0, Rad Onc 2011; 31: 2093-2105.


## APPENDIX B. ECOG PERFORMANCE SCALE

**Table 14: ECOG Performance Scale** 

| Grade | Description |
|---|---|
| 0 | Normal activity. Fully active, able to carry on all predisease performance without restriction. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (eg, light housework, office work). |
| 2 | In bed < 50% of the time. Ambulatory and capable of all selfcare, but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | In bed > 50% of the time. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair. |
| 5 | Dead |

ECOG=Eastern Cooperative Oncology Group.


# APPENDIX C. PROPHYLAXIS AND MANAGEMENT OF NAUSEA AND VOMITING AND HYPERSENSITIVITY REACTIONS, CYTOKINE RELEASE SYNDROME, AND NEUROLOGICAL TOXICITY

## Prophylaxis and Management of Nausea and Vomiting



Sites may also choose to use other/additional antinausea/vomiting medications for prophylaxis or treatment of symptoms, according to their practice and assessment of the subject's responses.

# Guidelines for Prophylaxis and Management of Hypersensitivity Reactions, Cytokine Release Syndrome, and Neurological Toxicity Attributed to XmAb18087

Because administration of XmAb18087 has been associated with symptoms of infusion reaction/CRS in some subjects, it is required that all subjects receive the following medications before at least the first 4 doses of XmAb18087:

- c. Acetaminophen (Tylenol®): 650 mg PO once before dosing with XmAb18087
- d. Diphenhydramine (Benadryl®): 50 mg PO once before dosing with XmAb18087
- e. 10 to 20 mg IV dexamethasone (Decadron®) before dosing with XmAb18087

If a subject receives 4 consecutive doses of XmAb18087 without  $\geq$  Grade 1 infusion reaction/CRS, the prophylaxis described above may be modified, prophylactic medications are to be administered to all subjects before at least the first 4 doses of the study drug.

## **Introduction and Grading**

Grading of toxicity, including allergic/hypersensitivity reactions, is by CTCAE version 5.0, except for CRS, which is using the ASTCT CRS Consensus Grading (Lee, 2019). See Table 15 for these definitions.

All sites should review and implement the general guidelines for the use of tocilizumab and IV fluids discussed below. Otherwise, management of CRS and other infusion-related reactions


should be per standard investigational site procedures. Or, if there are no local standards or if they are incomplete, the approaches discussed here may be used.


Table 15. American Society for Transplantation and Cellular Therapy Cytokine Release Syndrome Consensus Grading

| CRS Parameter | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Fever <sup>a</sup> | Temperature ≥ 38 °C | Temperature ≥ 38 °C | Temperature ≥ 38 °C | Temperature ≥ 38 °C |
| | | With | | |
| Hypotension | None | Not requiring vasopressors | Requiring a vasopressor with or without vasopressin | Requiring multiple<br>vasopressors<br>(excluding<br>vasopressin) |
| | | And/or <sup>b</sup> | | |
| Hypoxia | None | Requiring low-flow<br>nasal cannula <sup>c</sup> or<br>blow-by | Requiring high-flow<br>nasal cannula <sup>c</sup> ,<br>facemask,<br>nonrebreather mask,<br>or Venturi mask | Requiring positive<br>pressure (eg, CPAP,<br>BiPAP, intubation<br>and mechanical<br>ventilation) |

BiPAP = bilevel positive airway pressure; CPAP = continuous positive airway pressure; CRS = cytokine release syndrome; CTCAE = Common Terminology Criteria for Adverse Events.

Organ toxicities associated with CRS may be graded according to CTCAE v5.0, but they do not influence CRS grading.

## Cytokine Release Syndrome Versus Allergic or Hypersensitivity Reactions

Cytokine release syndrome is mechanistically different from allergic/hypersensitive reactions (Lee, 2014), although some of the manifestations are common to both AEs and both have been reported to occur with therapeutic antibodies. An acute infusion reaction is often caused by a type 1 hypersensitivity mechanism due to IgE-mediated release of histamines and prostaglandins, although a direct interaction with mast cells and basophils can also occur. It is less clear how cytokine release is triggered, although it is likely to be associated with immune cell activation; in this case, there is evidence that immunologic cascade is initiated by triggering of CD3-expressing T lymphocytes, resulting in TNF-α mediated monocyte/macrophage activation and systemic toxic cytokine release (Li, 2019).

Signs and symptoms usually develop during or shortly after drug infusion in hypersensitivity reactions, are more likely to occur after several doses of the drug and are largely related to histamine release. Typical signs and symptoms of hypersensitivity reaction include rash/urticaria,


<sup>&</sup>lt;sup>a</sup> Fever is defined as temperature ≥ 38 °C not attributable to any other cause. In patients who have CRS then receive antipyretic or anticytokine therapy such as tocilizumab or steroids, fever is no longer required to grade subsequent CRS severity. In this case, CRS grading is driven by hypotension and/or hypoxia.

<sup>&</sup>lt;sup>b</sup> CRS grade is determined by the more severe event: hypotension or hypoxia not attributable to any other cause. For example, a patient with temperature of 39.5 °C, hypotension requiring 1 vasopressor, and hypoxia requiring low-flow nasal cannula is classified as grade 3 CRS.

<sup>&</sup>lt;sup>c</sup> Low-flow nasal cannula is defined as oxygen delivered at  $\leq$  6 L/minute. Low flow also includes blow-by oxygen delivery, sometimes used in pediatrics. High-flow nasal cannula is defined as oxygen delivered at  $\geq$  6 L/minute.

flushing, pruritus, fever, dyspnea, cough, and hypotension, although the following may also occur (Lenz, 2007):

- Arthralgia
- Bronchospasm
- Confusion, mental status changes, and/or delirium
- Dizziness
- Fatigue (asthenia, lethargy, malaise)
- Hallucinations
- Headache
- Hypertension
- Myalgia
- Nausea and/or vomiting
- Rigors/chills
- Diaphoresis
- Tachycardia

Cytokine release syndrome, on the other hand, is more likely to occur after the first dose or first escalated dose of drug than after subsequent doses. It may begin somewhat later and is more likely to be associated with hepatic and neurologic complications, including the following:

- Any of the hypersensitivity signs or symptoms listed above
- Aphasia or word-finding difficulty
- Elevated d-dimer and/or hypofibrinogenemia
- Fatigue (asthenia, lethargy, malaise)
- Gait disturbance/dysmetria
- Hallucinations
- Seizures
- Transaminitis and/or hyperbilirubinemia
- Tremor

The Xencor Medical Monitor should be contacted immediately if questions arise concerning the grade and/or treatment of the infusion reaction.

## **Treatment Guidelines for Cytokine Release Syndrome**

## Use of Tocilizumab for Cytokine Release Syndrome

Tocilizumab is a therapeutic antibody that interferes with binding of IL-6 to the IL-6 receptor. It has been used to decrease the severity and possibly mortality of severe CRS (Frey, 2017), and


early administration may be useful in improving outcomes. Below are suggested guidelines for its use:

- Sufficient tocilizumab (dose of 8 mg/kg) should be readily available to the area where subjects are receiving their infusions and being observed post infusion.
- Prompt tocilizumab therapy should be strongly considered if:
  - Oxygen saturation falls below 90% on room air, **OR**
  - Systolic blood pressure falls 20 mm Hg below predose measurements and below 100 mm Hg, **OR**
  - Temperature of > 38 °C (100.4 °F) in the presence of new or worsening dyspnea and/or tachypnea and/or rigors and/or tachycardia (HR > 110 bpm), OR
  - Early discovery of hepatic transaminase elevation. (Note that peak transaminase elevation appears to occur within 24 hours, so that it is unlikely that tocilizumab treatment on the day after study drug administration would affect the course or outcome in the absence of concurrent symptoms or signs of CRS).
- Repeat dosing of tocilizumab may be necessary if signs and symptoms persist or return after initial treatment.

## Fluid Management

Cytokine release syndrome is sometimes associated with myocardial dysfunction, pulmonary edema, or capillary leak syndrome (Shimabukuro-Vornhagen, 2018). Although there are little or no data regarding use of anti-CD3 antibodies and the need for fluid management, it seems prudent to monitor subjects for weight gain and limit IV fluid administration in the acute setting.

- If a subject is noted to have had a ≥ 10% increase in body weight over the previous 2 weeks in association with new or significantly increased bilateral lower extremity edema, dosing should be delayed until this finding is evaluated and, if indicated, treated
- For acute hypotension, an IV fluid bolus should be limited to 500 mL of normal saline or the equivalent.
- If there is not an adequate response to fluids, treatment with tocilizumab (and vasopressors, if necessary) should be considered rather than additional fluid boluses.

## Cytokine Release Syndrome Treatment Guidelines by Grade

The following are treatment guidelines for XmAb18087 treatment-related infusion reactions (Lee, 2014); since it can be difficult to differentiate between different infusion reaction etiologies, both are included here.

#### Grade 1:

- Administer acetaminophen and/or diphenhydramine or dexamethasone to treat signs and symptoms if clinically indicated.
- Vital signs should be measured every 15 minutes or less as clinically indicated.


- Obtain a blood sample for cytokine analysis during the event and approximately 4 hours later, unless scheduled cytokine monitoring is already in progress.
- Monitor the subject for worsening of condition; if severity of event increases to a higher grade, stop the infusion, administer appropriate treatment, and refer to guidelines below for more severe infusion reactions.
- It may be useful to premedicate the subject with acetaminophen and antihistamines prior to the next infusion.

#### Grade 2:

- Hypotension responsive to fluids or a low dose of a single pressor, or mild respiratory symptoms treatable with low-flow oxygen are signs of Grade 2 toxicity. Older subjects or those with significant comorbidities may be at higher risk of decompensation in this situation.
- **Discontinue the infusion** and administer acetaminophen and/or diphenhydramine or dexamethasone to treat signs and symptoms if clinically indicated. Once symptoms have resolved, slow the infusion rate by 50% of the baseline rate. If after 1 hour, the subject's symptoms do not return and vital signs are stable, the infusion rate may be increased every 30 minutes, as tolerated, to the baseline rate.
- Note that older subjects or those with significant comorbidities may be at higher risk of decompensation in this situation. When reactions occur in these vulnerable subjects, or in the case of rapidly escalating reactions, consider treatment with **tocilizumab** 4 to 8 mg/kg IV over 1 hour, with or without dexamethasone 10 to 20 mg IV (or equivalent).
- Vital signs should be measured every 15 minutes or less as clinically indicated. For subjects who are able to tolerate an increase in the infusion rate back to baseline and maintain normal blood pressure for 30 minutes after the rate increase then, at the discretion of the Investigator, the frequency of vital sign assessment may be reduced to every 30 minutes during the infusion.
- Obtain a blood sample for cytokine analysis during the event and approximately 4 hours later, in addition to scheduled cytokine monitoring if already in progress.
- Monitor the subject for worsening of condition; if severity of event increases to a higher grade, stop the infusion, administer appropriate treatment, and refer to guidelines below for Grades 3 and 4 infusion reactions.
- Subjects with maximum Grade 2 infusion reaction may continue on study and should receive prophylactic premedication with acetaminophen 650 mg PO and diphenhydramine hydrochloride 25 to 50 mg IV or PO prior to all subsequent XmAb18087 infusions

#### Grade 3 and 4:

• Stop the infusion and disconnect the infusion tubing from the subject.


- Aggressive supportive care should be given immediately. Vasopressors, fluids, oxygen, epinephrine or bronchodilators, ventilatory support, antipyretics, and analgesics should be used as indicated.
- Treatment with tocilizumab 4 to 8 mg/kg IV over 1 hour with or without dexamethasone 10 mg IV (or equivalent) is strongly encouraged for CRS due to the high risk of progression and permanent organ dysfunction.
- Hospital admission for observations is almost always indicated, usually to an intensive care unit, since an initial appearance of improvement may quickly yield to rapid decompensation.
- Subjects with Grade 3 CRS or infusion reaction may be rechallenged once resolved. Subjects with recurrent Grade 3 or any Grade 4 infusion reaction should not receive further XmAb18087 treatment but will continue to be followed on the protocol (ie, for 4 weeks after last dose).
- Obtain a blood sample for cytokine analysis during the event and approximately 4 hours later, in addition to scheduled cytokine monitoring if already in progress.
- Obtain a sample for ADA testing as close to the onset of the event as possible, at the resolution of the event, and 28 days following the event.
- Notify the Xencor Safety Monitor or Xencor Medical Monitor, (Telephone: ; Email: ), immediately.

## Neurotoxicity

In addition to CRS, another toxicity observed after CAR-T cell therapy and CD3 bispecific antibodies is neurotoxicity. ICANS may manifest as delirium, encephalopathy, aphasia, lethargy, difficulty concentrating, agitation, tremor, seizures, and, rarely, cerebral edema (Lee, 2019). Neurotoxicity was previously considered in aggregate with CRS, but is now treated separately, due to its timing and response to treatment.

Neurologic symptoms may occur during or after CRS symptoms, but rarely precede CRS symptoms. The earliest manifestations of ICANS are tremor, dysgraphia, mild difficulty with expressive speech (especially in naming objects), impaired attention, apraxia, and mild lethargy. Headache is a nonspecific symptom, frequently occurring during fever or after chemotherapy in patients without other neurologic dysfunction. Thus, headache alone is not a useful marker of ICANS. Expressive aphasia, on the other hand, appears to be a very specific symptom of ICANS (Lee, 2019).

A consensus grading scheme, which is a slightly modified version of the CARTOX-10 screening tool, which incorporated key elements of the MMSE, the ICE score, will be used for the grading of ICANS (Table 9). It is important to note that the 10-point ICE screening tool is helpful for assessing patients for encephalopathy; however, the grading of ICANS requires assessment of the 10-point ICE score as well as evaluation of other neurologic domains, such as level of consciousness, motor symptoms, seizures, and signs of elevated ICP/cerebral edema, which may occur with or without encephalopathy. The ASTCT ICANS toxicity grading system is shown in Table 16. This grading scale will be used to assess neurotoxicity, rather than the CTCAE 5.0.


## Table 16: Immune Effector Cell-associated Encephalopathy Scoring

#### **ICE**

Orientation: orientation to year, month, city, hospital: 4 points

Naming: ability to name 3 objects (eg, point to clock, pen, button): 3 points

**Following commands:** ability to follow simple commands (eg, "Show me 2 fingers" or "Close your eyes and stick out your tongue"): 1 point

Writing: ability to write a standard sentence (eg, "Our national bird is the bald eagle"): 1 point

Attention: ability to count backwards from 100 by 10: 1 point

ICANS = immune effector cell-associated neurotoxicity syndrome; ICE = Immune Effector Cell-Associated Encephalopathy (score).

Scoring: 10, no impairment;

- 7 9, Grade 1 ICANS;
- 3 6, Grade 2 ICANS;
- 0 2, Grade 3 ICANS;

0 due to patient unarousable and unable to perform ICE assessment, Grade 4 ICANS (Lee, 2019).


Table 17: American Society for Transplantation and Cellular Therapy Immune Effector Cell-associated Neurotoxicity Syndrome Consensus Toxicity Grading for Adults

| Neurotoxicity<br>Domain | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| ICE score <sup>a</sup> | 7 – 9 | 3 - 6 | 0-2 | 0 (patient is<br>unarousable and<br>unable to perform<br>ICE) |
| Depressed level of consciousness <sup>b</sup> | Awakens spontaneously | Awakens to voice | Awakens only to tactile stimulus | Patient is<br>unarousable or<br>requires vigorous or<br>repetitive tactile<br>stimuli to arouse.<br>Stupor or coma |
| Seizure | N/A | N/A | Any clinical seizure focal or generalized that resolves rapidly or nonconvulsive seizures on EEG that resolve with intervention | Life-threatening prolonged seizure (> 5 min); or Repetitive clinical or electrical seizures without return to baseline in between |
| Motor findings <sup>c</sup> | N/A | N/A | N/A | Deep focal motor<br>weakness such as<br>hemiparesis or<br>paraparesis |
| Elevated ICP/cerebral edema | N/A | N/A | Focal/local edema on neuroimaging <sup>d</sup> | Diffuse cerebral edema on neuroimaging; decerebrate or decorticate posturing; or cranial nerve VI palsy; or papilledema; or Cushing's triad |

EEG = electroencephalogram; ICANS = immune effector cell-associated neurotoxicity syndrome; ICE = Immune Effector Cell-Associated Encephalopathy (score); ICP = intracranial pressure; N/A = not applicable; VI = sixth.

ICANS grade is determined by the most severe event (ICE score, level of consciousness, seizure, motor findings, raised ICP/cerebral edema) not attributable to any other cause; for example, a patient with an ICE score of 3 who has a generalized seizure is classified as grade 3 ICANS.

It has been speculated that high levels of IL-6 may directly mediate neurotoxicity in this situation (Lee, 2014).


<sup>&</sup>lt;sup>a</sup> A patient with an ICE score of 0 may be classified as Grade 3 ICANS if awake with global aphasia, but a patient with an ICE score of 0 may be classified as Grade 4.

<sup>&</sup>lt;sup>b</sup> Depressed level of consciousness should be attributable to no other cause (eg, no sedating medication).

<sup>&</sup>lt;sup>c</sup> Tremors and myoclonus associated with immune effector cell therapies may be graded according to CTCAE v5.0, but they do not influence ICANS grading.

<sup>&</sup>lt;sup>d</sup> Intracranial hemorrhage with or without associated edema is not considered a neurotoxicity feature and is excluded from ICANS grading. It may be graded according to CTCAE v5.0 (Lee, 2019).

Clinical management of neurotoxicity consists of the following:

- Monitor subjects closely for signs and symptoms of these events (including administration of mental status and neurologic examinations when these seem clinically warranted).
- If neurotoxicity becomes evident, a blood sample for cytokine analysis should be drawn at that time, and again 4 hours later, in addition to scheduled cytokine monitoring if already in progress.
- If neurologic toxicity is Grade 4, discontinue XmAb18087, if still infusing.
- For Grade 3 neurologic toxicity, withhold both drugs until the toxicity has recovered to ≤ Grade 1 (mild) and has remained at ≤ Grade 1 for at least 3 days before restarting therapy. Restart XmAb18087 at 75% of the previous dose. Restart pembrolizumab at the full dose. Escalate back to full dose at the time of the next dose if ≥ Grade 2 toxicity does not recur. If ≥ Grade 2 toxicity reoccurs at 75% dose, or if < Grade 2 toxicity takes more than 7 days to resolve, discontinue permanently.
- For severe neurologic symptoms, administer additional dexamethasone 10 mg intravenously and repeat every 12 hours if symptoms do not abate rapidly, or treat according to the clinical site's institutional protocol for such reactions.
- For recurrent seizures, anticonvulsant therapy may be necessary.


# Appendix D. DOSE MODIFICATION AND TOXICITY MANAGEMENT FOR IMMUNE-RELATED ADVERSE EVENTS

IRAEs may occur shortly after the first dose of pembrolizumab or up to several months after the last dose. Based on existing clinical data for pembrolizumab and other checkpoint inhibitors, most IRAEs were reversible and could be managed with dose interruptions, administration of corticosteroids, and/or other supportive care. For suspected IRAEs, ensure adequate evaluation to confirm etiology or exclude other causes. Additional procedures or tests such as bronchoscopy, endoscopy, or skin biopsy may be included as part of the evaluation. IRAEs known to be associated with pembrolizumab, as well as guidelines for dose modification and management when they occur, are described in the Keytruda Prescribing Information (Keytruda® Package Insert, 2020); these guidelines are summarized in Table 18.

For additional information on diagnosis and management of IRAEs, see the NCCN Guidelines – Management of Immunotherapy-Related Toxicities (Appendix E).


## Table 18: Dose Modification and Toxicity Management Guidelines for Immune-Related Adverse Events in Patients Receiving Pembrolizumab

#### **General Instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, it can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered.
- 3. For severe and life-threatening IRAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if IRAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity Grade or<br>Conditions (CTCAE<br>v5.0) | Action Taken with<br>Pembrolizumab | IRAE Management with Corticosteroid and/or Other Therapies | Monitor and Follow-up |
|---|---|---|---|---|
| Pneumonitis | Grade 2 | Withhold | Administer corticosteroids (initial dose of | Monitor participants for signs and symptoms of pneumonitis Evaluate participants with |
| | Grade 3 or 4, or recurrent Grade 2 | Permanently discontinue | 1 - 2 mg/kg<br>prednisone or<br>equivalent)<br>followed by taper | suspected pneumonitis with radiographic imaging and initiate corticosteroid treatment Add prophylactic antibiotics for opportunistic infections |
| Diarrhea/Colitis | Grade 2 or 3 | Withhold | Administer<br>corticosteroids<br>(initial dose of<br>1 - 2 mg/kg<br>prednisone or<br>equivalent)<br>followed by taper | Monitor participants for signs and symptoms of enterocolitis (ie, diarrhea, abdominal pain, blood or mucus in stool with or without fever) and of bowel perforation (ie, peritoneal signs and ileus). Participants with ≥ Grade 2 diarrhea suspecting colitis should consider GI consultation and performing endoscopy to rule out |
| | Grade 4 | Permanently discontinue | | colitis. Participants with diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion. |
| Immune-mediated hepatitis | AST or ALT greater than 3 but no more than 5 times the ULN or total bilirubin greater than 1.5 but no more than 3 times the ULN | Withhold | Administer corticosteroids (initial dose of 0.5 - 1 mg/kg prednisone or equivalent) followed by taper | Monitor with liver function tests<br>(consider weekly or more<br>frequently until liver enzyme<br>value returned to baseline or is<br>stable) |


| Immune-related<br>AEs | Toxicity Grade or<br>Conditions (CTCAE<br>v5.0) | Action Taken with<br>Pembrolizumab | IRAE Management with Corticosteroid and/or Other Therapies | Monitor and Follow-up |
|---|---|---|---|---|
| | In patients without liver metastases, AST or ALT greater than 5 times ULN or total bilirubin greater than 3 times ULN In patients with liver metastasis and Grade 2 AST or ALT at baseline, with an increase in AST or ALT of 50% or more relative to baseline that persists for at least 1 week | Permanently discontinue | Administer corticosteroids (initial dose of 1 - 2 mg/kg prednisone or equivalent) followed by taper | |
| Immune-mediated endocrinopathies | Grades 3 or 4 | Withhold until clinically stable | Administer<br>corticosteroids and<br>hormone<br>replacement as<br>clinically indicated | Monitor participants for signs and symptoms of endocrinopathies |
| Nephritis and<br>Renal dysfunction | Grade 2 Grade 3 or 4 | Withhold Permanently discontinue | Administer corticosteroids (prednisone 1 – 2 mg/kg or equivalent) followed by taper | Monitor changes of renal function |
| All other immune-related | Intolerable/persistent<br>Grade 2 | Withhold | Based on type and severity of AE, | Ensure adequate evaluation to confirm etiology and/or exclude |
| AEs | Grade 3 | Withhold or<br>discontinue based on<br>the type of event.<br>Events that require<br>discontinuation<br>include, but are not<br>limited to:<br>Guillain-Barré<br>Syndrome,<br>encephalitis | administer<br>corticosteroids | other causes |
| | Grade 4 or recurrent<br>Grade 3 | Permanently discontinue | | |

AE = adverse event; ALT = alanine aminotransferase; AST = aspartate aminotransferase; CTCAE = Common Terminology Criteria for Adverse Events; GI = gastrointestinal; IRAE = immune-related adverse event; IV = intravenous; ULN = upper limit of normal.


APPENDIX E. NATIONAL COMPREHENSIVE CANCER NETWORK AND AMERICAN SOCIETY OF CLINICAL ONCOLOGY:
MANAGEMENT OF IMMUNOTHERAPY-RELATED TOXICITIES (IMMUNE CHECKPOINT INHIBITOR-RELATED TOXICITIES)


## **NCCN: Continuing Education**

**Target Audience:** This activity is designed to meet the educational needs of oncologists, nurses, pharmacists, and other healthcare professionals who manage patients with cancer.

#### **Accreditation Statements**

In support of improving patient care, National Comprehensive Cancer Network (NCCN) is jointly accredited by the Accreditation Council for Continuing Medical Education (ACCME), the Accreditation Council for Pharmacy Education (ACPE), and the American Nurses Credentialing Center (ANCC), to provide continuing education for the healthcare team.

**Medicine (ACCME):** NCCN designates this journal based CME ac tivity for a maximum of 1.0 *AMA PRA Category 1 Credit*<sup>™</sup>. Physicians should claim only the credit commensurate with the extent of their participation in the activity.

**Nursing (ANCC):** NCCN designates this educational activity for a maximum of 1.0 contact hour.

**Pharmacy (ACPE):** NCCN designates this knowledge based continuing education activity for 1.0 contact hour (0.1 CEUs) of continuing education credit. UAN: JA4008196 0000 20 004 H01 P

All clinicians completing this activity will be issued a certificate of participation. To participate in this journal CE activity: (1) review the educational content; (2) take the posttest with a 66% minimum passing score and complete the evaluation at https://education.nccn.org/node/86963; and (3) view/print certificate.

Pharmacists: You must complete the posttest and evaluation within 30 days of the activity. Continuing pharmacy education credit is reported to the CPE Monitor once you have completed the posttest and evalu ation and claimed your credits. Before completing these requirements, be sure your NCCN profile has been updated with your NAPB e profile ID and date of birth. Your credit cannot be reported without this in formation. If you have any questions, please e mail education@nccn.org.

Release date: March 10, 2020; Expiration date: March 10, 2021

#### Learning Objectives:

Upon completion of this activity, participants will be able to:

- Integrate into professional practice the updates to the NCCN Guidelines for Management of Immunotherapy Related Toxicities
- Describe the rationale behind the decision making process for de veloping the NCCN Guidelines for Management of Immunotherapy Related Toxicities

## **Disclosure of Relevant Financial Relationships**

The NCCN staff listed below discloses no relevant financial relationships:

Kerrin M. Rosenthal, MA; Kimberly Callan, MS; Genevieve Emberger Hartzman, MA; Erin Hesler; Kristina M. Gregory, RN, MSN, OCN; Rashmi Kumar, PhD; Karen Kanefield; and Kathy Smith.

#### Individuals Who Provided Content Development and/or Authorship Assistance:

John A. Thompson, MD, Panel Chair, has disclosed that he receives honoraria from AstraZeneca Pharmaceuticals LP; is a scientific advisor for and has equity interest/stock options in Alpine Immune Sciences; and receives consulting fees from Calithera Biosciences, Inc. and Synthorx, Inc.

Bryan J. Schneider, MD, Panel Vice Chair, has disclosed that he receives grant/research support from Bristol-Myers Squibb Company, Genentech, Inc., and Incyte Corporation.

Julie Brahmer, MD, Panel Member, has disclosed that she receives consulting fees from Amgen Inc., AstraZeneca Pharmaceuticals LP, Bristol-Myers Squibb Company, Genentech, Inc., Merck & Co., Inc., and Syndax Pharmaceuticals Inc.; and she receives grant/research support from Bristol-Myers Squibb Company.

Philippe Armand, MD, PhD, Panel Member, has disclosed that he receives consulting fees from ., Merck & Co., Inc., Bristol-Myers Squibb Company, Pfizer Inc., Affimed, Adaptive Biotechnologies Corp., Infinity Pharmaceuticals, ADC Therapeutics, Celgene Corporation, MorphoSys AG, Daiichi Sankyo, Inc., Miltenyi Biotec; receives grant/research support from Merck & Co., Inc., Bristol-Myers Squibb Company, Affimed, Adaptive Biotechnologies Corp., Roche, Tensha Therapeutics, Otsuka Pharmaceutical Co., Ltd, Sigma-Tau Pharmaceuticals, Inc., Genentech, Inc., and IGM Biosciences, Inc.; and receives honoraria from Merck & Co., Inc. and Bristol-Myers Squibb Company.

Marianne Davies, DNP, RN, AOCNP, Panel Member, has disclosed that she is on the product/speakers bureau for AstraZeneca Pharmaceuticals LP, Bristol-Myers Squibb Company, Genentech, Inc., and Merck & Co., Inc.

Marc S. Ernstoff, MD, Panel Member, has disclosed that he receives consulting fees from Bristol-Myers Squibb Company, Alkermes plc, and ImmuNext Inc.; and receives grant/research support from EMD Serono, Merck & Co., Inc., and Alkermes plc.

Jeffrey A. Sosman, MD, Panel Member, has disclosed that he is a scientific advisor for and receives honoraria from Bristol-Myers Squibb Company, and receives consulting fees from Genentech, Inc.

Alyse Johnson-Chilla, MS, Guidelines Coordinator, NCCN, has disclosed that she has no relevant financial relationships.

Griselda Zuccarino-Catania, PhD, Oncology Scientist/Medical Writer, NCCN, has disclosed that her spouse is employed by Janssen Pharmaceuticals, Inc.

Anita Engh, PhD, Oncology Scientist/Medical Writer, NCCN, has disclosed that she has no relevant financial relationships.

To view all of the conflicts of interest for the NCCN Guidelines panel, go to NCCN.org/disclosures/guidelinepanellisting.aspx.

This activity is supported by educational grants from AstraZeneca; Celgene Corporation; Coherus BioSciences; Genentech, a member of the Roche Group; and TESARO, a GSK Company. This activity is supported in part by an educational grant from Bayer Healthcare Pharmaceuticals. This activity is supported by an independent medical education grant from Bristol-Myers Squibb. This activity is supported by a medical education grant from Exelixis, Inc. This activity is supported by an independent educational grant from Merck & Co., Inc.

# Management of Immunotherapy-Related Toxicities, Version 1.2020

## Featured Updates to the NCCN Guidelines

John A. Thompson, MD¹,\*; Bryan J. Schneider, MD²,\*; Julie Brahmer, MD³,\*; Stephanie Andrews, MS, ANP BC⁴; Philippe Armand, MD, PhD⁵,\*; Shailender Bhatia, MD¹; Lihua E. Budde, MD, PhD⁶; Luciano Costa, MD, PhD⁶; Marianne Davies, DNP, RN, AOCNP®,\*; David Dunnington, MA⁰; Marc S. Ernstoff, MD¹⁰,\*; Matthew Frigault, MD¹¹; Benjamin H. Kaffenberger, MD¹²; Matthew Lunning, DO¹³; Suzanne McGettigan, MSN, CRNP¹⁴; Jordan McPherson, PharmD, MS, BCOP¹⁵; Nisha A. Mohindra, MD¹⁶; Jarushka Naidoo, MD³; Anthony J. Olszanski, MD, RPh¹⁻; Olalekan Oluwole, MD¹®; Sandip P. Patel, MD¹⁰; Nathan Pennell, MD, PhD²⁰; Sunil Reddy, MD²¹; Mabel Ryder, MD²²; Bianca Santomasso, MD, PhD²³; Scott Shofer, MD, PhD²⁴; Jeffrey A. Sosman, MD¹⁶,\*; Yinghong Wang, MD, PhD²⁵; Ryan M. Weight, DO, MS²⁶; Alyse Johnson Chilla, MS²⁷,\*; Griselda Zuccarino Catania, PhD²⁷,\*; and Anita Engh, PhD²⁷,\*

#### **ABSTRACT**

The NCCN Guidelines for Management of Immunotherapy Related Toxicities provide interdisciplinary guidance on the management of immune related adverse events (irAEs) resulting from cancer immunotherapy. These NCCN Guidelines Insights describe symptoms that may be caused by an irAE and should trigger further investigation, and summarize the NCCN Management of Immunotherapy Related Toxicities Panel discussions for the 2020 update to the guidelines regarding immune checkpoint inhibitor related diarrhea/colitis and cardiovascular irAEs.

J Natl Compr Canc Netw 2020;18(3):230–241 doi: 10.6004/jnccn.2020.0012

<sup>1</sup>Fred Hutchinson Cancer Research Center/Seattle Cancer Care Alliance; <sup>2</sup>University of Michigan Rogel Cancer Center; <sup>3</sup>The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; <sup>4</sup>Moffitt Cancer Center; <sup>5</sup>Dana-Farber/Brigham and Women's Cancer Center; <sup>6</sup>City of Hope National Medical Center; <sup>7</sup>O'Neal Comprehensive Cancer Center at UAB; <sup>8</sup>Yale Cancer Center/Smilow Cancer Hospital; 9Patient Advocate; 10Roswell Park Comprehensive Cancer Center; 11 Massachusetts General Hospital Cancer Center; <sup>12</sup>The Ohio State University Comprehensive Cancer Center - James Cancer Hospital and Solove Research Institute; <sup>13</sup>Fred & Pamela Buffett Cancer Center; 14Abramson Cancer Center at the University of Pennsylvania; <sup>15</sup>Huntsman Cancer Institute at the University of Utah; <sup>16</sup>Robert H. Lurie Comprehensive Cancer Center of Northwestern University; <sup>17</sup>Fox Chase Cancer Center; <sup>18</sup>Vanderbilt-Ingram Cancer Center; <sup>19</sup>UC San Diego Moores Cancer Center; <sup>18</sup>Vanderbilt-Ingram Cancer Center; <sup>19</sup>UC San Diego Moores Cancer Center; <sup>20</sup>Case Comprehensive Cancer Center/University Hospitals Seidman Cancer Center and Cleveland Clinic Taussig Cancer Institute; 21 Stanford Cancer Institute; <sup>22</sup>Mayo Clinic Cancer Center; <sup>23</sup>Memorial Sloan Kettering Cancer Center; <sup>24</sup>Duke Cancer Institute; <sup>25</sup>The University of Texas MD Anderson Cancer Center; <sup>26</sup>University of Colorado Cancer Center; and <sup>27</sup>National Comprehensive Cancer Network.

#### NCCN CATEGORIES OF EVIDENCE AND CONSENSUS

**Category 1:** Based upon high level evidence, there is uniform NCCN consensus that the intervention is appropriate.

**Category 2A:** Based upon lower level evidence, there is uni form NCCN consensus that the intervention is appropriate.

**Category 2B:** Based upon lower level evidence, there is NCCN consensus that the intervention is appropriate.

**Category 3:** Based upon any level of evidence, there is major NCCN disagreement that the intervention is appropriate.

All recommendations are category 2A unless otherwise noted.

Clinical trials: NCCN believes that the best management of any patient with cancer is in a clinical trial. Participation in clinical trials is especially encouraged.

#### **PLEASE NOTE**

The NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®) are a statement of evidence and consensus of the authors regarding their views of currently accepted approaches to treatment. The NCCN Guidelines Insights highlight important changes in the NCCN Guidelines recommendations from previous versions. Colored markings in the algorithm show changes and the discussion aims to further the understanding of these changes by summarizing salient portions of the panel's discussion, including the literature reviewed.

The NCCN Guidelines Insights do not represent the full NCCN Guidelines; further, the National Comprehensive Cancer Network® (NCCN®) makes no representations or warranties of any kind regarding their content, use, or application of the NCCN Guidelines and NCCN Guidelines Insights and disclaims any responsibility for their application or use in any way.

# The complete and most recent version of these NCCN Guidelines is available free of charge at NCCN.org.

© National Comprehensive Cancer Network, Inc. 2020. All rights reserved. The NCCN Guidelines and the illustrations herein may not be reproduced in any form without the express written permission of NCCN.

<sup>\*</sup>Provided content development and/or authorship assistance.

#### PRINCIPLES OF ROUTINE MONITORING FOR IMMUNE-CHECKPOINT INHIBITORS

| Pre-Therapy Assessment <sup>a</sup> | Monitoring Frequency <sup>b</sup> | Evaluation for Abnormal Findings/Symptoms |
|---|---|---|
| Clinical - Physical examination - Comprehensive patient history of any autoimmune/organ-specific disease, endocrinopathy, or infectious disease - Neurologic examination - Bowel habits (typical frequency/consistency) | Clinical exam at each visit with adverse event (AE) symptom assessment | Follow-up testing based on findings, symptoms |
| Imaging Cross-sectional imaging Brain MRI if indicated | Periodic imaging as indicated | Follow-up testing as indicated based on imaging findings |
| General bloodwork CBC with differential Comprehensive metabolic panel | Repeat prior to each treatment or every 4 weeks during immunotherapy, then in 6–12 weeks or as indicated | HbA1c for elevated glucose |
| Dermatologic (ICI_DERM-1) • Examination of skin and mucosa if history of immune-related skin disorder | Conduct/repeat as needed based on symptoms | Monitor affected BSA and lesion type; photographic documentation. Skin biopsy if indicated. |
| Pancreatic (ICI_ENDO-1) • Baseline testing is not required. | No routine monitoring needed if asymptomatic | Amylase, lipase, and consider abdominal CT with contrast or MRCP for suspected pancreatitis. |
| Thyroid (ICI_ENDO-2) • Thyroid-stimulating hormone (TSH), free thyroxine (T4) <sup>C</sup> | Every 4–6 weeks during immunotherapy, then follow-up every 12 weeks as indicated | Total T3 and free T4 if abnormal thyroid function suspected. |
| Adrenal/Pituitary (ICI_ENDO-4) • Adrenal: Serum cortisol (morning preferred) <sup>C</sup> • Pituitary: TSH, free thyroxine (T4) <sup>C</sup> | Repeat prior to each treatment or every 4 weeks during immunotherapy, then follow-up every 6–12 weeks | Luteinizing hormone (LH), follicle-stimulating hormone (FSH), testosterone (males), estradiol (females), adrenocorticotropic hormone (ACTH) |
| Pulmonary (ICI_PULM-1) • Oxygen saturation (resting and with ambulation) • Pulmonary function tests (PFTs) for high-risk patients | Repeat oxygen saturation tests based on symptoms | Chest CT with contrast to evaluate for pneumonitis, biopsy if needed to exclude other causes. |
| Cardiovascular (ICL_CARDIO-1) Consider baseline EKG Individualized assessment in consultation with cardiology as indicated | Consider periodic testing for those with abnormal baseline or symptoms | Individualized follow-up in consultation with cardiology as indicated |
| Musculoskeletal (ICI_MS-1) • Joint examination/functional assessment as needed for patients with pre-existing disease | No routine monitoring needed if asymptomatic | Consider rheumatology referral. Depending on clinical situation, consider C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), or creatine phosphokinase (CPK) |

<sup>&</sup>lt;sup>a</sup> Prior to initiating treatment, counsel patients and caregivers on the warning signs and symptoms of immune-related adverse events (irAEs). See Principles of Immunotherapy Patient Education (IMMUNO-B).

Version 1.2020 ® National Comprehensive Cancer Network, Inc. 2020. All rights reserved.

The NCCN Guidelines® and this illustration may not be reproduced in any form without the express written permission of NCCN.

IMMUNO-1

#### **Overview**

Immune checkpoints are part of the natural balance of the immune system to prevent autoimmunity and are exploited by cancer cells to suppress the immune response. Immune checkpoint inhibitors (ICIs) block proteins—namely PD-1, PD-L1, and CTLA-4—that allow tumor cells to evade detection and killing by T cells. <sup>1-6</sup> Since the FDA-approval of the CTLA-4 inhibitor ipilimumab in 2011, ICIs have become a treatment option for several advanced cancers. ICIs significantly improve overall survival and delay progression of tumors in patients with a variety of cancers. <sup>7</sup> Indications for ICIs have expanded dramatically and now include a wide array of cancer types. <sup>1-8</sup>

A major drawback of ICI therapy is the potential for immune-related adverse events (irAEs), which can affect any organ or tissue. The pharmacodynamics and pharmacokinetics of ICI immunotherapy differ greatly from those of cytotoxic chemotherapy or targeted anticancer therapy. Traditional cytotoxic chemotherapy often results in acute-onset emetic and myelosuppressive effects, whereas irAEs tend to be relatively delayed in onset and inflammatory or autoimmune in nature. Although the pathophysiology of ICI-related irAEs is not yet fully elucidated, knowledge regarding the role of immune checkpoint pathways in autoimmune disease provides

some clues. Many autoimmune diseases are related to failure of T-cell tolerance and subsequent uncontrolled activation of immune effector cells. Early- and lateronset irAEs may result from distinct mechanisms that have yet to be elucidated. Typical earlier-onset, common irAEs appear to involve generalized epithelial inflammation and may be observed in the form of rash, colitis, and pneumonitis. Later-onset irAEs, which are typically less common, tend to be more-localized, organspecific reactions. Research is ongoing into the specific mechanisms underlying irAEs associated with specific ICIs. The reported incidence of any-grade irAEs associated with single-agent ICI treatment ranges widely across agents and trials, from approximately 15% to 90%, 14,15 and patterns of toxicity may differ between specific ICI agents. 16 Severe irAEs leading to discontinuation of treatment have occurred in up to 13% of patients receiving anti-PD-1 monotherapy in clinical trials. 17-24 Although combination regimens offer the potential for enhanced efficacy, in general, observed toxicity with ICI-based combination regimens is greater than that for ICI monotherapy.

### **Recognizing Immune-Related Symptoms**

Onset of irAEs can be immediate or delayed by as much as 2 years, and can affect any organ system.<sup>25</sup> Early

bCloser monitoring may be required for patients with combination immunotherapy regimens. Refer to prescribing information for each individual immunotherapy agent for monitoring recommendations.

<sup>&</sup>lt;sup>c</sup> After first four doses of immunotherapy, only as clinically indicated.



Version 1.2020 © National Comprehensive Cancer Network, Inc. 2020. All rights reserved.

The NCCN Guidelines® and this illustration may not be reproduced in any form without the express written permission of NCCN.

ICI GI-1

recognition of symptoms and prompt intervention are key goals for the successful management of immunotherapy-related toxicity. When encountering one or more of these symptoms, asking appropriate questions can help discern whether the patient is experiencing a symptom due to disease progression, an infection, some other condition, or an irAE. Symptoms that may cause clinical suspicion of an irAE include (main symptoms are bold and underlined; associated symptoms are underlined; possible irAE type/diagnoses are in italics):

- Change in bowel pattern compared with baseline, especially if it is watery diarrhea, stool contains blood or mucus, or cramping or severe abdominal pain develop, may indicate *colitis*. However, blood in the stools and/or fever may be because of other causes of gastrointestinal bleeding, such as *infection* or *peptic ulcer disease* or *bleeding due to tumor*.
- <u>Cough</u> may be due to an upper respiratory infection, but especially if the cough is dry or is coupled with shortness of breath, it could indicate *pneumonitis*.
- <u>Headaches</u> can be indicative of brain metastases, but when presenting with <u>fatigue</u>, <u>visual symptoms</u>, <u>nausea</u>, and other symptoms, may be indicative of *hypophysitis*

- (inflammation of the pituitary). <sup>26</sup> <sup>28</sup> Headaches may also be indicative of *meningitis* when coupled with a <u>stiff neck</u>, <u>photophobia</u>, <u>nausea</u>, or <u>fever</u>. Headaches can also be indicative of *encephalitis* if coupled with <u>fever</u>, <u>tiredness</u>, <u>confusion</u>, <u>mood change</u>, <u>memory problems</u>, <u>stiff neck</u>, and other symptoms. Headaches, <u>head pain</u>, and <u>scalp tenderness</u>, may be indicative of *giant cell arteritis*.
- Nausea is a common symptom that can accompany certain cancer therapies. Nausea with abdominal pain/bloating could indicate pancreatitis. Nausea that occurs during infusion of an ICI, accompanied by fever/chills, hypertension, hypotension, sweating, myalgia, cough, or shortness of breath, may indicate an infusion-related reaction.
- Rashes are very common and may be accompanied by <a href="itteling">itching</a> that can lead to scratching and severe *skin toxicities* causing edema, oozing, papulation, excoriations, <a href="lichenification">lichenification</a>, which may indicate *bullous dermatitis*, or separation of the dermis, a sign of *Stevens-Johnson syndrome/toxic epidermal necrolysis (SJS/TEN)*.
- <u>Fatigue</u> is a common symptom that alone or coupled with <u>weight change</u>, <u>nausea</u>, or other nonspecific symptoms may indicate a *thyroid disorder*,<sup>26</sup> *hypophysitis*, or,





<sup>9</sup> See Principles of Immunosuppression (IMMUNO-A)

Version 1.2020 © National Comprehensive Cancer Network, Inc. 2020. All rights reserved.
The NCCN Guidelines® and this illustration may not be reproduced in any form without the express written permission of NCCN

ICI\_GI-2

rarely, adrenal insufficiency.<sup>28</sup> Fatigue with tachycardia, palpitations, increased stool frequency, and other symptoms may be thyrotoxicosis.27 Fatigue accompanied by nausea, chest pain, shortness of breath, arrhythmias, and other potentially nonspecific symptoms may be indicative of *myocarditis*. However, fatigue may also be attributed to depression, an infection, disease progression, a hematologic abnormality, or another condition.

- Muscle or joint pain may be indicative of musculoskeletal toxicities. Muscle pain alone or with fatigue, chest pain, and shortness of breath may be due to a cardiac toxicity, because myocarditis may occur concurrently with myositis.29 32
- Muscle weakness may be indicative of neurologic toxicities, such as Guillain-Barré syndrome, or, if coupled with vision changes, myasthenia gravis. Myasthenia gravis related to immunotherapy may be associated with myositis and myocarditis.31,33,34
- Weight loss and nausea may be due to disease progression, but may also indicate a hepatic toxicity or an endocrine toxicity.

For many patients, routine laboratory monitoring, comparisons to baseline, and targeted questions by the treating healthcare providers will help identify some of the less common but serious irAEs. The primary facets of irAE management include early recognition and grading of toxicity, immunosuppression, and individualized modification to ICI administration. See the complete version of the NCCN Guidelines (available at NCCN.org) for management strategies for these and other ICI-related irAEs updated for 2020.

## 2020 Updates to the NCCN Guidelines

The NCCN Guidelines for Management of Immunotherapy-Related Toxicities provide guidance on the management of irAEs resulting from cancer immunotherapy, specifically ICI and CAR T-cell therapies. During the meeting to update the guidelines for 2020, the panel discussed updates to the management of many irAEs. These NCCN Guidelines Insights highlight recommendations for the assessment and treatment of ICI-related irAEs related to the gastrointestinal and cardiovascular systems.

#### Gastrointestinal Adverse Events: Diarrhea/Colitis

The most common gastrointestinal irAE presents as diarrhea and/or symptoms of colitis, which include watery

f More than 6 bowel movements above baseline per day, colitis symptoms, interfering with ADLs, hemodynamic instability, hospitalization, other serious complications (eg, ischemic bowel, perforation, toxic mega-colon).

h See Principles of Immunotherapy Rechallenge (IMMUNO-C).

k Treat until symptoms improve to Grade ≤1 then taper over <4–6 weeks. In cases where infliximab or vedolizumab is used, an attempt to taper steroids in <4 weeks

Duration of therapy with tumor necrosis factor alpha (TNF-alpha) blockers or integrin blocker is not clearly defined; evidence supports up to three doses (at weeks 0, 2, and 6) and is associated with reduced recurrence rates. Repeat end optional. See Principles of Immunosuppression (IMMUNO-A).

Man FDA-approved biosimilar is an appropriate substitute for infliximab. Repeat endoscopy to assess endoscopic healing may be helpful to guide colitis treatment duration, but

Obtain TB test before receiving first dose of infliximab or vedolizumab.Treatment does not need to be held for results.

<sup>&</sup>lt;sup>o</sup> Fecal transplantation may be considered for immunosuppressant refractory colitis based on institutional availability and expertise



- a Myocarditis symptoms are nonspecific. It is rare, but potentially severe, not viral in etiology, associated with myositis/myasthenia gravis, and is more common with combination therapy. In fatal cases, conduction abnormalities were mode of death and ejection fraction was preserved
- b No evidence specific to immunotherapy-related myocarditis; recommendations drawn from other causes of myocarditis.
- <sup>c</sup> Arrhythmia, significant echo findings without hypotension, cardiac markers >ULN.
- <sup>d</sup> Arrhythmia, hemodynamic instability (hypotension/cardiomyopathy), cardiac markers >3xULN. <sup>e</sup> See Principles of Immunosuppression (IMMUNO-A).
- f See Principles of Immunotherapy Rechallenge (IMMUNO-C).
- <sup>9</sup>Successful outcomes have been reported with other suppressive agents, such as alemtuzumab or abatacept
- h An FDA-approved biosimilar is an appropriate substitute for infliximab
- Total dosing should be 2 g/kg, administered in divided doses per package insert
- Mycophenolate mofetil treatment (0.5–1 g every 12 hours).

Version 1.2020 © National Comprehensive Cancer Network, Inc. 2020. All rights reserved.

The NCCN Guidelines® and this illustration may not be reproduced in any form without the express written permission of NCCN.

ICI\_CARDIO-1

diarrhea, cramping, urgency, abdominal pain, blood or mucus in the stool, fever, or nocturnal bowel movements. Diarrhea and/or colitis are the second most commonly reported AEs with ICIs, and symptoms typically develop within 6 to 8 weeks of starting treatment. 35,36 These gastrointestinal irAEs have been reported more frequently with anti-CTLA-4 monotherapy than with PD-1/PD-L1 inhibitors. In studies of CTLA-4 blockade, diarrhea has been reported in up to half of patients, with incidence typically reported between 30% and 40%. 14,37 The highest rates of ICI-mediated diarrhea/colitis have been observed with the addition of a PD-1/PD-L1 inhibitor to CTLA-4 blockade.38-40

### Detection, Initial Assessment, and Grading of Diarrhea/Colitis

To facilitate early detection of diarrhea/colitis, patient education is key. It is important to determine the patient's baseline bowel habits prior to initiation of immunotherapy. Patients are encouraged to report changes in their bowel habits to the treatment team in order to facilitate early detection of colitis that may occur before the next scheduled clinic visit (see IMMUNO-1, page 232). Most cases present as diarrhea (increased frequency of bowel movements), but as described earlier, a variety of other colitis symptoms often occur. Severity of the diarrhea (ie, increase in number bowel movements per day compared with baseline) and the presence and severity of other colitis symptoms determine the grade of the gastrointestinal irAE (Table 1). Hemodynamic instability and life-threatening complications (eg, ischemic bowel, perforation, toxic mega-colon) may be associated with high-grade gastrointestinal irAEs. Table 1 shows grading for these adverse events, based on elements from CTCAE version 5.0 (colitis, enterocolitis, diarrhea),41 Brahmer et al,42 and additions from the NCCN Panel (see ICI GI-1 footnotes, page 233).

Stool evaluation to rule out infectious etiology, specifically Clostridium difficile, ova, parasites, and viral pathogens, is an important element of workup for patients with suspected immunotherapy-related diarrhea and/or colitis. For patients presenting with grade 1 diarrhea (increase of <4 bowel movements per day above baseline) and no symptoms of colitis, some panel members defer stool testing until diarrhea has persisted and not improved with conservative treatment (loperamide or diphenoxylate for 2–3 days), or symptoms

## Table 1. Grading<sup>a</sup> for Colitis/Diarrhea<sup>b</sup>

#### erms

**Diarrhea:** increase in frequency and/or loose or watery bowel movements

Colitis: inflammation of the colon

Enterocolitis: inflammation of the small and large intestines

#### Grade 1

- Increase of <4 bowel movements per day above baseline</li>
   Mild increase in ostomy output compared with baseline
- No symptoms of colitis (watery diarrhea, cramping, urgency, abdominal pain, blood and mucus in the stool, fever, nocturnal bowel movements)

#### Grade 2

- Increase of 4-6 bowel movements per day above baseline
- Moderate increase in ostomy output compared with baseline
- Mild/moderate colitis symptoms: watery diarrhea, cramping, urgency, abdominal pain, blood and mucus in the stool, fever, nocturnal bowel movements
- Limiting instrumental ADLs<sup>d</sup>

#### Grade 3

- Increase of >6 bowel movements per day above baseline
- Severe increase in ostomy output compared with baseline
- Severe colitis symptoms: watery diarrhea, incontinence, cramping, urgency, abdominal pain, blood and mucus in the stool, fever, ileus, nocturnal bowel movements, peritoneal signs
- Limiting self-care ADLs
- Hemodynamic instability
- Hospitalization indicated

#### Grade 4

- Same as grade 3, but with:
- Other serious/life-threatening complications (eg, ischemic bowel, perforation, toxic mega-colon)
- Urgent intervention indicated

Abbreviation: ADLs, activities of daily living.

<sup>a</sup>For all adverse events, grade 5 is defined as death.

<sup>b</sup>Definitions incorporate elements from CTCAE version 5.0 (colitis,

enterocolitis, diarrhea), $^{41}$  Brahmer et al, 2018, $^{42}$  plus additions from the NCCN Panel (ICI GI-1 footnotes, page 233).

dInstrumental ADLs refer to preparing meals, shopping for groceries or clothes, managing money, etc.

eSelf-care ADLs include bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

have progressed (frequency of bowel movements increased and/or colitis symptoms developed). Blood or mucus in the stools, fever, and/or other symptoms of colitis (watery diarrhea, cramping, urgency, abdominal pain, nocturnal bowel movements) should prompt a thorough workup for infection, including stool evaluation. Patients presenting with blood in the stool should also be evaluated for other causes of gastrointestinal bleeding, including peptic ulcer disease and malignant bleeding, among others (eg, diverticulosis, angiodysplasia, hemorrhoids, ischemia). Diarrhea/colitis associated with immunotherapy can rapidly increase in severity, and therefore therapy to manage these gastrointestinal irAEs can be initiated while awaiting test results.

Measurement of fecal lactoferrin and calprotectin, 2 markers of inflammation, should also be considered as part of initial workup, depending on institutional availability. Calprotectin provides a quantitative measure of inflammation; low levels indicate mild inflammation or normal endoscopy and high levels correlate with ulceration.<sup>43</sup> Fecal lactoferrin is a noninvasive, qualitative biomarker that can predict colitis risk.<sup>44,45</sup>

For patients who present with diarrhea/colitis grade 2 or higher (as defined in Table 1), abdominal/pelvic CT with contrast and gastrointestinal consultation for further evaluation (ie, colonoscopy or flexible sigmoidoscopy ± esophagogastroduodenoscopy [EGD] with biopsy) should be considered. Symptom-based grading (listed in Table 1) may guide prompt initiation of therapy (eg, steroids); however, imaging and biopsy results can help establish the etiology of the problem and assess the likelihood that more aggressive management approaches will be needed. Although retrospective case reviews suggest that symptom grade may not correlate with colitis severity as observed by endoscopy and histology, 46,47 results from a recent retrospective study suggest that lactoferrin results may be used to inform prioritization of endoscopy.43 This study found that among patients with immune-mediated diarrhea/ colitis, lactoferrin levels were strongly correlated with inflammation observed by endoscopy (70% sensitivity), and even more strongly correlated with inflammation detected by histologic evaluation of endoscopy biopsy specimens (90% sensitivity).43 Histologic findings were correlated with the need for intravenous steroids and/or infliximab/vedolizumab for irAE management.43 Early endoscopy, defined as ≤7 days after onset of immunemediated diarrhea/colitis compared with >7 days, was associated with significantly shorter duration of symptoms (47 vs 19 days; P .026) and shorter steroid treatment duration (49 vs 74 days; P .053), 43 presumably because earlier endoscopy triggered earlier initiation of management. Performing endoscopy ≤30 days from onset of diarrhea/colitis (vs >30 days) was associated with significantly shorter duration of steroid treatment, a trend toward shorter duration of symptoms, and a significant reduction in recurrence of symptoms (50% vs 21.8% of patients; P .001). Better outcomes for patients who undergo endoscopy within 30 days of onset may be due to the earlier initiation of infliximab/vedolizumab (15 vs 31 days from onset; P .030). Given the results of this recent study,43 early endoscopy with biopsy within the first 2 weeks of the onset of symptoms is strongly recommended for all patients with positive lactoferrin results, even those who have only grade 1 symptoms (per Table 1). Fever and tenderness upon abdominal examination may be an indication of bowel perforation warranting immediate imaging and treatment.

#### Management of Mild (Grade 1) Events

For patients presenting with mild diarrhea (grade 1, defined as an increase of <4 bowel movements per day) with no other symptoms of colitis (Table 1), the NCCN Guidelines recommend hydration, considering holding immunotherapy, and monitoring the patient closely to determine whether diarrhea is worsening or other

symptoms of colitis develop (see ICI GI-1, page 233). Loperamide or diphenoxylate/atropine may be used, although some panel members prefer to wait before starting, out of concern about obscuring signs of worsening diarrhea, which may delay initiation of treatment (eg, steroids) that actually reverses underlying immunotherapy-related inflammation, if present. If diarrhea persists or progresses, or no improvement is seen after 2 to 3 days of loperamide or diphenoxylate/atropine, tests for infections workup should be obtained and levels of fecal lactoferrin should be checked if not already done. Cases of grade 1 diarrhea (increase of <4 bowel movements per day) with no other symptoms of colitis, documented absence of infection, and a negative lactoferrin result, may be managed conservatively (hydration and loperamide or diphenoxylate/atropine), with the addition of mesalamine or cholestyramine, if necessary. If lactoferrin results are positive, however, endoscopy should be strongly considered, if not already performed, even if the only symptom is grade 1 diarrhea. Patients with a positive lactoferrin result and persistent/progressive diarrhea should be treated as those with moderate (grade 2) diarrhea/colitis (see next section), because these cases are likely to require more aggressive management, even if the diarrhea has not yet reached the grade 2 threshold (increase of  $\geq 4$  bowel movements per day above baseline) and no other colitis symptoms have yet developed.

## Tools for Management of Grade 2 or Higher Events

Corticosteroids are typically the first line of treatment of diarrhea/colitis of grade 2 or higher. In retrospective reviews of patients with ICI-related diarrhea/colitis, symptoms resolved with corticosteroid treatment in approximately half of individuals. However, for some cases, corticosteroids fail to control symptoms and the diarrhea/colitis may persist or worsen and become life-threatening in the absence of more aggressive management.

Infliximab is a monoclonal anti–tumor necrosis factor alpha (TNF- $\alpha$ ) antibody used for treating various autoimmune diseases, including Crohn's disease, ulcerative colitis, rheumatoid and psoriatic arthritis, and psoriasis.<sup>49–51</sup> Infliximab has become a commonly used agent for treating steroid-refractory irAEs that develop during ICI therapy.<sup>25,52</sup> Case studies report on the successful use of infliximab for treating severe, steroid-refractory colitis associated with ipilimumab.<sup>48,53,54</sup> An FDA-approved biosimilar is an appropriate substitute for infliximab.

Vedolizumab is an integrin antagonist that binds to  $\alpha 4\beta 7$  integrin, blocking its interaction with mucosal addressin cell adhesion molecule-1 (MAdCAM-1), inhibiting the migration of T cells across the endothelium into inflamed gastrointestinal tissues. Vedolizumab is currently indicated for treating gastrointestinal

inflammation due to ulcerative colitis and Crohn's disease. 55,56 Case reports have described the use of vedolizumab for the treatment of ICI-induced diarrhea/colitis. 56–58 Vedolizumab binds to gut homing lymphocytes and may provide more specific immune suppression for the inflamed gastrointestinal mucosa, thereby theoretically avoiding suppression of antitumor immune responses.

Introduction of either infliximab or vedolizumab within 10 days of onset of colitis can reduce the duration of symptoms and improve steroid taper success.<sup>59</sup> Treatment with ≥3 doses of infliximab or vedolizumab, and achieving endoscopic or histologic remission are associated with lower risk of colitis relapse. This is important because endoscopic remission is often a better predictor of a cure than clinical remission, in which cases repeat endoscopy may be helpful.

Case studies suggest that transplantation of fecal microbiota from healthy donors may resolve cases of diarrhea/colitis that are resistant to corticosteroids, infliximab, and vedolizumab.<sup>60</sup>

#### Management of Moderate (Grade 2) Diarrhea/Colitis

For moderate diarrhea/colitis (grade 2), defined as an increase of 4 to 6 bowel movements per day above baseline and/or mild to moderate symptoms of colitis (as detailed in Table 1), the NCCN Guidelines recommend holding immunotherapy and administering prednisone/methylprednisolone (1–2 mg/kg/d) (see ICI GI-1, page 233). If no improvement is noted within 2 to 3 days of starting steroid treatment, the NCCN Guidelines recommend continuing steroids and considering adding infliximab (or FDA-approved biosimilar) or vedolizumab, preferably within 2 weeks from onset of diarrhea. A tuberculosis test (blood test preferred) should be obtained before administering the first dose of infliximab or vedolizumab, although treatment can be initiated before results are received.

#### Management of Severe (Grade 3-4) Events

For severe diarrhea/colitis (grade 3–4), defined as an increase of >6 bowel movements per day above baseline and/or severe symptoms of colitis (Table 1), inpatient care should be considered if needed to provide adequate supportive care (see ICI GI-2, page 234). Intravenous methylprednisolone, 1 to 2 mg/kg/d, should be administered. After improvement in diarrhea/colitis is noted, the steroid dose may be tapered, usually over 4 to 6 weeks (see later discussion). For diarrhea/colitis related to ipilimumab, the NCCN panel recommends permanent discontinuation if serious or life-threatening diarrhea/colitis occurs. For diarrhea/colitis associated with PD-1/PD-L1 inhibitors, therapy should be held for grade 3, with consideration of rechallenge upon resolution of symptoms

below grade 1. The immunotherapy agent(s) responsible for immune-related grade 4 diarrhea/colitis should be permanently discontinued.

If no improvement is noted within 2 to 3 days on intravenous methylprednisolone (1–2 mg/kg/d), the NCCN Guidelines recommend continuing steroids and strongly considering adding infliximab (or FDA-approved biosimilar) or vedolizumab, preferably within 2 weeks of onset, especially for patients with high-risk endoscopic features.<sup>43</sup> Fecal transplantation may be considered for colitis refractory to immunosuppressant therapy, based on institutional availability and expertise.<sup>60</sup>

# Duration of Treatment of Immune-Related Diarrhea/Colitis

For disease monitoring after receiving colitis treatment, checking the levels of calprotectin provides a quantitative measure of inflammation; low levels indicate mild inflammation or normal endoscopy and high levels correlate with ulceration.<sup>43</sup> Repeat endoscopy to assess endoscopic healing may be helpful to guide colitis treatment duration, but is optional. Endoscopy has revealed colonic ulcerations more commonly in steroid-refractory cases.<sup>36,46,48</sup>

Retrospective analysis of patients with refractory diarrhea/colitis found higher infection rates among patients treated with long-duration steroids (>30 days). Long-duration corticosteroid without infliximab was associated with increased infection risk compared with short-duration steroid plus infliximab, suggesting that earlier nonsteroid immunosuppressive therapy may confer better outcomes.<sup>47</sup> If a systemic corticosteroid is given, treatment should be continued until symptoms improve to grade 1 or better, then dose tapered over 4 to 6 weeks. In cases in which infliximab or vedolizumab is used, a shorter taper may help minimize the complication of infection, provided that the diarrhea/ colitis (or other concomitant irAEs) does not worsen during the taper. Intravenous methylprednisolone should be converted to oral prednisone when appropriate.

The duration of therapy with TNF- $\alpha$  blocker (infliximab) or integrin blocker (vedolizumab) is not clearly defined. Evidence supports the use of up to 3 doses (at weeks 0, 2, and 6) to reduce risk of recurrence and increase likelihood of endoscopic/histologic remission.<sup>59</sup>

#### Cardiovascular Adverse Events

Efforts to characterize cardiac irAEs associated with ICI therapy have begun to provide a better understanding of ICI-associated myocarditis. Case series reveal a variety of potential manifestations of cardiovascular irAEs, including myocarditis, pericarditis, arrhythmias, cardiomyopathy, cardiac fibrosis, heart failure, and cardiac arrest.<sup>61-65</sup> Data collected over

4 years from 8 sites revealed 35 cases of ICI-mediated myocarditis, which were compared with a sample of patients on ICI therapy without myocarditis.<sup>62</sup> Prevalence was 1.14% in this patient population, with a median onset of 34 days from initiation of treatment. However, recent evidence suggests that ICI-associated cardiovascular toxicity, myocarditis in particular, is more common than initially thought.<sup>33,34,62,66</sup>

Myocarditis symptoms are nonspecific, such as myalgia, shortness of breath, and chest pain, which could also be attributed to pneumonitis or other irAEs.<sup>29</sup> It is rare, but potentially severe, associated with myositis/myasthenia gravis, and is more common with anti–CTLA-4/anti–PD-(L)1 combination therapy. A recent report analyzed a total of 40 case reports describing cardiac irAEs and found that even with rapid assessment and initiation of immunosuppression, mortality was still high at 23%.<sup>67</sup> In fatal cases, conduction abnormalities were the mode of death and ejection fraction was preserved.

Cardiac irAEs have been associated with ipilimumab, pembrolizumab, and nivolumab. Based on multicenter registry data, myocarditis was observed more often in patients receiving combination ICI therapy and in those with diabetes.<sup>62</sup> Recent analysis of the WHO database revealed 101 individual case safety reports of severe myocarditis following initiation of ICI therapy.<sup>34</sup> Of these cases, 57% had received anti PD-1 monotherapy and 27% received combination PD-1/PD-L1 plus CTLA-4 inhibitor. For cases with available dosing information (n 59), 64% (n 38) had received only 1 or 2 ICI doses at the time of toxicity onset. Concurrent severe irAEs, most commonly myositis and myasthenia gravis, were reported for 42% of cases. Data on cardiovascular comorbidities were not available, but only 25% of patients with myocarditis were on medication to treat cardiovascular disease or diabetes.34

Preexisting cardiovascular pathology was identified in more than half of patients (5/8) in one case series. <sup>61</sup> Co-occurrence with noncardiac irAEs was also observed in >50% of patients. Corticosteroids and/or supportive care measures were helpful to improve symptoms in most cases, although permanent cardiotoxicity and fatalities also occurred despite intervention. <sup>61</sup> Myositis and myocarditis were observed to co-occur in a recent study of ICI-related fatalities. Notably, myasthenia gravis also co-occurred in 10% of fatal myocarditis cases. <sup>33</sup> Case reports of ICI-related myocarditis have reported irAE flare during steroid taper or ICI rechallenge. <sup>68,69</sup>

#### Management

Baseline EKG and individualized assessment in consultation with cardiology should be considered as indicated. Periodic testing should be considered for patients with abnormal baseline or symptoms (see IMMUNO-1, page 232).

Once a cardiac irAE is suspected, immediate cardiology consultation and intensive care unit–level monitoring is recommended (see ICI CARDIO-1, page 235). Assessment should include telemetry monitoring and electrocardiogram. Recommended laboratory testing includes cardiac biomarkers (creatine kinase and troponin levels) and inflammatory biomarkers (erythrocyte sedimentation rate, C-reactive protein level, and WBC count). To rule out other potential causes, evaluation may include viral titers, echocardiogram, or biopsy in the case of severe symptoms. When feasible, cardiac MRI may provide additional diagnostic information.<sup>70</sup>

Table 2 summarizes grading for cardiovascular adverse events that may be associated with ICI therapy, based on elements from CTCAE version 5.0 (myocarditis, pericarditis, ventricular arrhythmia),<sup>41</sup> Brahmer et al,<sup>42</sup> and additions from the NCCN Panel (see ICI CARDIO-1 footnotes, page 235). In the setting of severe (grade 3) cardiac irAE, arrhythmia may be accompanied by significant echocardiogram findings without hypotension, and cardiac biomarkers above the upper limit of normal (ULN). Life-threatening (grade 4) cardiac irAEs are denoted by arrhythmia, hemodynamic instability, and cardiac biomarkers >3 times the ULN. Transient pacemaker may be recommended in patients with arrhythmia.<sup>67</sup> Immunotherapy should be permanently discontinued for any grade 3 or 4 cardiovascular irAEs. The panel recommends methylprednisolone pulse dosing (1 g/d for 3–5 days). In a multicenter registry report, corticosteroids were administered in 89% of cases with myocarditis, with high-dose steroids resulting in better treatment response.<sup>62</sup> Elevated troponin and higher rates of major adverse cardiac events, which were defined as "the composite of cardiovascular death, cardiogenic shock, cardiac arrest, and hemodynamically significant complete heart block," were observed more commonly among patients who were treated with lower-dose corticosteroid.62 The NCCN Panel recommends treating with steroids until cardiac function returns to baseline, then dose taper over 4 to 6 weeks.

Beyond treatment with high-dose steroids, there are few data to suggest the optimal subsequent therapy should steroids fail. Treatment options for both severe (grade 3) or life-threatening cases (grade 4) are the same given the rapid progression of cardiac irAE. If no improvement is noted within 24 hours, the addition of other potent immunosuppressive agents should be considered, such as antithymocyte globulin (ATG),<sup>62,67,71–73</sup> infliximab<sup>61,67,71,74</sup> or an FDA-approved biosimilar, intravenous immunoglobulin (IVIG),<sup>67,73,75</sup> or mycophenolate.<sup>76</sup>

ATG is a polyclonal antibody derived from lymphoid cell immunized horses or rabbits, which reverses immunotoxicity by inducing T-cell depletion. Data supporting use of ATG to treat myocarditis and arrhythmia

#### Table 2. Grading<sup>a</sup> for Select Cardiovascular Events<sup>b</sup>

#### Terms

Myocarditis: inflammation of the muscle tissue of the heart

Pericarditis: irritation to the layers of the pericardium (the
protective sac around the heart)

Other cardiovascular irAEs: arrhythmias, impaired ventricular function, conduction abnormalities

Grade 1 • Asymptomatic

- Abnormal cardiac biomarkers (creatine kinase, troponin)
- Abnormal ECG or physical findings (eg, rub) consistent with pericarditis
- Grade 2
- Mild symptoms or symptoms with moderate activity or exertion: may include chest pain, myalgia, dyspnea, arrhythmia, palpitations, peripheral edema, pleural effusion, fatigue
- Abnormal screening tests: cardiac biomarkers (creatine kinase, troponin), ECG
- For arrhythmia: expedited cardiology evaluation indicated
- Grade 3
- Symptoms at rest or with minimal activity or exertion, or new onset of symptoms: may include chest pain, myalgia, dyspnea, arrhythmia, palpitations, peripheral edema, pleural effusion, fatigue
- Pericarditis with physiologic consequences (eg, pericardial constriction)
- Cardiac biomarkers (creatine kinase and troponin) >ULN
- Significant echocardiogram findings without hypotension

#### Grade 4

- Moderate to severe decompensation (worsening signs and symptoms): may include congestive heart failure, chest pain, myalgia, dyspnea on exertion, arrhythmia, palpitations, peripheral edema, pleural effusion, fatigue
- Hemodynamic instability (hypotension/cardiomyopathy)
- ullet Cardiac biomarkers (creatine kinase and troponin)  $> 3 \times$  ULN
- Life-threatening
- Urgent intervention indicated (eg, continuous intravenous therapy or mechanical hemodynamic support for myocarditis)

Abbreviations: ECG, electrocardiogram; irAEs, immune-related adverse events; ULN, upper limit of normal.

<sup>a</sup>For all adverse events, grade 5 is defined as death.

<sup>b</sup>Cardiovascular events that can be associated with cancer immunotherapy. Definitions incorporate elements from CTCAE version 5.0 (myocarditis, pericarditis, ventricular arrhythmia),<sup>41</sup> Brahmer et al,<sup>42</sup> and additions from the NCCN Panel (see ICI CARDIO-1 footnotes, page 235).

are limited to a number of single case reports with favorable outcomes. <sup>62,67,71</sup> Infliximab has also been used in cases studies to treat cardiotoxicities, <sup>61,67,71,74</sup> but it is important to note that it is contraindicated for patients who have heart failure. <sup>29,77</sup> IVIG is used to reduce the levels of antibodies that may be causing damage. IVIG was successfully used in a case report of smoldering ICI-related myocarditis that initially responded to corticosteroids but flared upon taper, <sup>68</sup> and has been used for years in the setting of cardiac rejection. <sup>73,75</sup> Mycophenolate mofetil is an antiproliferative agent that is used for cardiac transplant patients. <sup>76</sup>

Two additional immunosuppressive agents may be used based on case studies. A case report of a patient on pembrolizumab with confirmed myositis—myasthenia gravis overlap syndrome with worsening cardiac arrhythmia after methylprednisolone, mycophenolate, plasmapheresis, and rituximab described a successful outcome after treatment with alemtuzumab, 65 a monoclonal antibody that binds to

CD52 on some immune cells and leads to destruction of peripheral immune cells. Similarly, one case reported success using abatacept<sup>78</sup> (a CTLA-4 agonist that affects T cells and may lead to rapid inactivation of the normal immune response) in a patient receiving nivolumab who developed glucocorticoid-refractory myocarditis with concurrent myositis, who had also been treated with plasmapheresis.

#### **Conclusions**

Proper management of ICI-related toxicities requires early identification of potential irAEs in order to administer adequate treatment. Recent case studies and clinical experience have changed irAE management strategies, which have been incorporated in the 2020 update of NCCN Guidelines for Management of Immunotherapy-Related Toxicities. These NCCN Guidelines Insights provide context for topics that were discussed by the panel during the 2020 update meeting.



To participate in this journal CE activity, go to https://education.nccn.org/node/86963

#### References

- Keytruda (pembrolizumab) for injection, for intravenous use [prescribing information]. Whitehouse Station, NJ: Merck & Co, Inc.; 2019. Available at: https://www.accessdata.fda.gov/drugsatfda docs/label/2019/ 125514s065lbl.pdf. Accessed September 1, 2019.
- Opdivo (nivolumab) injection, for intravenous use [prescribing information]. Princeton, NJ: Bristol-Myers Squibb Company; 2019. Available at: https:// www. access data.fda.gov/drugs atf da.docs/label/2019/125554s075lbl.pdf.Accessed September 1, 2019.
- Tecentriq (atezolizumab) injection, for intravenous use [prescribing information]. South San Francisco, CA: Genentech, Inc.; 2019. Available at: https://www.accessdata.fda.gov/drugsatfda docs/label/2019/ 761034s021lbl.pdf. Accessed December 1, 2019.
- Bavencio (avelumab) injection, for intravenous use [prescribing information]. Rockland, MA: EMD Serono, Inc; 2019. Available at: https:// www.accessdata.fda.gov/drugsatfda docs/label/2019/761049s006lbl. pdf. Accessed May 1, 2019.
- Yervoy (ipilimumab) injection, for intravenous use [prescribing information]. Princeton, NJ: Bristol-Myers Squibb Company; 2019. Available at: https:// www.accessdata.fda.gov/drugsatfda docs/label/2019/125377s104lbl.pdf. Accessed September 1, 2019.
- Imfinzi (durvalumab) injection, for intravenous use [prescribing information]. Cambridge, England: AstraZeneca UK Limited; 2019. Available at: https://www.accessdata.fda.gov/drugsatfda docs/label/2019/ 761069s013lbl.pdf. Accessed July 2019.
- Seidel JA, Otsuka A, Kabashima K. Anti-PD-1 and anti-CTLA-4 therapies in cancer: mechanisms of action, efficacy, and limitations. Front Oncol
- Libtayo (cemiplimab) injection, for intravenous use [prescribing Information]. Tarrytown, NY: Regeneron Pharmaceuticals, Inc.; 2019. Available at: https://www.accessdata.fda.gov/drugsatfda docs/label/ 2019/761097s001lbl.pdf. Accessed Mar 2019.
- Lam LH, Lin SD, Sun J. Pharmacokinetics and pharmacodynamics of immunotherapy. In: Patel SP, Kurzrock R, eds. Early Phase Cancer Immunotherapy. Manhattan, NY: Springer International Publishing, 2018:29-67.
- Gangadhar TC, Vonderheide RH. Mitigating the toxic effects of anticancer immunotherapy. Nat Rev Clin Oncol 2014;11:91-99
- Kong YC, Flynn JC. Opportunistic autoimmune disorders potentiated by immune-checkpoint inhibitors anti-CTLA-4 and anti-PD-1. Front Immunol
- Ledezma B, Heng A. Real-world impact of education: treating patients with ipilimumab in a community practice setting. Cancer Manag Res 2013;6:5–14.
- Maude SL, Barrett D, Teachey DT, et al. Managing cytokine release syndrome associated with novel T cell-engaging therapies. Cancer J 2014;20:119-122.
- Kumar V, Chaudhary N, Garg M, et al. Current diagnosis and management of immune related adverse events (irAEs) induced by immune checkpoint inhibitor therapy. Front Pharmacol 2017;8:49.
- Puzanov I, Diab A, Abdallah K, et al. Managing toxicities associated with immune checkpoint inhibitors: consensus recommendations from the Society for Immunotherapy of Cancer (SITC) Toxicity Management Working Group. J Immunother Cancer 2017;5:95.
- Boutros C, Tarhini A, Routier E, et al. Safety profiles of anti-CTLA-4 and anti-PD-1 antibodies alone and in combination. Nat Rev Clin Oncol 2016; 13:473-486.

- Robert C, Long GV, Brady B, et al. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med 2015;372:320-330.
- Ferris RL, Blumenschein G Jr, Fayette J, et al. Nivolumab vs investigator's choice in recurrent or metastatic squamous cell carcinoma of the head and neck: 2-year long-term survival update of CheckMate 141 with analyses by tumor PD-L1 expression. Oral Oncol 2018;81:45-51.
- Hodi FS, Chiarion-Sileni V, Gonzalez R, et al. Nivolumab plus ipilimumab or nivolumab alone versus ipilimumab alone in advanced melanoma (CheckMate 067): 4-year outcomes of a multicentre, randomised, phase 3 trial. Lancet Oncol 2018;19:1480-1492.
- Topalian SL, Hodi FS, Brahmer JR, et al. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med 2012;366: 2443-2454
- 21. Agrawal S, Feng Y, Roy A, et al. Nivolumab dose selection: challenges, opportunities, and lessons learned for cancer immunotherapy. J Immunother Cancer 2016;4:72.
- 22. Hamid O, Robert C, Daud A, et al. Five-year survival outcomes for patients with advanced melanoma treated with pembrolizumab in KEYNOTE-001. Ann Oncol 2019;30:582-588.
- 23. Hamid O, Puzanov I, Dummer R, et al. Final analysis of a randomised trial comparing pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory advanced melanoma. Eur J Cancer 2017;86:37–45.
- 24. Schachter J, Ribas A, Long GV, et al. Pembrolizumab versus ipilimumab for advanced melanoma: final overall survival results of a multicentre randomised, open-label phase 3 study (KEYNOTE-006). Lancet 2017;390: 1853-1862
- Postow MA, Sidlow R, Hellmann MD. Immune-related adverse events associated with immune checkpoint blockade. N Engl J Med 2018;378: 158-168.
- Weber JS, Postow M, Lao CD, et al. Management of adverse events following treatment with anti-programmed death-1 agents. Oncologist 2016;21:1230-1240.
- $Ryder\ M,\ Callahan\ M,\ Postow\ MA,\ et\ al.\ Endocrine-related\ adverse\ events$ following ipilimumab in patients with advanced melanoma: a comprehensive retrospective review from a single institution. Endocr Relat Cancer 2014;21:371-381.
- 28. González-Rodríguez E, Rodríguez-Abreu D. Immune checkpoint inhibitors: review and management of endocrine adverse events. Oncologist 2016;21:804-816.
- 29. Ganatra S, Neilan TG. Immune checkpoint inhibitor-associated myocarditis. Oncologist 2018;23:879-886.
- Kadota H, Gono T, Shirai Y, et al. Immune checkpoint inhibitor-induced 30 myositis: a case report and literature review. Curr Rheumatol Rep 2019;21:10.
- Anquetil C, Salem JE, Lebrun-Vignes B, et al. Immune checkpoint inhibitor-associated myositis. Circulation 2018;138:743-745.
- Touat M, Maisonobe T, Knauss S, et al. Immune checkpoint inhibitorrelated myositis and myocarditis in patients with cancer. Neurology 2018; 91:e985-994.
- Wang DY, Salem JE, Cohen JV, et al. Fatal toxic effects associated with immune checkpoint inhibitors: a systematic review and meta-analysis. JAMA Oncol 2018;4:1721-1728.
- Moslehi JJ, Salem JE, Sosman JA, et al. Increased reporting of fatal immune checkpoint inhibitor-associated myocarditis. Lancet 2018;391:933.

- Weber JS, Dummer R, de Pril V, et al. Patterns of onset and resolution of immune-related adverse events of special interest with ipilimumab: detailed safety analysis from a phase 3 trial in patients with advanced melanoma. Cancer 2013;119:1675–1682.
- Wang Y, Abu-Sbeih H, Mao E, et al. Endoscopic and histologic features of immune checkpoint inhibitor-related colitis. Inflamm Bowel Dis 2018;24: 1695–1705.
- Gupta A, De Felice KM, Loftus EV Jr, et al. Systematic review: colitis associated with anti-CTLA-4 therapy. Aliment Pharmacol Ther 2015;42: 406–417
- Pernot S, Ramtohul T, Taieb J. Checkpoint inhibitors and gastrointestinal immune-related adverse events. Curr Opin Oncol 2016;28: 264–268.
- Tandon P, Bourassa-Blanchette S, Bishay K, et al. The risk of diarrhea and colitis in patients with advanced melanoma undergoing immune checkpoint inhibitor therapy: a systematic review and meta-analysis. J Immunother 2018;41:101–108.
- Wang DY, Ye F, Zhao S, et al. Incidence of immune checkpoint inhibitorrelated colitis in solid tumor patients: a systematic review and metaanalysis. Oncolmmunology 2017;6:e1344805.
- National Cancer Institute, Division of Cancer Treatment & Diagnosis. Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Bethesda, MD: US Department of Health and Human Services; 2017. Available at: https://ctep.cancer.gov/protocol/Development/electronic applications/ctc.htm#ctc 50. Accessed December 1, 2019.
- Brahmer JR, Lacchetti C, Schneider BJ, et al. Management of immunerelated adverse events in patients treated with immune checkpoint inhibitor therapy: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol 2018;36:1714–1768.
- Abu-Sbeih H, Ali FS, Luo W, et al. Importance of endoscopic and histological evaluation in the management of immune checkpoint inhibitorinduced colitis. J Immunother Cancer 2018;6:95.
- Dai C, Jiang M, Sun MJ, et al. Fecal lactoferrin for assessment of inflammatory bowel disease activity: a systematic review and meta-analysis [published online April 15, 2019]. J Clin Gastroenterol, doi: 10.1097/ MCG.000000000001212
- Wang Y, Pei F, Wang X, et al. Diagnostic accuracy of fecal lactoferrin for inflammatory bowel disease: a meta-analysis. Int J Clin Exp Pathol 2015;8: 12319–12332.
- Geukes Foppen MH, Rozeman EA, van Wilpe S, et al. Immune checkpoint inhibition-related colitis: symptoms, endoscopic features, histology and response to management. ESMO Open 2018;3:e000278.
- Wang Y, Abu-Sbeih H, Mao E, et al. Immune-checkpoint inhibitor-induced diarrhea and colitis in patients with advanced malignancies: retrospective review at MD Anderson. J Immunother Cancer 2018;6:37.
- Jain A, Lipson EJ, Sharfman WH, et al. Colonic ulcerations may predict steroid-refractory course in patients with ipilimumab-mediated enterocolitis. World J Gastroenterol 2017;23:2023–2028.
- Sfikakis PP. The first decade of biologic TNF antagonists in clinical practice: lessons learned, unresolved issues and future directions. Curr Dir Autoimmun 2010;11:180–210.
- 50. Reimold AM. TNFalpha as therapeutic target: new drugs, more applications. Curr Drug Targets Inflamm Allergy 2002;1:377–392.
- 51. Wolfe RM, Ang DC. Biologic therapies for autoimmune and connective tissue diseases. Immunol Allergy Clin North Am 2017;37:283–299.
- Friedman CF, Proverbs-Singh TA, Postow MA. Treatment of the immunerelated adverse effects of immune checkpoint inhibitors: a review. JAMA Oncol 2016;2:1346–1353.
- Pagès C, Gornet JM, Monsel G, et al. Ipilimumab-induced acute severe colitis treated by infliximab. Melanoma Res 2013;23:227–230.
- Merrill SP, Reynolds P, Kalra A, et al. Early administration of infliximab for severe ipilimumab-related diarrhea in a critically ill patient. Ann Pharmacother 2014;48:806–810.
- Entyvio (vedolizumab) for injection, for intravenous use [prescribing information]. Deerfield, IL: Takeda Pharmaceuticals America, Inc; 2019.
   Available at: https://www.accessdata.fda.gov/drugsatfda docs/label/2019/125476s024lbl.pdf. Accessed May 2019.

- Bergqvist V, Hertervig E, Gedeon P, et al. Vedolizumab treatment for immune checkpoint inhibitor-induced enterocolitis. Cancer Immunol Immunother 2017;66:581–592.
- Diana P, Mankongpaisarnrung C, Atkins MB, et al. Emerging role of vedolizumab in managing refractory immune checkpoint inhibitorinduced enteritis. ACG Case Rep J 2018;5:e17.
- Hsieh AH, Ferman M, Brown MP, Andrews JM. Vedolizumab: a novel treatment of ipilimumab-induced colitis. BMJ Case Rep 2016;2016: bcr2016216641.
- Abu-Sbeih H, Ali FS, Wang X, et al. Early introduction of selective immunosuppressive therapy associated with favorable clinical outcomes in patients with immune checkpoint inhibitor-induced colitis. J Immunother Cancer 2019;7:93.
- Wang Y, Wiesnoski DH, Helmink BA, et al. Fecal microbiota transplantation for refractory immune checkpoint inhibitor-associated colitis [errata appears in Nat Med 2019;25:188]. Nat Med 2018;24:1804–1808.
- Heinzerling L, Ott PA, Hodi FS, et al. Cardiotoxicity associated with CTLA4 and PD1 blocking immunotherapy. J Immunother Cancer 2016;4:50.
- Mahmood SS, Fradley MG, Cohen JV, et al. Myocarditis in patients treated with immune checkpoint inhibitors. J Am Coll Cardiol 2018;71:1755–1764.
- Johnson DB, Balko JM, Compton ML, et al. Fulminant myocarditis with combination immune checkpoint blockade. N Engl J Med 2016;375: 1749–1755.
- Yun S, Vincelette ND, Mansour I, et al. Late onset ipilimumab-induced pericarditis and pericardial effusion: a rare but life threatening complication. Case Rep Oncol Med 2015;2015:794842.
- Esfahani K, Buhlaiga N, Thébault P, et al. Alemtuzumab for immune-related myocarditis due to PD-1 therapy. N Engl J Med 2019;380:2375–2376.
- Varricchi G, Marone G, Mercurio V, et al. Immune checkpoint inhibitors and cardiac toxicity: an emerging issue. Curr Med Chem 2018;25:1327–1339.
- Agrawal N, Khunger A, Vachhani P, et al. Cardiac toxicity associated with immune checkpoint inhibitors: case series and review of the literature. Case Rep Oncol 2019;12:260–276.
- Norwood TG, Westbrook BC, Johnson DB, et al. Smoldering myocarditis following immune checkpoint blockade. J Immunother Cancer 2017;5:91.
- Tajmir-Riahi A, Bergmann T, Schmid M, et al. Life-threatening autoimmune cardiomyopathy reproducibly induced in a patient by checkpoint inhibitor therapy. J Immunother 2018;41:35–38.
- Aquaro GD, Perfetti M, Camastra G, et al. Cardiac MR with late gadolinium enhancement in acute myocarditis with preserved systolic function: ITAMY study. J Am Coll Cardiol 2017;70:1977–1987.
- 71. Tay RY, Blackley E, McLean C, et al. Successful use of equine antithymocyte globulin (ATGAM) for fulminant myocarditis secondary to nivolumab therapy. Br J Cancer 2017;117:921–924.
- Jain V, Bahia J, Mohebtash M, et al. Cardiovascular complications associated with novel cancer immunotherapies. Curr Treat Options Cardiovasc Med 2017;19:36.
- Kobashigawa J, Crespo-Leiro MG, Ensminger SM, et al. Report from a consensus conference on antibody-mediated rejection in heart transplantation. J Heart Lung Transplant 2011;30:252–269.
- Frigeri M, Meyer P, Banfi C, et al. Immune checkpoint inhibitor-associated myocarditis: a new challenge for cardiologists. Can J Cardiol 2018;34: 92.e1–92.e3.
- Rodriguez ER, Skojec DV, Tan CD, et al. Antibody-mediated rejection in human cardiac allografts: evaluation of immunoglobulins and complement activation products C4d and C3d as markers. Am J Transplant 2005; 5:2778, 2785
- Kobashigawa JA, Miller LW, Russell SD, et al. Tacrolimus with mycophenolate mofetil (MMF) or sirolimus vs. cyclosporine with MMF in cardiac transplant patients: 1-year report. Am J Transplant 2006;6:1377–1386.
- Kwon HJ, Coté TR, Cuffe MS, et al. Case reports of heart failure after therapy with a tumor necrosis factor antagonist. Ann Intern Med 2003; 138:807–811.
- Salem JE, Allenbach Y, Vozy A, et al. Abatacept for severe immune checkpoint inhibitor-associated myocarditis. N Engl J Med 2019;380: 2377–2379

## Signature Page for VV-CLIN-001702 v1.0 Prot\_XmAb18087-02\_v1.0\_18Aug2020\_CLEAN

| Approval | |
|----------|-------------------------------|
| | 20-Aug-2020 23:36:07 GMT+0000 |

## Signature Page for VV-CLIN-001702 v1.0 Prot\_XmAb18087-02\_v1.0\_18Aug2020\_CLEAN

| Approval | |
|----------|-------------------------------|
| | 20-Aug-2020 23:36:07 GMT+0000 |